# Replication of the DAPA-CKD (Chronic Kidney Disease) Trial in Healthcare Claims Data

DUPLICATE DAPA-CKD

September 14, 2021

NCT04882813

#### 1. RCT Details

This section provides a high-level overview of an RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Dapagliflozin in Patients with Chronic Kidney Disease (<u>DAPA-CKD</u> trial)

### 1.2 <u>Intended aim(s)</u>

The objective of the study is to assess the long-term efficacy and safety of dapagliflozin, a sodium-glucose cotransporter 2 (SGLT2) inhibitor in patients with chronic kidney disease, with or without type 2 diabetes

### 1.3 Primary endpoint for replication and RCT finding

Composite of a sustained decline in the estimated glomerular filtration rate (GFR) of at least 50%, end-stage kidney disease, or death from renal or cardiovascular causes.

### 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

With the recruitment of at least 4000 patients, the trial will have 90% power to detect a relative risk reduction of 22% in the primary endpoint based on primary events being observed in 681 patients and a two-sided P-value of 0.05.

### 1.5 <u>Trial estimate</u>

HR = 0.64 (95% CI 0.52–0.79) comparing dapagliflozin to placebo among patients with Type 2 DM and HR = 0.61 (95% CI 0.51-0.75) among patients with and without Type 2 DM (Heerspink et al., 2020, NEJM)

### 2. Person responsible for implementation of replication in Aetion

Helen Tesfaye, Pharm.D, ScM implemented the study design in the Aetion Evidence Platform. She is not responsible for the validity of design and analytic choices. All implementation steps are recorded, and implementation history is archived in the platform.

### 3. Data Source(s)

Optum Cliniformatics Data Mart, IBM MarketScan, Medicare

Effectiveness research with Real World Data to support FDA's regulatory decision making

### 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expediated review.

### Design Diagram - DAPA-CKD TRIAL REPLICATION



#### 5. Cohort Identification

#### 5.1 Cohort Summary

This study will involve a new user, parallel group retrospective cohort study design comparing dapagliflozin to sitagliptin. Although the trial compared dapagliflozin to placebo, for the current emulation we used an active comparator, sitagliptin, which is a dipeptidyl peptidase-4 (DPP-4) inhibitor. This is because both dapagliflozin and sitagliptin are guideline recommended as second to third line therapies used for the treatment of type 2 diabetes at the same stage of the disease and sitagliptin is not expected to have an effect on the primary outcome.

The patients will be required to have continuous enrollment during baseline period of 180 days before initiation of dapagliflozin or sitagliptin (cohort entry).

### 5.2 Important steps for cohort formation

New users (defined as no use in 180 days prior to index date) of an exposure, dapagliflozin and a comparator, sitagliptin, will be identified.

### 5.2.1 Eligible cohort entry date

Dapagliflozin was approved by FDA for market availability on January 8, 2014.

- Optum: January 8, 2014 March 31, 2020 (end of data availability)
- Marketscan: January 8, 2014 December 31, 2018 (end of data availability)
- Medicare: January 8, 2014 December 31, 2017 (end of data availability)

### 5.2.2 Specify inclusion/exclusion criteria for cohort entry and define the index date

Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

### 5.3 Flowchart of the study cohort assembly

| | Optum | | Marke | tscan | Medi | care |
|---|---|---|---|---|---|---|
| | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients |
| All patients | | 78,202,636 | | 200,203,908 | | 23,466,175 |
| Did not meet cohort entry criteria | -77,797,182 | 405,454 | -199,563,302 | 640,606 | -22,268,953 | 1,197,222 |
| Excluded due to insufficient enrollment | -66,483 | 338,971 | -58,936 | 581,670 | -333,159 | 864,063 |
| Excluded due to prior use of referent | -245,915 | 93,056 | -397,135 | 184,535 | -679,548 | 184,515 |
| Excluded due to prior use of exposure | -21,695 | 71,361 | -95,936 | 88,599 | -27,223 | 157,292 |
| Excluded because patient qualified in >1 exposure category | -36 | 71,325 | -346 | 88,253 | -108 | 157,184 |
| Excluded based on Age | 0 | 71,325 | 0 | 88,253 | -28 | 157,156 |
| Excluded based on Gender | -7 | 71,318 | 0 | 88,253 | 0 | 157,156 |
| Excluded based on Inclusion #1 - Age ≥ 18 years or older | -7 | 71,311 | -54 | 88,199 | -692 | 156,464 |
| Excluded based on Inclusion #2 - eGFR ≥30 and ≤75 mL/min/1.73 m2 (CKD-EPI formula)_ONLY STAGE II & III | -41,866 | 29,445 | -73,659 | 14,540 | -82,143 | 74,321 |
| Excluded based on Inclusion #4 - Treatment with ACEi or ARB for at least 4 weeks, if not medically contraindicated | -4,797 | 24,648 | -2,385 | 12,155 | -12,272 | 62,049 |
| Excluded based on Inclusion #5 - Type 2 DM | -32 | 24,616 | -29 | 12,126 | -45 | 62,004 |
| Excluded based on Exclusion #2 - Autosomal dominant or autosomal recessive polycystic kidney disease, lupus nephritis or Antineutrophil cytoplasmic antibody (ANCA) | -1,060 | 23,556 | -650 | 11,476 | -3,273 | 58,731 |
| Excluded based on Exclusion #3 - Receiving cytotoxic therapy, immunosuppresive therapy or other immunotherapy | -65 | 23,491 | -15 | 11,461 | -97 | 58,634 |
| Excluded based on Exclusion #4 - NYHA class IV CHF - measured as LVAD/Implantable heart | -1 | 23,490 | -1 | 11,460 | -14 | 58,620 |
| Excluded based on Exclusion #5 - MI, Unstable angina, Stroke, Transient Ischemic Attack | -248 | 23,242 | -151 | 11,309 | -1,427 | 57,193 |
| Excluded based on Exclusion # 6-Coronary revascularization (PCI or CABG) or valvular repair/replacement | -18 | 23,224 | -7 | 11,302 | -58 | 57,135 |
| Excluded based on Exclusion #8 - Presence of hepatic impairment | -195 | 23,029 | -65 | 11,237 | -472 | 56,663 |

| Excluded based on Exclusion #9 - History of Organ Transplant | -33 | 22,996 | -14 | 11,223 | -98 | 56,565 |
|---|---|---|---|---|---|---|
| Excluded based on Exclusion #10 - Receiving therapy with SGLT2 inhibitor | -170 | 22,826 | -83 | 11,140 | -219 | 56,346 |
| Excluded based on Exclusion #11a - Acute kidney injury (AKI) | -327 | 22,499 | -82 | 11,058 | -798 | 55,548 |
| Excluded based on Exclusion #11b - Baseline CKD IV & V, ESRD, HD/PD | -360 | 22,139 | -118 | 10,940 | -949 | 54,599 |
| Final cohort | | 22,139 | | 10,940 | | 54,599 |

#### 6 Variables

#### 6.1 Exposure-related variables:

#### Study drug:

The study exposure of interest is initiation of dapagliflozin (SGLT2i at any dose and frequency. Initiation will be defined by no use of dapagliflozin during the prior 180 days before treatment initiation (washout period). Patients are required to be incident users with respect both exposure groups.

### **Comparator agents:**

Initiators of sitagliptin, any dose and frequency.

### 6.2 Preliminary Covariates:

- Age
- Sex
- Combined Comorbidity Index (CCI), measured over the default baseline covariate assessment period of 180 days prior to and including the index prescription date

Covariates listed above are a small subset of covariates that will ultimately be controlled in the design and analysis phase of the study. They are included in the preliminary assessment to determine the presence of adequate overlap between the two population of patients to proceed to the next phase of the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and initial power assessment and are listed in Table 1 (Appendix B).

### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcome variables of interest (definitions provided in **Appendix A**):

- Primary outcome: Composite of end stage renal disease (ESRD) or all-cause mortality
- Secondary outcomes:
  - o ESRD
  - All-cause death

Control outcomes of interest (control outcomes only serve to assess aspects of study validity but are not further interpreted):

#### Control outcome definitions

Genital infections

### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analysis will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real-world databases is expected to be much worse than in the trial, the AT analysis is the **primary** analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analysis, the follow-up will start the day after the initiation of dapagliflozin or sitagliptin and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest,
- The date of end of continue registration in the database,
- End of the study period,
- Death (for ESRD outcome only),
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.

- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (dapagliflozin or sitagliptin) + a 30-day grace period,
- The date of switching from an exposure to comparator and vice versa,
- The date of switching to or initiation of other SGLT2i (excluding dapagliflozin) and other DPP4i (excluding sitagliptin).

For the ITT analyses, the censoring based on the switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

### 7 Initial Feasibility Analysis

#### Aetion report name:

Optum- <a href="https://bwh-dope.aetion.com/projects/details/1379/results/66309/result/0">https://bwh-dope.aetion.com/projects/details/1379/results/66309/result/0</a>
Marketscan- <a href="https://bwh-dope.aetion.com/projects/details/1400/results/66311/result/0">https://bwh-dope.aetion.com/projects/details/1379/results/66311/result/0</a>
Medicare - <a href="https://bwh-dope.aetion.com/projects/details/1377/results/66055/result/0">https://bwh-dope.aetion.com/projects/details/1379/results/66311/result/0</a>

Date conducted: 2/25/2021

#### 8 Initial Power Assessment

### Aetion report name:

Optum- <a href="https://bwh-dope.aetion.com/projects/details/1379/results/66310/result/0">https://bwh-dope.aetion.com/projects/details/1379/results/66310/result/0</a>
Marketscan- <a href="https://bwh-dope.aetion.com/projects/details/1377/results/66056/result/0">https://bwh-dope.aetion.com/projects/details/1379/results/66310/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/projects/details/1377/results/66056/result/0">https://bwh-dope.aetion.com/projects/details/1379/results/66310/result/0</a>

Date conducted: 2/25/2021

• Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: | 2/26/2021 |
|-------------------------|----------------|----------------|-----------|
| Reviewed by FDA: | Kenneth Quinto | Date reviewed: | 3/16/2021 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 9. Balance Assessment

Optum- https://bwh-dope.aetion.com/projects/details/1379/rwrs/68008

Marketscan-https://bwh-dope.aetion.com/projects/details/1400/rwrs/68510

Medicare- https://bwh-dope.aetion.com/projects/details/1377/rwrs/68010

<u>Date conducted</u>: 4/02/2021, 4/16/2021 (Enrollment corrected for Marketscan)

After review of initial feasibility and power analyses, complete creation of the remaining covariates from Section 6.2. Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates.

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

• Report covariate balance after matching.

Note- For Table 1, please refer to Appendix B.

### • Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy outcome | 0 (0%) | 0 (0%) | 0 (0%) |
| Death | 64 (0.62%) | 44 (0.86%) | 20 (0.39%) |
| Start of an additional exposure | 638 (6.20%) | 41 (0.80%) | 597 (11.60%) |
| End of Index Exposure | 4,738 (46.04%) | 2,567 (49.89%) | 2,171 (42.20%) |
| Specified date reached | 2,374 (23.07%) | 1,323 (25.71%) | 1,051 (20.43%) |
| End of patient enrollment | 913 (8.87%) | 479 (9.31%) | 434 (8.44%) |
| Switch to other SGLT-2i + Switch to other DPP-4i + Nursing<br>Home admission occurred | 1,563 (15.19%) | 691 (13.43%) | 872 (16.95%) |

### • Report follow-up time by treatment group.

| Patient Group | Optum<br>Median<br>Follow-Up Time<br>(Days) [IQR] | Marketscan<br>Median<br>Follow-Up Time<br>(Days) [IQR] | Medicare<br>Median<br>Follow-Up Time<br>(Days) [IQR] |
|---|---|---|---|
| Overall Patient Population | 113 [58, 221] | 118 [58, 267] | 118 [58, 220] |
| Referent - Sitagliptin | 118 [58, 254] | 127 [69, 285] | 118 [58, 257] |
| Exposure - Dapagliflozin | 79 [52, 183] | 118 [58, 240] | 88 [55, 181] |

### • Report overall risk of the primary outcome.

| | Optum | MarketScan | Medicare | Pooled |
|-------------------------|-------|------------|----------|--------|
| Risk per 1,000 patients | 15.6 | 3.3 | 25.5 | 20.2 |

### **10. Final Power Assessment**

<u>Date conducted</u>: 4/02/2021, 4/16/2021 (Marketscan only)

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8.

| Superiority Analysis (Booled) | |
|-------------------------------|----------|
| Superiority Analysis (Pooled) | |
| Number of patients matched | |
| Reference | 5145.0 |
| Exposed | 5145.0 |
| Risk per 1,000 patients | 20.22 |
| Desired HR from RCT | 0.64 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 208.0638 |
| Power | 0.90 |

| Superiority Analysis (Optum) | |
|------------------------------|-------------|
| Number of patients matched | |
| Reference | 828 |
| Exposed | 828 |
| Risk per 1,000 patients | 15.60 |
| Desired HR from RCT | 0.64 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 25.8336 |
| Power | 0.205446437 |

| Superiority Analysis (Marketscan) | |
|-----------------------------------|-------------|
| Number of patients matched | |
| Reference | 1,687 |
| Exposed | 1,687 |
| Risk per 1,000 patients | 3.30 |
| Desired HR from RCT | 0.64 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 11.1342 |
| Power | 0.115530515 |

| Superiority Analysis (Medicare) | |
|---------------------------------|-------------|
| Number of patients matched | |
| Reference | 2,630 |
| Exposed | 2,630 |
| Risk per 1,000 patients | 25.50 |
| Desired HR from RCT | 0.64 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 134.13 |
| Power | 0.733807835 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Date reviewed: |
|-------------------------|----------------|
| Reviewed by FDA: | Date reviewed: |
| Reasons for stopping | |
| analysis (if required): | |

### Appendix A: Composite of ESRD or all-cause mortality

Measured 1 day after drug initiation in diagnosis position specified below and inpatient and outpatient care setting -

#### **Composite of ESRD or All-Cause Mortality**

#### **ESRD**

ICD-9 diagnosis: 585.5, 585.6 ICD-10 diagnosis: N18.5, N18.6

AND

#### **Dialysis**

ICD-9 diagnosis: V45.1x, V56.0x, V56.1, V56.8x ICD-10 diagnosis: Z49.01, Z49.31, Z49.32, Z99.2

ICD-9 procedure: 39.95, 54.98

ICD-10 procedure: 3E1M39z, 5A1D00z, 5A1D60Z

CPT: S9339, 90945, 90947, 90999

-----

OR

#### CV death

Inpatient mortality - renal or CV causes --

Mortality- Dependent on data source.

1. CV mortality

Information on CV mortality through data linkage with the National Death Index (NDI) will be available for Medicare and Optum Clinformatics.

2. All-cause inpatient mortality

Identified using the discharge status codes-

Optum-

- 20 = EXPIRED
- 21 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 22 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 23 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 24 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 25 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 26 = EXPIRED TO BE DEFINED AT STATE LEVEL

- 27 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 28 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 29 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 40 = EXPIRED AT HOME (HOSPICE)
- 41 = EXPIRED IN A MEDICAL FACILITY (HOSPICE)
- 42 = EXPIRED PLACE UNKNOWN (HOSPICE)

#### Truven-

- 20 Died
- 22 Died
- 23 Died
- 24 Died
- 25 Died
- 26 Died
- 27 Died
- 28 Died
- 29 Died
- 40 Other died status or Expired at home (Hospice claims only) (depends on year)
- 41 Other died status or Expired in medical facility (Hospice claims only) (depends on year)
- 42 Other died status or Expired place unknown (Hospice claims only) (depends on year)
- 21 Died or Disch./Transf. to court/law enforcement (depends on year)

| # | DAPA-CKD trial definitions | Implementation in routine care | References/Rationale | Color coding |
|---|---|---|---|---|
| | Trial details - Intended S with label change - 2 | Please see the following Google Drive for further details or<br>any missing information:<br>https://drive.google.com/open?id=1WD618wrywYjEaXrfLT<br>cuK-VCcnb6b_gV | Criteria | |
| | EXPOSURE vs. COMPARISON | ICD-10 codes are not listed in this document because of excel cell size limitations and excessive number of ICD-10 codes. Full ICD-10 code lists will be available in the above Google Drive Folder (link above). ICD-9 to ICD-10 code conversions were completed using a SAS macro that implements forward/ backward mapping based on the CMS ICD-9 to ICD-10 mapping: https://www.nber.org/data/icd9-icd-10-cm-and-pcs-crosswalk-general-equivalence-mapping.html | Adequate mapping in claims | |
| | Dapagliflozin 10 mg or 5 mg tablets once daily vs. placebo matching dapagliflozin 10 mg or 5 mg <u>Aim</u> : To evaluate the effect of dapagliflozin on renal outcomes and CV mortality in patients with CKD | Dapagliflozin 10 mg or 5 mg vs.Sitagliptin (any dose) <u>Exposure</u> : new-use dapagliflozin <u>Reference</u> : Sitagliptin | | Intermediate mapping in claims |
| | PRIMARY OUTCOME | | | Poor mapping or cannot be measured in claims |
| | Primary endpoint: A composite of sustained decline in eGFR of >= 50%, ESRD, renal death or CV death 1) time to >=50% eGFR decline from baseline (confirmed by >=28-day SCr) 2) time to ESRD defined as eGFR <15 ml/min/1.73 m2, need for chronic dialysis (both confirmed after >= 28 days) and renal transplantation 3) time to renal or CV death | Measured 1 day after drug initiation in any diagnosis position in inpatient and outpatient care setting: Composite of ESRD or All-Cause Mortality ESRD ICD-9 diagnosis: 585.5, 585.6 ICD-10 diagnosis: N18.5, N18.6 AND Dialysis ICD-9 diagnosis: V45.1x, V56.0x, V56.1, V56.8x ICD-10 diagnosis: 249.01, Z49.31, Z49.32, Z99.2 ICD-9 procedure: 39.95, 54.98 ICD-10 procedure: 38.1M39z, 5A.1D00z, 5A.1D60z CPT: S9339, 90945, 90947, 90999 OR CV death Inpatient mortality - renal or CV causes Mortality- Dependent on data source. | | Can't be measured in claims but not important for the analysis |
| | Dapagliflozin 10 mg or 5 mg tablets once daily vs. placebo matci | | | |
| | Aim: To evaluate the effect of dapagliflozin on renal outcomes and | | | |
| 1 | 18 years of age | Measured on the day of drug initiation<br>Age >= 18 | | |

| 2 | eGFR ≥25 and ≤75 mL/min/1.73 m2 (CKD-EPI formula) at visit 1 | Measured any time prior to and including the day of drug initiation in any diagnosis position and inpatient and outpatient care setting: CKD Stage III (eGFR 60 - 89 mL/min/1.73 m2) ICD-9 diagnosis: 585.2 ICD-10 diagnosis: N18.2 ICD-10 diagnosis: N18.2 ICD-9 diagnosis: 585.3 ICD-10 diagnosis: S85.3 ICD-10 diagnosis: N18.3 ICD-9 diagnosis: N18.3 ICD-10 diagnosis: N | |
|---|---|---|---|
| 3 | Evidence of increased albuminuria for 3 months or more before visit 1 and UACR ≥200 and ≤5000 mg/g at visit 1 | ICD-9 diagnosis: 585.4 ICD-10 diagnosis: N18.4 Measured from the start of all available data until 90 days prior to the date of drug initiation in any diagnosis position and inpatient and outpatient care setting: Proteinuria ICD-9 diagnosis: 791.0 ICD-10 diagnosis: R80.x | |
| 4 | Stable, and for the patient maximum tolerated labelled daily dose, treatment with ACEI or ARB for at least 4 weeks before visit 1, if not medically contraindicated | Measured 45 days prior to index drug initiation in prescription claims requiring 28 days supply of ACE or ARB: <u>ACE inibitors' generic names for prescription claims:</u> Enalapril, Captopril, Ciazapril, Fosinopril, Lisinopril, Moexipril, Perindopril, Quinapril, Ramipril, Trandolapril, Zofenopril, Benazepril OR <u>ARBs generic names for prescription claims:</u> Candesartan, Eprosartan, Irbesartan, Losartan, Olmesartan, Telmisartan, Valsartan, Azilsartan | |
| | EXCLUSION CRITERIA | <u> </u> | |
| 1 | Type I diabetes mellitus | Measured from the start of all available data to and including the day of drug initiation in any diagnosis position and inpatient and outpatient care setting: Type I DIM ICD-9 diagnosis: 250.01, 250.03, 250.11, 250.13, 250.21, 250.23, 250.31, 250.33, 250.41, 250.43, 250.51, 250.53, 250.61, 250.63, 250.71, 250.73, 250.91, 250.93 ICD-10 diagnosis: E10.x | |
| 2 | Autosomal dominant or autosomal recessive polycystic kidney disease, lupus nephritis or Antineutrophil cytoplasmic antibody<br>(ANCA) -associated vasculitis | Measured from the start of all available data to and including the day of drug initiation in any diagnosis position and inpatient and outpatient care setting: Autosomal dominant or recessive PKD ICD-9 diagnosis: 753.12, 753.13, 753.14 ICD-10 diagnosis: Q61.3, Q61.2, Q61.19 Lupus nephritis ICD-9 diagnosis: 710.0, 583.x ICD-10 diagnosis: N05.2, N05.5, N05.9 ANCA-associated vasculitis ICD-9 diagnosis: 446.0, 446.4, 447.6, 446.7 ICD-10 diagnosis: M30.3, M31.30, M31.4, I77.6 | Sreih AG, Annapureddy N, Springer J, et al. Development and validation of case-finding algorithms for the identification of patients with anti-neutrophil cytoplasmic antibody-associated vasculitis in large healthcare administrative databases. Pharmacoepidemiol Drug Saf. 2016;25(12):1368–1374. doi:10.1002/pds.4116 Chibnik LB, Massarotti EM, Costenbader KH. Identification and validation of lupus nephritis cases using administrative data. Lupus. 2010;19(6):741–743. doi:10.1177/0961203309356289 |

| _ | | Measured 180 days prior to and including the day of drug initiation in prescription claims: |
|---|---|---|
| | | Membranous nephropathy |
| | | ICD-9 diagnosis: 583.1, 583.2 |
| | | ICD-10 diagnosis: N05.2, N05.5 |
| | | Glomerular disease (except chronic glomerulonephritis) |
| | | ICD-9 diagnosis: 580.x |
| | | ICD-10 dlagnosis: N00.x, N01.x, N02.x, N03.x, N04.x, N05.x, N06.x, N07.x, N08.x |
| | | Immunoglobulin A nephropathy (Berger's disease) |
| | Receiving cytotoxic therapy, immunosuppressive therapy or other immunotherapy for primary or secondary renal disease within | ICD-9 diagnosis: 583.9 ICD-10 diagnosis: N02.8 |
| 3 | 6 months prior to enrollment | TCP-10 diagnosis. Noz.o |
| | | Focal segmental glomerulosclerosis (FSGS) |
| | | ICD-9 diagnosis: 581.1 |
| | | ICD-10 diagnosis: N02.2 |
| 1 | | Conductive quidams |
| 1 | | Goodpasture syndrome ICD-9 diagnosis: 446.2x |
| | | 1CD-10 diagnosis: M3.0 |
| 1 | | ' |
| | | Hemolytic uremic syndrome (HUS) |
| | | ICD-9 diagnosis: 283.11 |
| | | ICD-10 diagnosis: D59.3 |
| | | Measured 180 days prior to and including the day of drug initiation in any diagnosis position |
| | | and inpatient and outpatient care setting: |
| | | LVAD/Implantable Heart |
| | | LVRL//milanture treat/<br>ICD-9 diagnosis: V43.2x |
| 4 | NYHA class IV congestive heart failure at the time of enrollment | ICD-10 diagnosis: 295.811, 295.812 |
| | | ICD-9 procedure: 37.60, 37.66 |
| | | ICD-10 procedure: 02HA0RS, 02HA3RS, 02HA4RS, 5A02116, 5A02216, 02HA0QZ, 02HA3QZ, |
| | | 02HA4QZ<br>CPT-4 code: 33975, 33976, 33979, 33981 - 33983, 33977, 33978, 33980 |
| | | LT 1-4 LUUE. 333/3, 333/6, 333/3, 33361 - 33363, 333/6, 333/6, 333/6 |
| 1 | | Measured 56 days prior to including the day of drug initiation in any diagnosis position and |
| 1 | | inpatient and ED care setting: |
| 1 | | Myocardial Infarction/STEMI |
| 1 | | ICD-9 diagnosis: 410.xx (exclude 410.x2), 411.0 |
| 1 | | ICD-10 diagnosis: I21.xx, I22.xx, I23.xx |
| 1 | | Lea |
| | | ACS: Unstable Angina<br>ICD-9 diagnosis: 413.xx (exclude 413.1), 411.1, 411.8, 411.81, 411.89 |
| 5 | MI, unstable angina, stroke, transient ischemic attack within 8 weeks prior to enrollment | ICD-10 diagnosis: 413.xx (exclude 413.1), 411.8, 411.81, 411.89<br>ICD-10 diagnosis: 120.xx (exclude 120.1), 124.xx (exclude 124.1) |
| 1 | | 1 |
| 1 | | <u>Stroke</u> |
| 1 | | ICD-9 diagnosis: 430.xx, 431.xx, 433.x1, 434.xx (excluding 434.x0), 436.x, 997.02 |
| 1 | | ICD-10 diagnosis: G97.3x, I60.xx, I61.xx I62.xx, I63.xx, I97.81x, I97.82x |
| 1 | | TIA. |
| 1 | | ICD-9 diagnosis: 435.xx |
| 1 | | ICD-10 diagnosis: G45.xx |
| 1 | | |
| | | I |


| 10 | <b>Receiving therapy with SGLT2 inhibitor</b> within 8 weeks prior to enrollment or previous intolerance of an SGLT2 inhibitor | Measured from 56 days prior to 1 day prior to drug initiation in prescription claims: SGIT2 Inhibitors (including combination products containing any of the following) - Canagliflozin (INVOKANA*) - Canagliflozin/metformin (INVOKAMET*, INVOKAMET* XR) - Empagliflozin/Larabin/metformin (SYNJARDY*, SYNJARDY* XR) - Empagliflozin/metformin (SYNJARDY*, SYNJARDY* XR) - Empagliflozin/linagliptin (GLYXAMBI*) - Dapagliflozin/linagliptin (GLYXAMBI*) - Dapagliflozin/metformin (XIGDUO* XR) - Dapagliflozin/metformin (XIGDUO* XR) - Dapagliflozin/saxagliptin (QTERN*) - Dapagliflozin/saxagliptin/metformin (QTERNMET* XR) - Ertugliflozin (STEGLATRO*) - Ertugliflozin/metformin (SEGLUROMET*) - Ertugliflozin/metformin (SEGLUROMET*) - Ertugliflozin/sitagliptin (STEGLUJAN*) |
|---|---|---|
| 11a | Exclude patients that have <b>AKI</b> during the baseline period | Measured from 14 days prior to and including the day of drug intiation in any diagnosis position and any care setting: <u>Acute kidney injury (AKI)</u> ICD-9 diagnosis: 584.xx, 586 ICD-10 diagnosis: NJ7.x, N19 |
| 11b | Exclude patients that have <b>CKD-V, ESRD and are on HD/PD</b> during the baseline period | Measured from 180 days prior to and including the day of drug intiation in any diagnosis position and any care setting: Chronic Kidney Disease (CKD)-V ICD-9 diagnosis: 585.5 ICD-10 diagnosis: N18.5 ESRD. ICD-9 diagnosis: 403.01, 403.11, 403.91, 404.03, 404.13, 585.6 ICD-10 diagnosis: 112.0, N18.6 Hemodialysis/Peritoneal Dialysis ICD-9 diagnosis: V45.1x, V56.xx, 996.56, 996.68, 996.73 ICD-10 diagnosis: 29.9x, 549.1x, 785.611x, 785.621x, 785.631x, 785.691x, 785.71x ICD-9 procedure: 39.9x, 54, 58.8 ICD-10 procedure: 5A1D702, 5A1D802, 5A1D902, 3E1M392 ICD-10 procedure: 5A1D702, 5A1D802, 5A1D902, 3E1M392 ICD-10 code: 90935, 90937, 90939 |

### Mortality-Dependent on data source. 1. All-cause mortality / inpatient mortality Identified using the vital status file-Medicare Identified using the discharge status codes-Optum-• 20 = EXPIRED • 21 = EXPIRED TO BE DEFINED AT STATE LEVEL • 22 = EXPIRED TO BE DEFINED AT STATE LEVEL • 23 = EXPIRED TO BE DEFINED AT STATE LEVEL • 24 = EXPIRED TO BE DEFINED AT STATE LEVEL • 25 = EXPIRED TO BE DEFINED AT STATE LEVEL • 26 = EXPIRED TO BE DEFINED AT STATE LEVEL • 27 = EXPIRED TO BE DEFINED AT STATE LEVEL • 28 = EXPIRED TO BE DEFINED AT STATE LEVEL • 29 = EXPIRED TO BE DEFINED AT STATE LEVEL • 40 = EXPIRED AT HOME (HOSPICE) • 41 = EXPIRED IN A MEDICAL FACILITY (HOSPICE) • 42 = EXPIRED - PLACE UNKNOWN (HOSPICE) Truven-• 20 - Died • 22 - Died • 23 - Died • 24 - Died • 25 - Died • 26 - Died • 27 - Died • 28 - Died • 29 - Died • 40 - Other died status or Expired at home (Hospice claims only) (depends on year) • 41 - Other died status or Expired in medical facility (Hospice claims only) (depends on year) • 42 - Other died status or Expired - place unknown (Hospice claims only) (depends on year) • 21 - Died or Disch./Transf. to court/law enforcement (depends on year)


| 1 | | | | | | | | 1 | | | - | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| March 1971 1971 1972 | | | | | | Bypass Coronary Artery, Four or More Arteries from | | | | | | | |
| March 1 | Backward (ICD10 to ICD9) | 0213083 | 02 13083 | 3619 | 36.19 | | Other hypass anastomosis for heart revascularization | Coronary artery hypass surgery Py | 2 Δnnroy 1·1 | 1 | 0 | 0 | 0 |
| March Marc | Sackward (res to to ress) | 0213003 | 02.13003 | 3013 | 30.13 | - Ab | Other bypass and to most stories and the control of | coronary artery bypass surgery i x | 2_74piox 1.1 | - | - | | |
| March Marc | | | | | | | | | | | | | |
| Company Comp | Backward (ICD10 to ICD9) | 0213088 | 02.13088 | 3616 | 36.16 | | | Coronary artery bypass surgery Px | 2_Approx 1:1 | 1 | 0 | 0 0 | 0 |
| 1996 | | | | | | | | | | | | | |
| Part | | | | | | | | | | | _ | | |
| Part | Backward (ICD10 to ICD9) | 0213089 | 02.13089 | 3616 | 36.16 | грргоден | Double internal mammary-coronary artery bypass | Coronary artery bypass surgery Px | 2_Approx 1:1 | 1 | 0 | 0 0 | 0 |
| State American (1976) 1,000 1,00 | | | | | | | | | | | | | |
| A PROPERTY REPORT OF THE PROPERTY AND A PROPERTY REPORT OF THE PROPERTY REPORT TO THE PROPERTY REPORT OF THE PROPERTY REPORT TO THE PROPERTY REPORT OF THE PROPERTY REPORT OF THE PROPERTY REPORT OF THE PROPERTY REPORT OF THE PROPERTY REPORT OF THE PROPE | Backward (ICD10 to ICD9) | 021308C | 02.1308C | 3616 | 36.16 | | Double internal mammary-coronary artery bypass | Coronary artery bypass surgery Px | 2 Approx 1:1 | 1 | 0 | 0 0 | 0 |
| Company Comp | | | | | | 1 | , | , | - 17 | | | | |
| Application Company | | | | | | | | | | | | | |
| According 1,000 | Backward (ICD10 to ICD9) | 021308F | 02.1308F | 3617 | 36.17 | Approach | Abdominal-coronary artery bypass | Coronary artery bypass surgery Px | 2_Approx 1:1 | 1 | 0 | 0 0 | 0 |
| April 1971 1972 | | | | | | | | | | | | | |
| Control of Control (1971) Control of Control (Control (Control of Control (Control (Control of Control (Control of Control (Control (Contr | Backward (ICD10 to ICD9) | 021308W | 02.1308W | 3614 | 36.14 | | (Aorto)coronary bypass of four or more coronary arter | Coronary artery bypass surgery Px | 2_Approx 1:1 | 1 | 0 | 0 0 | 0 |
| According Col. 1986 Col. | | | | | | | | | | | | | |
| Property | Rachward (ICD10 to ICD9) | 0213003 | 02 12002 | 3610 | 36.10 | | Other hypass anastomosis for heart revascularization | Coronary artery hypass surgery By | 2 Approx 1:1 | 1 | 0 | 0 | 0 |
| Secretary Control Co | Backward (ICD10 to ICD3) | 0213033 | 02.13033 | 3013 | 30.13 | The Process | Other bypass anastomosis for freat thevascularization | Coronary artery bypass surgery rx | 2_Approx 1.1 | | - | 0 | |
| According 1935 | | | | | | | | | | | | | |
| Page 1 1 1 1 1 1 1 1 1 | Backward (ICD10 to ICD9) | 0213098 | 02.13098 | 3616 | 36.16 | | Double internal mammary-coronary artery bypass | Coronary artery bypass surgery Px | 2 Approx 1:1 | 1 | 0 | 0 0 | 0 |
| Lett. tribers Lett. triber | | | | | | | , , , , | | | | | | |
| Page Company Prince | | | | | | | | | | | | | |
| Description Company Section Section Company Section | Backward (ICD10 to ICD9) | 0213099 | 02.13099 | 3616 | 36.16 | Tissue, Open Approach | Double internal mammary-coronary artery bypass | Coronary artery bypass surgery Px | 2_Approx 1:1 | 1 | 0 | 0 0 | 0 |
| Appendix | | | | | | | | | | | | | |
| Appendix Column Appe | | | | | | | | | | | _ | | _! |
| Address of ECRIT to 1 CRIT CRIT to 1 CRIT to 1 CRIT CRIT to 1 CRIT CRIT to 1 CRIT CRIT to 1 CRIT CRIT to 1 CRIT | Backward (ICD10 to ICD9) | 021309C | 02.1309C | 3616 | 36.16 | 11 | Double internal mammary-coronary artery bypass | Coronary artery bypass surgery Px | 2_Approx 1:1 | 1 | 0 | 0 0 | 0 |
| Part | Backward (ICD10 to ICD9) | 021309F | 02 1309F | 3617 | 36.17 | | Abdominal-coronary artery hypass | Coronary artery bypass surgery Py | 2 Approx 1:1 | 1 | 0 | 0 | 0 |
| Security (CO10 to CC0) CO11004 | Sackward (res to to ress) | 0213031 | 02.13031 | 5017 | 50.17 | Орентирически | y activity articly bypass | coronary artery bypass surgery i x | 2_7 ppi 0x 1:1 | - | - | | |
| Security (CO10 to CC0) CO11004 | | | | | | Bypass Coronary Artery, Four or More Arteries from | | | | | | | |
| Declared (CO10 to CO0) CO13004 CO13004 Sept. Sept. Consequent with Auditopops Anterior Stown, Owner Agreement of the System anadomous for heart reconcileration Owner Agreement of the System anad | Backward (ICD10 to ICD9) | 021309W | 02.1309W | 3614 | 36.14 | | (Aorto)coronary bypass of four or more coronary arte | Coronary artery bypass surgery Px | 2_Approx 1:1 | 1 | 0 | 0 0 | 0 |
| Decision (COD) Display | | | | | | Bypass Coronary Artery, Four or More Arteries from | | | | | | | |
| Pages Commany Afters Foundation Foun | | | | | | Coronary Artery with Autologous Arterial Tissue, | | | | | | | ļ |
| Reference Comment Co | Backward (ICD10 to ICD9) | 02130A3 | 02.130A3 | 3619 | 36.19 | | Other bypass anastomosis for heart revascularization | Coronary artery bypass surgery Px | 2_Approx 1:1 | 1 | 0 | 0 0 | 0 |
| Decision (COD) O211004 | | | | | | | | | | | | | |
| | Rackward (ICD10 to ICD0) | 0212049 | 02 12049 | 2616 | 26.16 | | Double internal mammary caronary artery hypars | Coronary artery bypace curgon, By | 3 Approx 1:1 | 1 | 0 | | |
| Lett internal Mammary virtue Autologous Arterial Tours (pen Agrosch 1) 10 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 | Backward (ICD10 to ICD9) | U213UA6 | U2.13UA6 | 3010 | 30.10 | | Double Internal mainmai y-coronal y artery bypass | Coronal y artery bypass surgery FX | 2_Approx 1.1 | | 0 | 0 0 | - 0 |
| Designate Company Co | | | | | | | | | | | | | ļ |
| Paginas Coronary Artery Four of More Arteries from Paginas Coronary Artery Four of More Arteries from Paginas Coronary Artery Four of More Arteries from Paginas Coronary Artery Four of More Arteries from Paginas Coronary Artery Paginas Surgery Px 2, Agenos 1: 1 0 0 0 0 | Backward (ICD10 to ICD9) | 02130A9 | 02.130A9 | 3616 | 36.16 | | Double internal mammary-coronary artery bypass | Coronary artery bypass surgery Px | 2_Approx 1:1 | 1 | 0 | 0 0 | 0 |
| | | | | | | Bypass Coronary Artery, Four or More Arteries from | | | | | | | |
| | | | | | | Thoracic Artery with Autologous Arterial Tissue, Oper | | | | | | | |
| Abdominal Action with Abdominal Active wit | Backward (ICD10 to ICD9) | 02130AC | 02.130AC | 3616 | 36.16 | 11 | Double internal mammary-coronary artery bypass | Coronary artery bypass surgery Px | 2_Approx 1:1 | 1 | 0 | 0 0 | 0 |
| Decision Color C | | | | | | | | | | | | | |
| Backward (CD10 to ICD9) | Rackward (ICD10 to ICD0) | 0212045 | 02.12045 | 2617 | 26 17 | | Abdominal coronary artery bypass | Coronary artery bypace curgon, By | 3 Approx 1:1 | 1 | 0 | | 0 |
| Active with Authorities Active (D10 to (CD9) 02130W | Backward (ICD10 to ICD9) | U213UAF | 02.130AF | 3017 | 30.17 | 1 | Abdominar-coronary artery bypass | Coronary artery bypass surgery FX | 2_Approx 1.1 | 1 | 0 | 0 0 | |
| Approach O2130AW O21 | | | | | | | | | | | | | |
| Spass Coronay Artery, Four or More Arteries from Coronay Artery by Substitute, Open Approach Spass Coronay Artery, Four or More Arteries from Right internal Mammary with Synthetic Substitute, Open Approach Spass Coronay Artery, Four or More Arteries from Left internal Mammary with Synthetic Substitute, Open Approach Spass Coronay Artery, Four or More Arteries from Left internal Mammary with Synthetic Substitute, Open Approach Spass Coronay Artery, Four or More Arteries from Left internal Mammary with Synthetic Substitute, Open Approach Spass Coronay Artery, Four or More Arteries from Left internal Mammary with Synthetic Substitute, Open Approach Spass Coronay Artery, Four or More Arteries from Left internal Mammary with Synthetic Substitute, Open Approach Spass Coronay Artery, Four or More Arteries from Location Coronary artery bypass surgery Px 2, Approx 1:1 1 0 0 0 0 0 0 0 0 | Backward (ICD10 to ICD9) | 02130AW | 02.130AW | 3614 | 36.14 | | (Aorto)coronary bypass of four or more coronary arter | Coronary artery bypass surgery Px | 2 Approx 1:1 | 1 | 0 | 0 0 | 0 |
| Coronary Artery with Synthetic Substitute, Open Sackward (ICD10 to ICD9) C213018 | · | | | | | Bypass Coronary Artery, Four or More Arteries from | | | | | | | |
| Suckward (ICD10 to ICD9) 0213018 02.13018 36.16 36.16 0 0 0 0 0 0 0 0 0 | | | | | | | | | | | | | |
| Section Company Comp | Backward (ICD10 to ICD9) | 02130J3 | 02.130J3 | 3619 | 36.19 | | Other bypass anastomosis for heart revascularization | Coronary artery bypass surgery Px | 2_Approx 1:1 | 1 | 0 | 0 0 | 0 |
| Double internal mammary-coronary artery bypass Coronary artery bypass Coronary artery bypass Coronary artery bypass Suggest Px 2, Approx 1:1 1 0 0 0 0 0 0 0 0 | | | | | | | | | | | | | |
| Bypass Coronary Artery, Four or More Arteries from Letternal Mammary with Synthetic Substitute, Open Approach Bypass Coronary Artery, Four or More Arteries from Thoracic Artery with Synthetic Substitute, Open Approach Bypass Coronary Artery, Four or More Arteries from Thoracic Artery with Synthetic Substitute, Open Approach Bypass Coronary Artery, Four or More Arteries from Abdominal Artery with Synthetic Substitute, Open Approach Bypass Coronary Artery, Four or More Arteries from Abdominal Artery with Synthetic Substitute, Open Approach Bypass Coronary Artery, Four or More Arteries from Abdominal Artery with Synthetic Substitute, Open Approach Bypass Coronary Artery, Four or More Arteries from Abdominal Artery with Synthetic Substitute, Open Approach Bypass Coronary Artery, Four or More Arteries from Abdominal Artery bypass Surgery Px Bypass Coronary Artery, Four or More Arteries from Abdomina | Bardonard (ICD104- ICD0) | 0242010 | 02.12010 | 2616 | 26.16 | | D | C | 2 41-1 | | | | |
| Left Internal Mammary with Synthetic Substitute, Open Approach Double internal mammary-coronary artery bypass Coronary artery bypass Surgery Px 2_Approx 1:1 1 0 0 0 0 0 0 0 0 | packwata (ICD10 to ICD3) | 0213038 | UZ.13UJ8 | 2010 | 50.16 | | Double Internal mammary-coronary artery bypass | Coronary artery bypass surgery Px | 2_Appr0X 1:1 | 1 | U | 0 | 0 |
| Jackward (ICD10 to ICD9) O2130/9 O2130/0 O2130/C O213 | | | | | 1 | | | | | | | | |
| Bypass Coronary Artery, Four or More Arteries from Thoracic Artery with Synthetic Substitute, Open Approach Bypass Coronary Artery, Four or More Arteries from Abdominal Artery with Synthetic Substitute, Open Approach Bypass Coronary Artery, Four or More Arteries from Abdominal Artery with Synthetic Substitute, Open Approach Bypass Coronary Artery bypass Surgery Px 2, Approx 1:1 1 0 0 0 0 0 0 0 0 0 0 0 0 | Backward (ICD10 to ICD9) | 0213019 | 02.130J9 | 3616 | 36.16 | | Double internal mammary-coronary artery bypass | Coronary artery bypass surgery Px | 2 Approx 1:1 | 1 | 0 | 0 0 | 0 |
| Thoracic Attery with Synthetic Substitute, Open Double internal mammary-coronary artery bypass Surgery Px 2, Approx 1:1 1 0 0 0 0 0 | , | | | | | 1 | ,,,, | , , | | | | 1 1 | |
| Sackward (ICD10 to ICD9) O2130/F O213 | | 1 1 | | | I | | | | | | | | |
| Sackward (ICD10 to ICD9) O2130JF O2.130JF O2.130JF O2.130JF O2.130JW O | Backward (ICD10 to ICD9) | 02130JC | 02.130JC | 3616 | 36.16 | | Double internal mammary-coronary artery bypass | Coronary artery bypass surgery Px | 2_Approx 1:1 | 1 | 0 | 0 0 | 0 |
| Approach | | | | | 1 | | | | | | | | |
| Sackward (ICD10 to ICD9) O2130JW O2.130JW O | | [] | | L | 1 | | | <u></u> | | | _ | | |
| Sackward (ICD10 to ICD9) 02130/W 02.130/W 3614 36.14 Acrta with Synthetic Substitute, Open Approach Acrta with Synthetic Substitute, Open Approach Acrta with Synthetic Substitute, Open Approach Acrta with Synthetic Substitute, Open Approach Synthetic Substitute, Open Approach Acrta with Synthetic Substitute, Open Approach Acrta with Synthetic Substitute, Open Approach Open Approach | Backward (ICD10 to ICD9) | 02130JF | 02.130JF | 3617 | 36.17 | | Abdominal-coronary artery bypass | Coronary artery bypass surgery Px | 2_Approx 1:1 | 1 | 0 | 0 0 | 0 |
| Bypass Coronary Artery, Four or More Arteries from Coronary Artery, Four or More Arteries from Coronary Artery, Four or More Arteries from Coronary Artery by Dass Surgery Px (2, Approx 1:1) 1 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 | Backward (ICD10 to ICD0) | 02420000 | 02 12004 | 2614 | 26.14 | | (Aarta)saranany hynass off | Coronary artony bypacs Pro | 3 Approvided | | 0 | | _ |
| Sackward (ICD10 to ICD9) O2130K3 O2.130K3 O2.130K8 O | packwala (ICD10 to ICD3) | 0213UJW | U2.13UJW | 3014 | 50.14 | | (nor to/coronary bypass or lour or more coronary arter | Coronary artery bypass surgery Px | 2_Appr 0X 1:1 | 1 | U | 0 | - 0 |
| Sackward (ICD10 to ICD9) 02130K3 02.130K3 3619 36.19 Substitute, Open Approach Other bypass anastomosis for heart revascularization Coronary artery bypass surgery PX 2_Approx 1:1 1 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 | | | | | 1 | | | | | | | | |
| Bypass Coronary Artery, Four or More Arteries from Right Internal Mammary with Nonautologous Tissue Sackward (ICD10 to ICD9) 02130K8 02.130K8 3616 36.16 Substitute, Open Approach Double internal mammary-coronary artery bypass Coronary Artery, bypass Surgery Px 2_Approx 1:1 1 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 | Backward (ICD10 to ICD9) | 02130K3 | 02.130K3 | 3619 | 36.19 | Substitute, Open Approach | Other bypass anastomosis for heart revascularization | Coronary artery bypass surgery Px | 2 Approx 1:1 | 1 | 0 | 0 0 | 0 |
| Right Internal Mammary with Nonautologous Tissue Sackward (ICD10 to ICD9) O2130K8 O2.130K8 O2.130KB O2 | | | | | | | | | | | | | |
| Sackward (ICD10 to ICD9) 02130K8 02.130K8 3616 36.16 Substitute, Open Approach Double internal mammary-coronary artery bypass Coronary artery bypass surgery PX 2_Approx 1:1 1 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 | | | | | 1 | Right Internal Mammary with Nonautologous Tissue | | | | | | | |
| Left Internal Mammary with Nonautologous Tissue | Backward (ICD10 to ICD9) | 02130K8 | 02.130K8 | 3616 | 36.16 | Substitute, Open Approach | Double internal mammary-coronary artery bypass | Coronary artery bypass surgery Px | 2_Approx 1:1 | 1 | 0 | 0 0 | 0 |
| | | 1 7 | | | 1 | | | | | | | | |
| ackward (ICD10 to ICD9) U2130K9 02.130K9 36.16 36.16 Substitute, Open Approach Double internal mammary-coronary artery bypass Coronary artery bypass surgery Px 2, Approx 1:1 1 0 0 0 0 0 | L | | | L | 1 - | | | <u></u> | | | _ | | J |
| | Backward (ICD10 to ICD9) | 02130K9 | 02.130K9 | 3616 | 36.16 | Substitute, Open Approach | Double internal mammary-coronary artery bypass | Coronary artery bypass surgery Px | 2_Approx 1:1 | 1 | U | 0 | 0 |




| | | | | | BEI | ORE MAT | CHING | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | OPTUM | 1 | | MARKETSCAN | | | MEDICARE | | | POOLED | |
| Variable | Reference - Sitagliptin | Exposure - Dapagliflozin | St. Diff | Reference - Sitagliptin | Exposure - Dapagliflozin | St. Diff | Reference - Sitagliptin | Exposure - Dapagliflozin | St. Diff | Reference -<br>Sitagliptin | Exposure -<br>Dapagliflozin | St. Diff |
| Number of patients | 21,224 | 871 | | 9,009 | 1,931 | | 51,898 | 2,701 | | 82,131 | 5,503 | |
| Age - Continuous mean (sd) | 73.04 (8.33) | 64.74 (10.17) | 0.8929 | 66.93 (11.32) | 59.00 (8.67) | 0.7865 | 76.27 (7.02) | 73.23 (6.25) | 0.4574 | 74.41 (7.95) | 66.89 (7.87) | 0.9507 |
| Age Categories | | | | | | | | | | | | |
| 18 - 54; n (%)<br>55 - 64; n (%) | 564 (2.7%)<br>1.973 (9.3%) | 155 (17.8%)<br>238 (27.3%) | -0.5140<br>-0.4787 | 1,146 (12.7%)<br>3.167 (35.2%) | 508 (26.3%)<br>1.093 (56.6%) | -0.3484<br>-0.4397 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1,710 (2.1%)<br>5,140 (6.3%) | 663 (12.0%)<br>1,331 (24.2%) | -0.3942<br>-0.5141 |
| 65 - 74: n (%) | 9,500 (44.8%) | 339 (38.9%) | 0.4787 | 2,238 (24.8%) | 241 (12.5%) | 0.3198 | 23,338 (45.0%) | 1,723 (63.8%) | -0.3844 | 32.838 (40.0%) | 2,062 (37.5%) | 0.0513 |
| > 75; n (%) | 9.187 (43.3%) | 139 (16.0%) | 0.6264 | 2,458 (27.3%) | 89 (4.6%) | 0.6521 | 28,560 (55.0%) | 978 (36.2%) | 0.3844 | 37,747 (46.0%) | 1,117 (20.3%) | 0.5675 |
| Gender | ., . , , | | | , , | | | .,, | | | | | |
| Male; n (%) | 10,060 (47.4%) | 487 (55.9%) | -0.1707 | 5,120 (56.8%) | 1,212 (62.8%) | -0.1226 | 24,233 (46.7%) | 1,385 (51.3%) | -0.0921 | 34,293 (41.8%) | 1,872 (34.0%) | 0.1613 |
| Female; n (%) | 11,164 (52.6%) | 384 (44.1%) | 0.1707 | 3,889 (43.2%) | 719 (37.2%) | 0.1226 | 27,665 (53.3%) | 1,316 (48.7%) | 0.0921 | 38,829 (47.3%) | 1,700 (30.9%) | 0.3409 |
| Geographic RegionNortheast: n (%) | 1.916 (9.0%) | 71 (8.2%) | 0.0285 | 1.605 (17.8%) | 214 (11.1%) | 0.1914 | 9.276 (17.9%) | 422 (15.6%) | 0.0616 | 11.192 (13.6%) | 493 (9.0%) | 0.1457 |
| Not theast, if (%) | 1,916 (9.0%) | 486 (55.8%) | -0.0823 | 4.157 (46.1%) | 1.168 (60.5%) | -0.2917 | 22.230 (42.8%) | 1.231 (45.6%) | -0.0564 | 33,205 (40.4%) | 1.717 (31.2%) | 0.1928 |
| Midwest; n (%) | 2.594 (12.2%) | 129 (14.8%) | -0.0761 | 2,159 (24.0%) | 288 (14.9%) | 0.2314 | 10.763 (20.7%) | 389 (14.4%) | 0.1662 | 13,357 (16.3%) | 518 (9.4%) | 0.2073 |
| West; n (%) | 5,730 (27.0%) | 185 (21.2%) | 0.1359 | 1,039 (11.5%) | 254 (13.2%) | -0.0517 | 9,502 (18.3%) | 655 (24.3%) | -0.1469 | 15,232 (18.5%) | 840 (15.3%) | 0.0855 |
| Unknown+missing; n (%) | 9 (0.0%) | 0 (0.0%) | #DIV/0! | 49 (0.5%) | 7 (0.4%) | 0.0149 | 127 (0.2%) | ** | - | 136 (0.2%) | | #VALUE! |
| Calendar Time - Year of Initiation (2014/15 - 2020) | | | | | | | | | | | | |
| 2014-2015; n (%) | 4,202 (19.8%) | 294 (33.8%) | -0.3201 | 3,943 (43.8%) | 576 (29.8%) | 0.2934 | 24,357 (46.9%) | 799 (29.6%) | 0.3617 | 28,559 (34.8%) | 1,093 (19.9%) | 0.3390 |
| 2016; n (%) | 2,845 (13.4%)<br>3,840 (18.1%) | 78 (9.0%)<br>135 (15.5%) | 0.1399 | 2,048 (22.7%)<br>1,743 (19.3%) | 473 (24.5%)<br>375 (19.4%) | -0.0424<br>-0.0025 | 13,886 (26.8%)<br>13,655 (26.3%) | 673 (24.9%)<br>1,229 (45.5%) | -0.4085 | 17,495 (21.3%) | 1,364 (24.8%) | -0.0832 |
| 2017, n (%) | 4.202 (19.8%) | 130 (14.9%) | 0.1297 | 1,743 (19.3%) | 507 (26.3%) | -0.3046 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 4,202 (5.1%) | 130 (2.4%) | 0.1425 |
| 2019 - March 2020; n (%) | 6,135 (28.9%) | 234 (26.9%) | 0.0446 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 6,135 (7.5%) | 234 (4.3%) | 0.1361 |
| Combined comorbidity score, 180 daysmean (sd) | 3.29 (2.46) | 2.52 (2.23) | 0.3280 | 2.30 (2.23) | 1.62 (1.81) | 0.3348 | 2.47 (2.48) | 2.02 (2.13) | 0.1947 | 2.66 (2.45) | 1.96 (2.04) | 0.3105 |
| Frailty Score: Empirical Version, 180 daysmean (sd) | 0.17 (0.05) | 0.16 (0.04) | 0.2209 | 0.16 (0.04) | 0.15 (0.03) | 0.2828 | 0.20 (0.06) | 0.19 (0.05) | 0.1811 | 0.19 (0.06) | 0.17 (0.04) | 0.3922 |
| DiabRen - CKD II; n (%) | 3,872 (18.2%) | 191 (21.9%) | -0.0925 | 1,306 (14.5%) | 391 (20.2%) | -0.1510 | 6,955 (13.4%) | 497 (18.4%) | -0.1371 | 10,827 (13.2%) | 688 (12.5%) | 0.0209 |
| DiabRen - CKD III; n (%) | 11,801 (55.6%) | 359 (41.2%) | 0.2912 | 4,193 (46.5%) | 563 (29.2%) | 0.3625 | 27,504 (53.0%) | 1,109 (41.1%) | 0.2401 | 39,305 (47.9%) | 1,468 (26.7%) | 0.4493 |
| DiabRen - Occurrence of Diabetic Nephropathy ; n (%) | 11,450 (53.9%) | 398 (45.7%) | 0.1646 | 3,050 (33.9%) | 669 (34.6%) | -0.0148 | 16,224 (31.3%) | 906 (33.5%) | -0.0470 | 27,674 (33.7%) | 1,304 (23.7%) | 0.2224 |
| DiabRen - Occurrence of Diabetic Neuropathy ; n (%) DiabRen - Diabetic retinopathy : n (%) | 6,254 (29.5%)<br>2,260 (10.6%) | 253 (29.0%)<br>95 (10.9%) | 0.0110<br>-0.0097 | 1,659 (18.4%)<br>577 (6.4%) | 392 (20.3%)<br>113 (5.9%) | -0.0481<br>0.0208 | 13,517 (26.0%)<br>4.571 (8.8%) | 847 (31.4%)<br>327 (12.1%) | -0.1196<br>-0.1080 | 19,771 (24.1%)<br>6.831 (8.3%) | 1,100 (20.0%)<br>422 (7.7%) | 0.0990 |
| DiabRen - Diabetic foot : n (%) | 713 (3.4%) | 27 (3.1%) | 0.0169 | 274 (3.0%) | 52 (2.7%) | 0.0180 | 2.084 (4.0%) | 94 (3.5%) | 0.0263 | 2,797 (3.4%) | 121 (2.2%) | 0.0728 |
| DiabRen - Diabetes with peripheral circulatory disorders ; n (%) | 3,190 (15.0%) | 90 (10.3%) | 0.1417 | 617 (6.8%) | 95 (4.9%) | 0.0810 | 5,924 (11.4%) | 343 (12.7%) | -0.0399 | 9,114 (11.1%) | 433 (7.9%) | 0.1093 |
| DiabRen - Hypertensive nephropathy; n (%) | 6,719 (31.7%) | 227 (26.1%) | 0.1238 | 1,940 (21.5%) | 363 (18.8%) | 0.0673 | 8,934 (17.2%) | 477 (17.7%) | -0.0132 | 15,653 (19.1%) | 704 (12.8%) | 0.1727 |
| DiabRen - Hypertension ; n (%) | 19,413 (91.5%) | 786 (90.2%) | 0.0451 | 7,700 (85.5%) | 1,635 (84.7%) | 0.0225 | 48,556 (93.6%) | 2,539 (94.0%) | -0.0166 | 67,969 (82.8%) | 3,325 (60.4%) | 0.5128 |
| DiabRen - Hypotension ; n (%) DiabRen - Gout (acute/chronic) : n (%) | 616 (2.9%)<br>430 (2.0%) | 20 (2.3%)<br>15 (1.7%) | 0.0377 | 181 (2.0%)<br>237 (2.6%) | 28 (1.5%)<br>43 (2.2%) | 0.0381 | 1,813 (3.5%)<br>1,334 (2.6%) | 72 (2.7%)<br>44 (1.6%) | 0.0462 | 2,429 (3.0%)<br>1,764 (2.1%) | 092 (1.7%)<br>059 (1.1%) | 0.0859 |
| DiabRen - Gout (acute/chronic); n (%) DiabRen - Nephrolithiasis: n (%) | 430 (2.0%)<br>362 (1.7%) | 15 (1.7%) | -0.0223 | 237 (2.6%) | 43 (2.2%)<br>35 (1.8%) | 0.0261 | 1,334 (2.6%) | 44 (1.6%) | 0.0098 | 1,499 (1.8%) | 066 (1.2%) | 0.0798 |
| DiabRen - Proteinuria: n (%) | 1,863 (8.8%) | 80 (9.2%) | -0.0140 | 328 (3.6%) | 44 (2.3%) | 0.0769 | 4.437 (8.5%) | 253 (9.4%) | -0.0315 | 6,300 (7.7%) | 333 (6.1%) | 0.0632 |
| DiabRen - Urinary tract infections (UTIs); n (%) | 2,823 (13.3%) | 80 (9.2%) | 0.1300 | 705 (7.8%) | 95 (4.9%) | 0.1191 | 9,351 (18.0%) | 408 (15.1%) | 0.0781 | 12,174 (14.8%) | 488 (8.9%) | 0.1833 |
| DiabRen - Genital infections; n (%) | 302 (1.4%) | 9 (1.0%) | 0.0367 | 123 (1.4%) | 28 (1.5%) | -0.0084 | 800 (1.5%) | 47 (1.7%) | -0.0159 | 1,102 (1.3%) | 056 (1.0%) | 0.0281 |
| DiabRen - Hypoglycemia v2 ; n (%) | 3,543 (16.7%) | 121 (13.9%) | 0.0778 | 651 (7.2%) | 175 (9.1%) | -0.0695 | 4,291 (8.3%) | 292 (10.8%) | -0.0851 | 7,834 (9.5%) | 413 (7.5%) | 0.0718 |
| DiabRen - Hyperglycemia; n (%) DiabRen - Hyperkalemia: n (%) | 1,039 (4.9%)<br>975 (4.6%) | 32 (3.7%)<br>33 (3.8%) | 0.0592 | 311 (3.5%)<br>312 (3.5%) | 70 (3.6%)<br>41 (2.1%) | -0.0054<br>0.0849 | 2,817 (5.4%)<br>2,589 (5.0%) | 148 (5.5%)<br>87 (3.2%) | -0.0044 | 3,856 (4.7%)<br>3,564 (4.3%) | 180 (3.3%)<br>120 (2.2%) | 0.0715 |
| DiabRen - Hyperkalemia; n (%) DiabRen - Hypovolemia/volume depletion; n (%) | 834 (3.9%) | 28 (3.2%) | 0.0339 | 263 (2.9%) | 44 (2.3%) | 0.0377 | 2,569 (5.0%) | 90 (3.3%) | 0.0853 | 3,403 (4.1%) | 118 (2.1%) | 0.1156 |
| NephroTox - ACE inhibitors ; n (%) | 11,816 (55.7%) | 458 (52.6%) | 0.0622 | 4,903 (54.4%) | 1,056 (54.7%) | -0.0060 | 28,838 (55.6%) | 1,361 (50.4%) | 0.1043 | 40,654 (49.5%) | 1,819 (33.1%) | 0.3378 |
| NephroTox - ARBs ; n (%) | 10,050 (47.4%) | 451 (51.8%) | -0.0881 | 4,429 (49.2%) | 956 (49.5%) | -0.0060 | 24,917 (48.0%) | 1,439 (53.3%) | -0.1062 | 34,967 (42.6%) | 1,890 (34.3%) | 0.1712 |
| NephroTox - Loop Diuretics ; n (%) | 4,691 (22.1%) | 166 (19.1%) | 0.0742 | 1,928 (21.4%) | 272 (14.1%) | 0.1919 | 15,531 (29.9%) | 647 (24.0%) | 0.1333 | 20,222 (24.6%) | 813 (14.8%) | 0.2483 |
| NephroTox - Thiazide diuretics ; n (%) | 4,144 (19.5%) | 165 (18.9%) | 0.0152 | 1,823 (20.2%) | 333 (17.2%) | 0.0770 | 10,001 (19.3%) | 484 (17.9%) | 0.0360 | 14,145 (17.2%) | 649 (11.8%) | 0.1538 |
| NephroTox - Mineralocorticoid receptor antagonist ; n (%) | 1,024 (4.8%) | 50 (5.7%) | -0.0404 | 590 (6.5%) | 97 (5.0%) | 0.0645 | 2,969 (5.7%) | 128 (4.7%) | 0.0451 | 3,993 (4.9%) | 178 (3.2%) | 0.0863 |
| NephroTox - NSAIDs; n (%) NephroTox - PPIs: n (%) | 2,651 (12.5%)<br>5.417 (25.5%) | 140 (16.1%)<br>201 (23.1%) | -0.1030<br>0.0560 | 1,182 (13.1%)<br>1.895 (21.0%) | 339 (17.6%)<br>380 (19.7%) | -0.1251<br>0.0323 | 5,826 (11.2%)<br>14.510 (28.0%) | 427 (15.8%)<br>688 (25.5%) | -0.1349<br>0.0565 | 8,477 (10.3%)<br>19.927 (24.3%) | 567 (10.3%)<br>889 (16.2%) | 0.0000 |
| NephroTox - PPIs; n (%) NeohroTox - H2RAs: n (%) | 5,417 (25.5%) | 201 (23.1%)<br>40 (4.6%) | 0.0560 | 1,895 (21.0%)<br>377 (4.2%) | 380 (19.7%)<br>67 (3.5%) | 0.0323 | 14,510 (28.0%)<br>3,801 (7.3%) | 688 (25.5%)<br>217 (8.0%) | -0.0263 | 5,423 (6.6%) | 257 (4.7%) | 0.2026 |
| NephroTox - Antivirals/Antiretrovirals/Antimicrobials; n (%) | 200 (0.9%) | 14 (1.6%) | -0.0630 | 85 (0.9%) | 19 (1.0%) | -0.0103 | 517 (1.0%) | 33 (1.2%) | -0.0192 | 717 (0.9%) | 047 (0.9%) | 0.0000 |
| DM Medications - 1st and 2nd Generation SUs ; n (%) | 9,808 (46.2%) | 380 (43.6%) | 0.0523 | 3,893 (43.2%) | 708 (36.7%) | 0.1330 | 24,534 (47.3%) | 1,180 (43.7%) | 0.0723 | 34,342 (41.8%) | 1,560 (28.3%) | 0.2858 |
| DM Medications - AGI & Meglinitides; n (%) | 487 (2.3%) | 17 (2.0%) | 0.0207 | 246 (2.7%) | 35 (1.8%) | 0.0607 | 1,767 (3.4%) | 136 (5.0%) | -0.0798 | 2,254 (2.7%) | 153 (2.8%) | -0.0061 |
| DM Medications - DPP-4 Inhibitors (excluding sitagliptin); n (%) | 1,253 (5.9%) | 134 (15.4%) | -0.3117 | 675 (7.5%) | 172 (8.9%) | -0.0510 | 4,025 (7.8%) | 426 (15.8%) | -0.2499 | 5,278 (6.4%) | 560 (10.2%) | -0.1381 |
| DM Medications - Glitazones ; n (%) DM Medications - Gl P-1 RA · n (%) | 1,969 (9.3%)<br>888 (4.2%) | 106 (12.2%)<br>228 (26.2%) | -0.0937<br>-0.6437 | 771 (8.6%)<br>469 (5.2%) | 242 (12.5%) | -0.1272<br>-0.6143 | 4,266 (8.2%) | 320 (11.8%) | -0.1202<br>-0.5360 | 6,235 (7.6%)<br>2,407 (2.9%) | 426 (7.7%)<br>743 (13.5%) | -0.0038 |
| DM Medications - GLP-1 RA ; n (%) DM Medications - Insulins: n (%) | 4,954 (23.3%) | 228 (26.2%) | -0.6437 | 469 (5.2%)<br>1,997 (22.2%) | 515 (26.7%)<br>633 (32.8%) | -0.6143 | 1,519 (2.9%) | 515 (19.1%)<br>1,005 (37.2%) | -0.5360 | 17,245 (21.0%) | 1,296 (23.6%) | -0.3938 |
| DM Medications - Insulins; in (%) DM Medications - Metformin ; n (%) | 11,179 (52.7%) | 529 (60.7%) | -0.2233 | 4,464 (49.6%) | 1,188 (61.5%) | -0.2331 | 24,769 (47.7%) | 1,510 (55.9%) | -0.2960 | 35,948 (43.8%) | 2,039 (37.1%) | 0.1368 |
| DM Medications - SGLT-2 Inhibitors (excluding dapagliflozin); n (%) | 443 (2.1%) | 60 (6.9%) | -0.2331 | 181 (2.0%) | 269 (13.9%) | -0.4509 | 473 (0.9%) | 181 (6.7%) | -0.3069 | 916 (1.1%) | 241 (4.4%) | -0.2028 |
| DM Medications - Number of antiDM medications at index datemean (sd) | 2.28 (0.84) | 2.84 (0.97) | -0.6172 | 2.25 (0.84) | 2.82 (0.99) | -0.6209 | ** | ** | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| CV Comorbidity - Acute and Old MI ; n (%) | 1,054 (5.0%) | 29 (3.3%) | 0.0853 | 215 (2.4%) | 27 (1.4%) | 0.0733 | 3,147 (6.1%) | 127 (4.7%) | 0.0620 | 4,201 (5.1%) | 156 (2.8%) | 0.1183 |
| CV Comorbidity - Any Heart failure (HF); n (%) | 3,264 (15.4%) | 90 (10.3%) | 0.1528 | 923 (10.2%) | 98 (5.1%) | 0.1928 | 10,227 (19.7%) | 389 (14.4%) | 0.1413 | 13,491 (16.4%) | 479 (8.7%) | 0.2340 |
| CV Comorbidity - Hospitalization for CHF; n (%) CV Comorbidity - Atrial fibrillation; n (%) | 715 (3.4%) | 23 (2.6%) | 0.0469<br>0.1505 | 315 (3.5%)<br>802 (8.9%) | 25 (1.3%)<br>82 (4.2%) | 0.1441 | 3,249 (6.3%)<br>8,791 (16.9%) | 79 (2.9%)<br>355 (13.1%) | 0.1628 | 3,964 (4.8%)<br>11,280 (13.7%) | 102 (1.9%)<br>419 (7.6%) | 0.1617 |
| CV Comorbidity - Atrial fibrillation; n (%) CV Comorbidity - Other dysrythmias ; n (%) | 2,489 (11.7%)<br>3,047 (14.4%) | 64 (7.3%)<br>109 (12.5%) | 0.1505 | 802 (8.9%)<br>948 (10.5%) | 82 (4.2%)<br>124 (6.4%) | 0.1908 | 8,791 (16.9%)<br>8,990 (17.3%) | 355 (13.1%)<br>422 (15.6%) | 0.1066 | 11,280 (13.7%) | 419 (7.6%)<br>531 (9.6%) | 0.1987 |
| CV Comorbidity - Other dysrytnimas ; n (%) CV Comorbidity - Valve disorder ; n (%) | 720 (3.4%) | 17 (2.0%) | 0.0337 | 168 (1.9%) | 20 (1.0%) | 0.0753 | 2.387 (4.6%) | 98 (3.6%) | 0.0504 | 3,107 (3.8%) | 115 (2.1%) | 0.1006 |
| CV Comorbidity - Implantable cardioverter defibrillator ; n (%) | 416 (2.0%) | 10 (1.1%) | 0.0729 | 156 (1.7%) | 12 (0.6%) | 0.1033 | 1,521 (2.9%) | 49 (1.8%) | 0.0727 | 1,937 (2.4%) | 059 (1.1%) | 0.0993 |
| CV Comorbidity - CABG/PCI ; n (%) | 1,691 (8.0%) | 60 (6.9%) | 0.0419 | 305 (3.4%) | 46 (2.4%) | 0.0596 | 5,727 (11.0%) | 268 (9.9%) | 0.0360 | 7,418 (9.0%) | 328 (6.0%) | 0.1141 |
| CV Comorbidity - Coronary atherosclerosis and other forms of chronic ischemic heart disease ; n (%) | 5,339 (25.2%) | 199 (22.8%) | 0.0562 | 1,914 (21.2%) | 295 (15.3%) | 0.1532 | 18,111 (34.9%) | 895 (33.1%) | 0.0380 | 23,450 (28.6%) | 1,094 (19.9%) | 0.2040 |

| | 16.913 (79.7%) | | -0.0955 | | 1.483 (76.8%) | -0.1456 | | 2.257 (83.6%) | -0.0732 | 58,868 (71.7%) | 2,983 (54.2%) | 0.000 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CV Comorbidity - Hyperlipidemia ; n (%) CV Comorbidity - Stable Angina : n (%) | 16,913 (79.7%) | 726 (83.4%)<br>33 (3.8%) | 0.0955 | 6,345 (70.4%)<br>216 (2.4%) | 1,483 (76.8%) | 0.0133 | 41,955 (80.8%)<br>1,933 (3.7%) | 2,257 (83.6%) | -0.0732 | 3.165 (3.9%) | 2,983 (54.2%)<br>170 (3.1%) | 0.3685 |
| CV Comorbidity - Stable Angina ; n (%) CV Comorbidity - Unstable Angina ; n (%) | 1,232 (5.8%)<br>331 (1.6%) | 33 (3.8%)<br>18 (2.1%) | -0.0371 | 216 (2.4%)<br>93 (1.0%) | 42 (2.2%)<br>15 (0.8%) | 0.0133 | 1,933 (3.7%)<br>846 (1.6%) | 137 (5.1%)<br>38 (1.4%) | 0.0165 | 1,177 (1.4%) | 056 (1.0%) | 0.0435 |
| CV Comorbidity - Oristable Alighta , It (%) CV Comorbidity - Peripheral Vascular Disease (PVD) or PVD Surgery ; n (%) | 2.604 (12.3%) | 91 (10.4%) | 0.0599 | 651 (7.2%) | 77 (4.0%) | 0.1395 | 8,166 (15.7%) | 421 (15.6%) | 0.0028 | 10,770 (13.1%) | 512 (9.3%) | 0.1207 |
| CV Comorbidity - Peripheral vascular Disease (PVD) of PVD surgery, It (%) | 927 (4.4%) | 25 (2.9%) | 0.0801 | 183 (2.0%) | 19 (1.0%) | 0.0823 | 2.043 (3.9%) | 84 (3.1%) | 0.0435 | 2,970 (3.6%) | 109 (2.0%) | 0.0973 |
| CV Comorbidity - Pulmonary hypertension/Other pulmonary heart disease; n (%) | 637 (3.0%) | 19 (2.2%) | 0.0503 | 179 (2.0%) | 18 (0.9%) | 0.0921 | 1,876 (3.6%) | 64 (2.4%) | 0.0704 | 2,513 (3.1%) | 083 (1.5%) | 0.1069 |
| , | 001 (01071) | (=:=,:) | | 2.0 (2.0,1.) | ( | | 2,010 (01011) | J - (Z) | | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | , | |
| CV Medication - Beta blockers; n (%) | 10,748 (50.6%) | 438 (50.3%) | 0.0060 | 4,664 (51.8%) | 823 (42.6%) | 0.1851 | 29,658 (57.1%) | 1,486 (55.0%) | 0.0423 | 40,406 (49.2%) | 1,924 (35.0%) | 0.2906 |
| CV Medication - CCB; n (%) | 8,243 (38.8%) | 274 (31.5%) | 0.1533 | 3,256 (36.1%) | 544 (28.2%) | 0.1698 | 20,572 (39.6%) | 987 (36.5%) | 0.0639 | 28,815 (35.1%) | 1,261 (22.9%) | 0.2713 |
| CV Medication - Digoxin; n (%) | 473 (2.2%) | 15 (1.7%) | 0.0362 | 198 (2.2%) | 17 (0.9%) | 0.1054 | 2,016 (3.9%) | 87 (3.2%) | 0.0378 | 2,489 (3.0%) | 102 (1.9%) | 0.0712 |
| CV Medication - Nitrates; n (%) | 1,651 (7.8%) | 74 (8.5%) | -0.0256 | 564 (6.3%) | 74 (3.8%) | 0.1144 | 5,317 (10.2%) | 255 (9.4%) | 0.0269 | 6,968 (8.5%) | 329 (6.0%) | 0.0965 |
| CV Medication - Use of Statins ; n (%) | 17,126 (80.7%) | 717 (82.3%) | -0.0412 | 6,804 (75.5%) | 1,470 (76.1%) | -0.0140 | 40,441 (77.9%) | 2,195 (81.3%) | -0.0844 | 57,567 (70.1%) | 2,912 (52.9%) | 0.3591 |
| CV Medication - Use of other lipid-lowering drugs ; n (%) | 2,741 (12.9%) | 161 (18.5%) | -0.1544 | 1,615 (17.9%) | 398 (20.6%) | -0.0685 | 8,062 (15.5%) | 497 (18.4%) | -0.0774 | 10,803 (13.2%) | 658 (12.0%) | 0.0362 |
| CV Medication - Use of other hypertension drugs; n (%) | 2,587 (12.2%) | 82 (9.4%) | 0.0903 | 1,156 (12.8%) | 181 (9.4%) | 0.1084 | 6,811 (13.1%) | 350 (13.0%) | 0.0030 | 9,398 (11.4%) | 432 (7.9%) | 0.1187 |
| | | | 4 | | | | | | | | | |
| Other Comorbidity - Anemia ; n (%) | 4,602 (21.7%) | 131 (15.0%) | 0.1737 | 1,550 (17.2%) | 240 (12.4%) | 0.1355 | 16,274 (31.4%) | 720 (26.7%) | 0.1037 | 20,876 (25.4%) | 851 (15.5%) | 0.2473 |
| Other Comorbidity - Cancer ; n (%) | 2,602 (12.3%)<br>2,845 (13.4%) | 93 (10.7%) | 0.0502<br>0.1059 | 1,053 (11.7%)<br>667 (7.4%) | 128 (6.6%)<br>60 (3.1%) | 0.1776<br>0.1937 | 8,190 (15.8%)<br>7.771 (15.0%) | 345 (12.8%)<br>364 (13.5%) | 0.0858 | 10,792 (13.1%)<br>10.616 (12.9%) | 438 (8.0%)<br>451 (8.2%) | 0.1534 |
| Other Comorbidity - COPD ; n (%) Other Comorbidity - Dementia : n (%) | 2,845 (13.4%) | 87 (10.0%)<br>28 (3.2%) | 0.1059 | 314 (3.5%) | 9 (0.5%) | 0.1937 | 7,771 (15.0%)<br>5.494 (10.6%) | 167 (6.2%) | 0.0429 | 6.947 (8.5%) | 451 (8.2%)<br>195 (3.5%) | 0.1534 |
| Other Comorbidity - Dementia ; n (%) Other Comorbidity - Depression ; n (%) | 3.072 (14.5%) | 28 (3.2%)<br>104 (11.9%) | 0.0769 | 701 (7.8%) | 9 (0.5%) | 0.0267 | 5,494 (10.6%)<br>6.957 (13.4%) | 350 (13.0%) | 0.0118 | 10,029 (12.2%) | 454 (8.3%) | 0.1289 |
| Other Comorbidity - Fractures ; n (%) | 772 (3.6%) | 24 (2.8%) | 0.0455 | 284 (3.2%) | 36 (1.9%) | 0.0825 | 2.685 (5.2%) | 101 (3.7%) | 0.0728 | 3.457 (4.2%) | 125 (2.3%) | 0.1073 |
| Other Comorbidity - Fractures ; n (%) Other Comorbidity - Hypothyroidism ; n (%) | 1,505 (7.1%) | 74 (8.5%) | -0.0522 | 711 (7.9%) | 152 (7.9%) | 0.0000 | 7,204 (13.9%) | 330 (12.2%) | 0.0728 | 8.709 (10.6%) | 404 (7.3%) | 0.1075 |
| Other Comorbidity - Pypothyroidism , II (%) | 1,618 (7.6%) | 47 (5.4%) | 0.0893 | 282 (3.1%) | 29 (1.5%) | 0.1069 | 4.961 (9.6%) | 304 (11.3%) | -0.0556 | 6,579 (8.0%) | 351 (6.4%) | 0.0619 |
| Other Comorbidity - Pneumonia ; n (%) | 825 (3.9%) | 21 (2.4%) | 0.0860 | 315 (3.5%) | 28 (1.5%) | 0.1284 | 2,793 (5.4%) | 96 (3.6%) | 0.0869 | 3,618 (4.4%) | 117 (2.1%) | 0.1300 |
| Other Comorbidity - Sleep apnea ; n (%) | 2,555 (12.0%) | 148 (17.0%) | -0.1424 | 1,255 (13.9%) | 329 (17.0%) | -0.0859 | 5,931 (11.4%) | 400 (14.8%) | -0.1009 | 8,486 (10.3%) | 548 (10.0%) | 0.0099 |
| | | | | | | | -,, | , | | | | |
| Other Medication - Use of anticonvulsants ; n (%) | 4,685 (22.1%) | 187 (21.5%) | 0.0145 | 1,476 (16.4%) | 312 (16.2%) | 0.0054 | 11,018 (21.2%) | 708 (26.2%) | -0.1178 | 15,703 (19.1%) | 895 (16.3%) | 0.0734 |
| Other Medication - Use of antidepressants ; n (%) | 5,538 (26.1%) | 228 (26.2%) | -0.0023 | 2,124 (23.6%) | 451 (23.4%) | 0.0047 | 14,254 (27.5%) | 799 (29.6%) | -0.0465 | 19,792 (24.1%) | 1,027 (18.7%) | 0.1320 |
| Other Medication - Use of antiparkinsonian meds ; n (%) | 668 (3.1%) | 25 (2.9%) | 0.0117 | 229 (2.5%) | 40 (2.1%) | 0.0267 | 2,031 (3.9%) | 118 (4.4%) | -0.0251 | 2,699 (3.3%) | 143 (2.6%) | 0.0414 |
| Other Medication - Use of dementia meds ; n (%) | 924 (4.4%) | 16 (1.8%) | 0.1504 | 217 (2.4%) | 3 (0.2%) | 0.1951 | 3,463 (6.7%) | 133 (4.9%) | 0.0771 | 4,387 (5.3%) | 149 (2.7%) | 0.1330 |
| Other Medication - Use of antipsychotics ; n (%) | 672 (3.2%) | 24 (2.8%) | 0.0235 | 200 (2.2%) | 25 (1.3%) | 0.0687 | 2,140 (4.1%) | 93 (3.4%) | 0.0369 | 2,812 (3.4%) | 117 (2.1%) | 0.0796 |
| Other Medication - Use of anxiolytics/hypnotics ; n (%) | 1,093 (5.1%) | 55 (6.3%) | -0.0518 | 534 (5.9%) | 130 (6.7%) | -0.0329 | 3,233 (6.2%) | 204 (7.6%) | -0.0553 | 4,326 (5.3%) | 259 (4.7%) | 0.0275 |
| Other Medication - Use of Benzodiazepines ; n (%) | 2,322 (10.9%) | 100 (11.5%) | -0.0190 | 920 (10.2%) | 197 (10.2%) | 0.0000 | 6,616 (12.7%) | 344 (12.7%) | 0.0000 | 8,938 (10.9%) | 444 (8.1%) | 0.0956 |
| Other Medication - Use of COPD/asthma meds; n (%) | 4,164 (19.6%) | 175 (20.1%) | -0.0125<br>0.0444 | 1,578 (17.5%) | 310 (16.1%) | 0.0375 | 10,663 (20.5%) | 601 (22.3%) | -0.0439 | 14,827 (18.1%) | 776 (14.1%) | 0.1090 |
| Other Medication - Use of antiplatelet agents; n (%) | 2,950 (13.9%) | 108 (12.4%) | 0.0444 | 1,478 (16.4%) | 271 (14.0%) | 0.0669<br>0.1720 | 8,311 (16.0%) | 447 (16.5%) | -0.0136<br>0.0295 | 11,261 (13.7%) | 555 (10.1%)<br>418 (7.6%) | 0.1114 |
| Other Medication - Use of oral anticoagulants ; n (%) Other Medication - Use of opioids : n (%) | 2,259 (10.6%)<br>5,237 (24.7%) | 72 (8.3%)<br>194 (22.3%) | 0.0566 | 875 (9.7%)<br>2,318 (25.7%) | 101 (5.2%)<br>461 (23.9%) | 0.1720 | 7,187 (13.8%)<br>14,731 (28.4%) | 346 (12.8%)<br>737 (27.3%) | 0.0295 | 9,446 (11.5%)<br>19,968 (24.3%) | 931 (16.9%) | 0.1330 |
| Other Medication - Use of opioids ; n (%) | 5,237 (24.7%) | 194 (22.3%) | 0.0566 | 2,318 (25.7%) | 461 (23.9%) | 0.0417 | 14,/31 (28.4%) | /3/(2/.3%) | 0.0245 | 19,968 (24.3%) | 931 (10.9%) | 0.1837 |
| Lifestyle - Alcohol/Drug Abuse or Dependence ; n (%) | 616 (2.9%) | 16 (1.8%) | 0.0727 | 110 (1.2%) | 18 (0.9%) | 0.0294 | 870 (1.7%) | 45 (1.7%) | 0.0000 | 1.486 (1.8%) | 061 (1.1%) | 0.0586 |
| Lifestyle - Obesity; n (%) | 4,620 (21.8%) | 273 (31.3%) | -0.2164 | 1,702 (18.9%) | 481 (24.9%) | -0.1455 | 10,685 (20.6%) | 795 (29.4%) | -0.2043 | 15,305 (18.6%) | 1,068 (19.4%) | -0.0204 |
| Lifestyle - Smoking; n (%) | 2,862 (13.5%) | 94 (10.8%) | 0.0827 | 508 (5.6%) | 93 (4.8%) | 0.0360 | 8,159 (15.7%) | 395 (14.6%) | 0.0307 | 11,021 (13.4%) | 489 (8.9%) | 0.1433 |
| HU - Number of Cardiologist visitsmean (sd) | 1.78 (4.22) | 1.67 (4.25) | 0.0260 | 1.10 (3.36) | 0.88 (2.46) | 0.0747 | 2.45 (5.55) | 2.07 (5.07) | 0.0715 | 2.13 (5.03) | 1.59 (4.20) | 0.1165 |
| HU - Number of Nephrologist visitmean (sd) | 0.60 (2.24) | 0.48 (1.72) | 0.0601 | 0.49 (1.99) | 0.38 (1.68) | 0.0597 | 0.74 (2.77) | 0.69 (3.95) | 0.0147 | 0.68 (2.57) | 0.55 (3.02) | 0.0464 |
| HU - Number of Endocrinologist visitsmean (sd) | 0.45 (2.10) | 1.18 (3.73) | -0.2412 | 0.49 (2.28) | 0.98 (2.96) | -0.1855 | 0.79 (3.61) | 1.32 (4.52) | -0.1296 | 0.67 (3.15) | 1.18 (3.91) | -0.1436 |
| HU - Number of Internal Medicine/Family Medicine Visitsmean (sd) | 15.91 (18.92) | 11.70 (15.83) | 0.2413 | 9.07 (12.72) | 7.67 (8.79) | 0.1281 | 10.09 (12.96) | 10.75 (14.87) | -0.0473<br>0.1146 | 11.48 (14.71)<br>0.66 (1.90) | 9.82 (13.24)<br>0.42 (1.50) | 0.1186 |
| HU - Number of Emergency Department (ED) visitsmean (sd) | 0.59 (1.60) | 0.52 (1.83) | | 0.27 (1.51) | 0.00 (0.00) | | 0.75 (2.06) | 0.55 (1.36) | | | | |
| HU - Number of Distinct Medication Prescriptions (not generalized to generics)mean (sd) HU - Number of Echocardiogrammean (sd) | 28.51 (19.80)<br>0.28 (1.42) | 33.44 (20.23)<br>0.30 (1.55) | -0.2463<br>-0.0135 | 25.94 (16.29)<br>0.22 (0.69) | 27.51 (16.84)<br>0.13 (0.46) | -0.0948<br>0.1535 | 31.26 (22.25)<br>0.28 (0.70) | 36.01 (26.11)<br>0.23 (0.65) | -0.1958<br>0.0740 | 29.97 (21.05)<br>0.27 (0.94) | 32.62 (22.34)<br>0.21 (0.81) | 0.0684 |
| | 0.83 (1.83) | | | 0.22 (0.69) | 0.13 (0.46) | | | | | | | |
| HU - Number of Electrocardiogram Performedmean (sd) HU - Number of HbAIc tests orderedmean (sd) | 0.03 (1.03) | | 0.0438 | 0.68/1.43\ | 0.47/1.00) | 0.1702 | 0.00 (1.00) | | | | | 0.1209 |
| | 1 50 (0 97) | 0.75 (1.82) | -0.0213 | 0.68 (1.43) | 0.47 (1.00) | 0.1702<br>-0.4455 | 0.98 (1.80) | 0.85 (1.58) | 0.0768 | 0.91 (1.77) | 0.70 (1.45) | -0.1152 |
| HU - Number of Hospitalizations during CAPmean (sd) | 1.50 (0.97)<br>0.15 (0.50) | 1.52 (0.91) | 0.0438<br>-0.0213<br>0.0637 | 0.96 (0.98) | 1.39 (0.95) | 0.1702<br>-0.4455<br>0.1576 | 1.53 (0.93) | 0.85 (1.58)<br>1.72 (0.98) | | | | 0.1298<br>-0.1152<br>0.1984 |
| HU - Number of Hospitalizations during CAPmean (sd) HU - Recent hospitalization (-30 days to Index Rx date) : n (%) | 1.50 (0.97)<br>0.15 (0.50)<br>617 (2.9%) | | -0.0213<br>0.0637 | | | -0.4455<br>0.1576 | | 0.85 (1.58) | 0.0768<br>-0.1989<br>0.2162 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59) | 0.70 (1.45)<br>1.57 (0.96)<br>0.11 (0.40) | -0.1152<br>0.1984 |
| HU - Recent hospitalization (-30 days to Index Rx date); n (%) | 0.15 (0.50) | 1.52 (0.91)<br>0.12 (0.44) | -0.0213 | 0.96 (0.98)<br>0.14 (0.44) | 1.39 (0.95)<br>0.08 (0.31) | -0.4455 | 1.53 (0.93)<br>0.25 (0.65)<br>2,465 (4.7%) | 0.85 (1.58)<br>1.72 (0.98)<br>0.13 (0.44) | 0.0768<br>-0.1989 | 0.91 (1.77)<br>1.46 (0.95) | 0.70 (1.45)<br>1.57 (0.96) | -0.1152 |
| HU - Recent hospitalization (-30 days to Index Rx date); n (%) HU - Old hospitalizations (-180 to -31 days); n (%) | 0.15 (0.50)<br>617 (2.9%)<br>2,008 (9.5%) | 1.52 (0.91)<br>0.12 (0.44)<br>13 (1.5%)<br>76 (8.7%) | -0.0213<br>0.0637<br>0.0956 | 0.96 (0.98)<br>0.14 (0.44)<br>254 (2.8%)<br>841 (9.3%) | 1.39 (0.95)<br>0.08 (0.31)<br>18 (0.9%)<br>110 (5.7%) | -0.4455<br>0.1576<br>0.1414 | 1.53 (0.93)<br>0.25 (0.65)<br>2,465 (4.7%)<br>7,233 (13.9%) | 0.85 (1.58)<br>1.72 (0.98)<br>0.13 (0.44)<br>36 (1.3%)<br>245 (9.1%) | 0.0768<br>-0.1989<br>0.2162<br>0.2003 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%) | 0.70 (1.45)<br>1.57 (0.96)<br>0.11 (0.40)<br>049 (0.9%) | -0.1152<br>0.1984<br>0.1923 |
| HU - Recent hospitalization (-30 days to Index Rx date); n (%) | 0.15 (0.50)<br>617 (2.9%) | 1.52 (0.91)<br>0.12 (0.44)<br>13 (1.5%) | -0.0213<br>0.0637<br>0.0956<br>0.0278 | 0.96 (0.98)<br>0.14 (0.44)<br>254 (2.8%) | 1.39 (0.95)<br>0.08 (0.31)<br>18 (0.9%) | -0.4455<br>0.1576<br>0.1414<br>0.1370 | 1.53 (0.93)<br>0.25 (0.65)<br>2,465 (4.7%) | 0.85 (1.58)<br>1.72 (0.98)<br>0.13 (0.44)<br>36 (1.3%) | 0.0768<br>-0.1989<br>0.2162<br>0.2003<br>0.1509 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%)<br>9,241 (11.3%) | 0.70 (1.45)<br>1.57 (0.96)<br>0.11 (0.40)<br>049 (0.9%)<br>321 (5.8%) | -0.1152<br>0.1984<br>0.1923<br>0.1977 |
| HU - Recent hospitalization (-30 days to Index Rx date); n (%) HU - Old hospitalizations (-180 to -31 days); n (%) HU - Mammogram ; n (%) | 0.15 (0.50)<br>617 (2.9%)<br>2,008 (9.5%)<br>2,561 (12.1%) | 1.52 (0.91)<br>0.12 (0.44)<br>13 (1.5%)<br>76 (8.7%)<br>108 (12.4%) | -0.0213<br>0.0637<br>0.0956<br>0.0278<br>-0.0092 | 0.96 (0.98)<br>0.14 (0.44)<br>254 (2.8%)<br>841 (9.3%)<br>754 (8.4%) | 1.39 (0.95)<br>0.08 (0.31)<br>18 (0.9%)<br>110 (5.7%)<br>181 (9.4%) | -0.4455<br>0.1576<br>0.1414<br>0.1370<br>-0.0351 | 1.53 (0.93)<br>0.25 (0.65)<br>2,465 (4.7%)<br>7,233 (13.9%)<br>5,207 (10.0%) | 0.85 (1.58)<br>1.72 (0.98)<br>0.13 (0.44)<br>36 (1.3%)<br>245 (9.1%)<br>293 (10.8%) | 0.0768<br>-0.1989<br>0.2162<br>0.2003<br>0.1509<br>-0.0262 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%)<br>9,241 (11.3%)<br>7,768 (9.5%) | 0.70 (1.45)<br>1.57 (0.96)<br>0.11 (0.40)<br>049 (0.9%)<br>321 (5.8%)<br>401 (7.3%) | -0.1152<br>0.1984<br>0.1923<br>0.1977<br>0.0794 |
| HU - Recent hospitalization (-30 days to Index Rx date); n (%) HU - Old hospitalizations (-180 to -31 days); n (%) HU - Mammogram; n (%) HU - Pap smear; n (%) | 0.15 (0.50)<br>617 (2.9%)<br>2,008 (9.5%)<br>2,561 (12.1%)<br>380 (1.8%) | 1.52 (0.91)<br>0.12 (0.44)<br>13 (1.5%)<br>76 (8.7%)<br>108 (12.4%)<br>19 (2.2%) | -0.0213<br>0.0637<br>0.0956<br>0.0278<br>-0.0092<br>-0.0286<br>0.0144<br>0.0446 | 0.96 (0.98)<br>0.14 (0.44)<br>254 (2.8%)<br>841 (9.3%)<br>754 (8.4%)<br>261 (2.9%) | 1.39 (0.95)<br>0.08 (0.31)<br>18 (0.9%)<br>110 (5.7%)<br>181 (9.4%)<br>84 (4.4%) | -0.4455<br>0.1576<br>0.1414<br>0.1370<br>-0.0351<br>-0.0801<br>-0.0558<br>0.0044 | 1.53 (0.93)<br>0.25 (0.65)<br>2,465 (4.7%)<br>7,233 (13.9%)<br>5,207 (10.0%)<br>916 (1.8%) | 0.85 (1.58)<br>1.72 (0.98)<br>0.13 (0.44)<br>36 (1.3%)<br>245 (9.1%)<br>293 (10.8%)<br>47 (1.7%) | 0.0768<br>-0.1989<br>0.2162<br>0.2003<br>0.1509<br>-0.0262<br>0.0076<br>-0.0679<br>-0.0093 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%)<br>9,241 (11.3%)<br>7,768 (9.5%)<br>1,296 (1.6%)<br>3,671 (4.5%)<br>3,501 (4.3%) | 0.70 (1.45)<br>1.57 (0.96)<br>0.11 (0.40)<br>049 (0.9%)<br>321 (5.8%)<br>401 (7.3%)<br>066 (1.2%)<br>220 (4.0%)<br>167 (3.0%) | -0.1152<br>0.1984<br>0.1923<br>0.1977<br>0.0794<br>0.0341<br>0.0248<br>0.0694 |
| HU - Recent hospitalization (-30 days to Index Rx date); n (%) HU - Old hospitalizations (-180 to -31 days); n (%) HU - Mammogram; n (%) HU - Pap smear; n (%) HU - Prostate exam for DRE; n (%) HU - Floxible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%) HU - Bone mineral density; n (%) | 0.15 (0.50)<br>617 (2.9%)<br>2,008 (9.5%)<br>2,561 (12.1%)<br>380 (1.8%)<br>1,007 (4.7%)<br>987 (4.7%)<br>1,026 (4.8%) | 1.52 (0.91)<br>0.12 (0.44)<br>13 (1.5%)<br>76 (8.7%)<br>108 (12.4%)<br>19 (2.2%)<br>38 (4.4%)<br>33 (3.8%)<br>38 (4.4%) | -0.0213<br>0.0637<br>0.0956<br>0.0278<br>-0.0092<br>-0.0286<br>0.0144<br>0.0446<br>0.0191 | 0.96 (0.98)<br>0.14 (0.44)<br>254 (2.8%)<br>841 (9.3%)<br>754 (8.4%)<br>261 (2.9%)<br>315 (3.5%)<br>497 (5.5%)<br>196 (2.2%) | 1.39 (0.95)<br>0.08 (0.31)<br>18 (0.9%)<br>110 (5.7%)<br>181 (9.4%)<br>84 (4.4%)<br>88 (4.6%)<br>104 (5.4%)<br>39 (2.0%) | -0.4455<br>0.1576<br>0.1414<br>0.1370<br>-0.0351<br>-0.0801<br>-0.0558<br>0.0044<br>0.0139 | 1.53 (0.93)<br>0.25 (0.65)<br>2,465 (4.7%)<br>7,233 (13.9%)<br>5,207 (10.0%)<br>916 (1.8%)<br>2,664 (5.1%)<br>2,514 (4.8%)<br>2,214 (4.3%) | 0.85 (1.58)<br>1.72 (0.98)<br>0.13 (0.44)<br>36 (1.3%)<br>245 (9.1%)<br>293 (10.8%)<br>47 (1.7%)<br>182 (6.7%)<br>134 (5.0%)<br>133 (4.9%) | 0.0768<br>-0.1989<br>0.2162<br>0.2003<br>0.1509<br>-0.0262<br>0.0076<br>-0.0679<br>-0.093<br>-0.0286 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%)<br>9,241 (11.3%)<br>7,768 (9.5%)<br>1,296 (1.6%)<br>3,671 (4.5%)<br>3,501 (4.3%)<br>3,240 (3.9%) | 0.70 (1.45)<br>1.57 (0.96)<br>0.11 (0.40)<br>049 (0.9%)<br>321 (5.8%)<br>401 (7.3%)<br>066 (1.2%)<br>220 (4.0%)<br>167 (3.0%)<br>171 (3.1%) | -0.1152<br>0.1984<br>0.1923<br>0.1977<br>0.0794<br>0.0341<br>0.0248<br>0.0694 |
| HU - Recent hospitalization (-30 days to index Rx date); n (%) HU - Old hospitalizations (-180 to -31 days); n (%) HU - Mammogram; n (%) HU - Pap smear; n (%) HU - Prostate exam for DRE; n (%) HU - Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%) HU - Bloome mineral density; n (%) HU - Hu vaccine; n (%) | 0.15 (0.50)<br>617 (2.9%)<br>2,008 (9.5%)<br>2,561 (12.1%)<br>380 (1.8%)<br>1,007 (4.7%)<br>987 (4.7%)<br>1,026 (4.8%)<br>4,955 (23.3%) | 1.52 (0.91)<br>0.12 (0.44)<br>13 (1.5%)<br>76 (8.7%)<br>108 (12.4%)<br>19 (2.2%)<br>38 (4.4%)<br>33 (3.8%)<br>38 (4.4%)<br>197 (22.6%) | -0.0213<br>0.0637<br>0.0956<br>0.0278<br>-0.0092<br>-0.0286<br>0.0144<br>0.0446<br>0.0191<br>0.0166 | 0.96 (0.98)<br>0.14 (0.44)<br>254 (2.8%)<br>841 (9.3%)<br>754 (8.4%)<br>261 (2.9%)<br>315 (3.5%)<br>497 (5.5%)<br>196 (2.2%)<br>1,562 (17.3%) | 1.39 (0.95)<br>0.08 (0.31)<br>18 (0.9%)<br>110 (5.7%)<br>181 (9.4%)<br>84 (4.4%)<br>88 (4.6%)<br>104 (5.4%)<br>39 (2.0%)<br>355 (18.4%) | -0.4455<br>0.1576<br>0.1414<br>0.1370<br>-0.0351<br>-0.0801<br>-0.0558<br>0.0044<br>0.0139<br>-0.0287 | 1.53 (0.93)<br>0.25 (0.65)<br>2,465 (4.7%)<br>7,233 (13.9%)<br>5,207 (10.0%)<br>916 (1.8%)<br>2,664 (5.1%)<br>2,514 (4.8%)<br>2,214 (4.3%)<br>18,258 (35.2%) | 0.85 (1.58)<br>1.72 (0.98)<br>0.13 (0.44)<br>36 (1.3%)<br>245 (9.1%)<br>293 (10.8%)<br>47 (1.7%)<br>182 (6.7%)<br>134 (5.0%)<br>133 (4.9%)<br>935 (34.6%) | 0.0768 -0.1989 0.2162 0.2003 0.1509 -0.0262 0.0076 -0.0679 -0.093 -0.0286 0.0126 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%)<br>9,241 (11.3%)<br>7,768 (9.5%)<br>1,296 (1.6%)<br>3,671 (4.5%)<br>3,501 (4.3%)<br>3,240 (3.9%)<br>23,213 (28.3%) | 0.70 (1.45)<br>1.57 (0.96)<br>0.11 (0.40)<br>049 (0.9%)<br>321 (5.8%)<br>401 (7.3%)<br>066 (1.2%)<br>220 (4.0%)<br>167 (3.0%)<br>171 (3.1%)<br>1,132 (20.6%) | 0.1152<br>0.1984<br>0.1923<br>0.1977<br>0.0794<br>0.0341<br>0.0248<br>0.0694<br>0.0435 |
| HU - Recent hospitalization (-30 days to Index Rx date); n (%) HU - Old hospitalizations (-180 to -31 days); n (%) HU - Mammogram; n (%) HU - Pap smear; n (%) HU - Prostate exam for DRE; n (%) HU - Floxible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%) HU - Bone mineral density; n (%) | 0.15 (0.50)<br>617 (2.9%)<br>2,008 (9.5%)<br>2,561 (12.1%)<br>380 (1.8%)<br>1,007 (4.7%)<br>987 (4.7%)<br>1,026 (4.8%) | 1.52 (0.91)<br>0.12 (0.44)<br>13 (1.5%)<br>76 (8.7%)<br>108 (12.4%)<br>19 (2.2%)<br>38 (4.4%)<br>33 (3.8%)<br>38 (4.4%) | -0.0213<br>0.0637<br>0.0956<br>0.0278<br>-0.0092<br>-0.0286<br>0.0144<br>0.0446<br>0.0191 | 0.96 (0.98)<br>0.14 (0.44)<br>254 (2.8%)<br>841 (9.3%)<br>754 (8.4%)<br>261 (2.9%)<br>315 (3.5%)<br>497 (5.5%)<br>196 (2.2%) | 1.39 (0.95)<br>0.08 (0.31)<br>18 (0.9%)<br>110 (5.7%)<br>181 (9.4%)<br>84 (4.4%)<br>88 (4.6%)<br>104 (5.4%)<br>39 (2.0%) | -0.4455<br>0.1576<br>0.1414<br>0.1370<br>-0.0351<br>-0.0801<br>-0.0558<br>0.0044<br>0.0139 | 1.53 (0.93)<br>0.25 (0.65)<br>2,465 (4.7%)<br>7,233 (13.9%)<br>5,207 (10.0%)<br>916 (1.8%)<br>2,664 (5.1%)<br>2,514 (4.8%)<br>2,214 (4.3%) | 0.85 (1.58)<br>1.72 (0.98)<br>0.13 (0.44)<br>36 (1.3%)<br>245 (9.1%)<br>293 (10.8%)<br>47 (1.7%)<br>182 (6.7%)<br>134 (5.0%)<br>133 (4.9%) | 0.0768<br>-0.1989<br>0.2162<br>0.2003<br>0.1509<br>-0.0262<br>0.0076<br>-0.0679<br>-0.093<br>-0.0286 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%)<br>9,241 (11.3%)<br>7,768 (9.5%)<br>1,296 (1.6%)<br>3,671 (4.5%)<br>3,501 (4.3%)<br>3,240 (3.9%) | 0.70 (1.45)<br>1.57 (0.96)<br>0.11 (0.40)<br>049 (0.9%)<br>321 (5.8%)<br>401 (7.3%)<br>066 (1.2%)<br>220 (4.0%)<br>167 (3.0%)<br>171 (3.1%) | -0.1152<br>0.1984<br>0.1923<br>0.1977<br>0.0794<br>0.0341<br>0.0248<br>0.0694 |
| HU - Recent hospitalization (-30 days to Index Rx date); n (%) HU - Old hospitalizations (-180 to -31 days); n (%) HU - Hu - Mammogram; n (%) HU - Pap smear; n (%) HU - Prostate exam for DRE; n (%) HU - Flexible Eigenioidoscopy or colonoscopy or CT virtual colonoscopy; n (%) HU - Bone mineral density; n (%) HU - Flu vaccine; n (%) HU - Pneumococcal vaccine; n (%) | 0.15 (0.50)<br>617 (2.9%)<br>2,008 (9.5%)<br>2,561 (12.1%)<br>380 (1.8%)<br>1,007 (4.7%)<br>987 (4.7%)<br>1,026 (4.8%)<br>4,955 (23.3%)<br>5,388 (25.4%) | 1.52 (0.91)<br>0.12 (0.44)<br>13 (1.5%)<br>76 (8.7%)<br>108 (12.4%)<br>19 (2.2%)<br>38 (4.4%)<br>33 (3.8%)<br>36 (4.4%)<br>197 (22.6%) | -0.0213<br>0.0637<br>0.0956<br>0.0278<br>-0.0092<br>-0.0286<br>0.0144<br>0.0446<br>0.0191<br>0.0166<br>0.0680 | 0.96 (0.98)<br>0.14 (0.44)<br>254 (2.8%)<br>841 (9.3%)<br>754 (8.4%)<br>261 (2.9%)<br>315 (3.5%)<br>497 (5.5%)<br>196 (2.2%)<br>1,562 (17.3%)<br>1,246 (13.8%) | 1.39 (0.95)<br>0.08 (0.31)<br>1.8 (0.9%)<br>1.10 (5.7%)<br>1.81 (9.4%)<br>8.84 (4.4%)<br>8.84 (4.5%)<br>1.04 (5.4%)<br>3.92 (2.0%)<br>3.55 (18.4%)<br>2.89 (15.0%) | -0.4455<br>0.1576<br>0.1414<br>0.1370<br>-0.0351<br>-0.0801<br>-0.0558<br>0.0044<br>0.0139<br>-0.0287<br>-0.0342 | 1.53 (0.93)<br>0.25 (0.65)<br>2,465 (4.7%)<br>7,233 (13.9%)<br>5,207 (10.0%)<br>916 (1.8%)<br>2,664 (5.1%)<br>2,514 (4.8%)<br>2,514 (4.3%)<br>18,258 (35.2%)<br>14,318 (27.6%) | 0.85 (1.58)<br>1.72 (0.98)<br>0.13 (0.44)<br>36 (1.3%)<br>245 (9.1%)<br>293 (10.8%)<br>47 (1.7%)<br>132 (5.0%)<br>133 (5.0%)<br>935 (34.6%)<br>856 (31.7%) | 0.0768<br>-0.1989<br>0.2162<br>0.2003<br>0.1509<br>-0.0262<br>0.0076<br>-0.0679<br>-0.0286<br>0.0126<br>-0.0899 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%)<br>9,241 (11.3%)<br>7,768 (9.5%)<br>1,296 (1.6%)<br>3,671 (4.5%)<br>3,671 (4.3%)<br>3,240 (3.9%)<br>23,213 (28.3%)<br>19,706 (24.0%) | 0.70 (1.45)<br>1.57 (0.96)<br>0.11 (0.40)<br>0.49 (0.9%)<br>321 (5.8%)<br>401 (7.3%)<br>066 (1.2%)<br>220 (4.0%)<br>167 (3.0%)<br>171 (3.1%)<br>1,132 (20.6%)<br>1,052 (19.1%) | 0.1152<br>0.1984<br>0.1923<br>0.1977<br>0.0794<br>0.0341<br>0.0248<br>0.0694<br>0.0435<br>0.1799 |
| HU - Recent hospitalization (-30 days to index Rx date); n (%) HU - Old hospitalizations (-180 to -31 days); n (%) HU - Mammogram; n (%) HU - Pap smear; n (%) HU - Prostate exam for DRE; n (%) HU - Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%) HU - Bloome mineral density; n (%) HU - Hu vaccine; n (%) | 0.15 (0.50)<br>617 (2.9%)<br>2,008 (9.5%)<br>2,08 (9.5%)<br>2,561 (12.1%)<br>380 (1.8%)<br>1,007 (4.7%)<br>987 (4.7%)<br>4,955 (23.3%)<br>5,388 (25.4%)<br>8,939 (42.1%) | 1.52 (0.91)<br>0.12 (0.44)<br>13 (1.5%)<br>76 (8.7%)<br>108 (12.4%)<br>19 (2.2%)<br>38 (4.4%)<br>38 (4.4%)<br>38 (4.4%)<br>197 (2.6%)<br>196 (22.5%) | -0.0213<br>0.0637<br>0.0956<br>0.0278<br>-0.0092<br>-0.0286<br>0.0144<br>0.0191<br>0.0166<br>0.0680 | 0.96 (0.98)<br>0.14 (0.44)<br>254 (2.8%)<br>841 (9.3%)<br>754 (8.4%)<br>261 (2.9%)<br>315 (3.5%)<br>497 (5.5%)<br>196 (2.2%)<br>1,562 (17.3%)<br>1,246 (13.8%)<br>2,455 (27.3%) | 1.39 (0.95)<br>0.08 (0.31)<br>18 (0.9%)<br>110 (5.7%)<br>181 (9.4%)<br>84 (4.4%)<br>88 (4.6%)<br>104 (5.4%)<br>39 (2.0%)<br>355 (18.4%)<br>289 (15.0%) | -0.4455<br>0.1576<br>0.1414<br>0.1370<br>-0.0351<br>-0.0801<br>-0.0558<br>0.0044<br>0.0139<br>-0.0287<br>-0.0342 | 1.53 (0.93)<br>0.25 (0.65)<br>2,465 (4.7%)<br>7,233 (13.9%)<br>5,207 (10.9%)<br>916 (1.8%)<br>2,664 (5.1%)<br>2,514 (4.8%)<br>2,214 (4.3%)<br>18,258 (35.2%)<br>14,318 (27.6%) | 0.85 (1.58)<br>1.72 (0.98)<br>0.13 (0.44)<br>36 (1.3%)<br>245 (9.1%)<br>293 (10.8%)<br>47 (1.7%)<br>132 (6.7%)<br>134 (5.0%)<br>133 (4.9%)<br>935 (34.6%)<br>856 (31.7%) | 0.0768 -0.1989 0.2162 0.2003 0.1509 -0.0262 0.0076 -0.0679 -0.0093 -0.0286 0.0126 -0.0899 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%)<br>9,241 (11.3%)<br>7,768 (9.5%)<br>1,296 (1.6%)<br>3,671 (4.5%)<br>3,501 (4.3%)<br>3,240 (3.9%)<br>23,213 (28.3%)<br>19,706 (24.0%) | 0.70 (1.45)<br>1.57 (0.96)<br>0.11 (0.40)<br>0.49 (0.9%)<br>321 (5.8%)<br>401 (7.3%)<br>066 (1.2%)<br>220 (4.0%)<br>167 (3.0%)<br>171 (3.1%)<br>1,132 (20.6%)<br>1,052 (19.1%) | 0.1152<br>0.1984<br>0.1923<br>0.1977<br>0.0794<br>0.0341<br>0.0248<br>0.0694<br>0.1799<br>0.1194 |
| HU - Recent hospitalization (-30 days to index Rx date); n (%) HU - Old hospitalizations (-180 to -31 days); n (%) HU - Hammorgam; n (%) HU - Pap smear; n (%) HU - Prostate exam for DRE; n (%) HU - Frostate exam for DRE; n (%) HU - Brostate exam for DRE; n (%) HU - Brostate exam for DRE; n (%) HU - Flow and the state of | 0.15 (0.50)<br>617 (2.9%)<br>2,008 (9.5%)<br>2,561 (12.1%)<br>380 (1.8%)<br>1,007 (4.7%)<br>987 (4.7%)<br>1,026 (4.8%)<br>4,955 (2.3%)<br>5,388 (25.4%)<br>1,202 (5.7%) | 1.52 (0.91)<br>0.12 (0.44)<br>13 (1.5%)<br>76 (8.7%)<br>108 (12.4%)<br>13 (4.4%)<br>38 (4.4%)<br>38 (4.4%)<br>38 (4.4%)<br>197 (22.6%)<br>196 (22.5%)<br>370 (42.5%)<br>53 (6.1%) | -0.0213<br>0.0637<br>0.0956<br>0.0278<br>-0.0092<br>-0.0286<br>0.0144<br>0.0191<br>0.0166<br>0.0680 | 0.96 (0.98)<br>0.14 (0.44)<br>254 (2.8%)<br>841 (9.3%)<br>754 (8.8%)<br>261 (2.9%)<br>315 (3.5%)<br>497 (5.5%)<br>196 (2.2%)<br>1,562 (17.3%)<br>1,246 (13.8%)<br>2,455 (27.3%)<br>466 (5.2%) | 1.39 (0.95)<br>0.08 (0.31)<br>18 (0.9%)<br>110 (5.7%)<br>181 (9.4%)<br>84 (4.4%)<br>88 (4.6%)<br>104 (5.4%)<br>39 (2.0%)<br>355 (18.4%)<br>289 (15.0%)<br>755 (39.1%)<br>80 (4.1%) | -0.4455<br>0.1576<br>0.1414<br>0.1370<br>-0.0351<br>-0.0801<br>-0.0558<br>0.0044<br>0.0139<br>-0.0287<br>-0.0342<br>-0.2526<br>0.0523 | 1.53 (0.93)<br>0.25 (0.65)<br>2.465 (4.7%)<br>7.233 (13.9%)<br>5.207 (10.9%)<br>916 (1.8%)<br>2.664 (5.1%)<br>2.514 (4.8%)<br>2.214 (4.3%)<br>18,258 (35.2%)<br>14,318 (27.6%)<br>19,220 (37.0%)<br>4,261 (8.2%) | 0.85 (1.58)<br>1.72 (0.98)<br>0.13 (0.44)<br>36 (1.3%)<br>245 (9.1%)<br>293 (10.8%)<br>47 (1.7%)<br>182 (6.7%)<br>133 (4.9%)<br>935 (34.6%)<br>856 (31.7%)<br>1,105 (40.9%)<br>195 (7.2%) | 0.0768 -0.1989 0.2162 0.2003 0.1509 -0.0262 0.0076 -0.0679 -0.093 -0.0286 0.0126 -0.0899 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%)<br>9,241 (11.3%)<br>7,768 (9.5%)<br>1,296 (1.6%)<br>3,671 (4.5%)<br>3,501 (4.3%)<br>3,240 (3.9%)<br>23,213 (28.3%)<br>19,706 (24.0%) | 0.70 (1.45)<br>1.57 (0.96)<br>0.31 (0.40)<br>049 (0.9%)<br>321 (5.8%)<br>401 (7.3%)<br>066 (1.2%)<br>167 (3.0%)<br>171 (3.1%)<br>1,132 (0.6%)<br>1,052 (19.1%)<br>1,475 (26.8%)<br>248 (4.5%) | 0.115;<br>0.1984<br>0.1923<br>0.1977<br>0.0794<br>0.0341<br>0.0248<br>0.0694<br>0.1799<br>0.1194<br>0.1634<br>0.0958 |
| HU - Recent hospitalization (-30 days to Index Rx date); n (%) HU - Old hospitalizations (-180 to -31 days); n (%) HU - Mammogram; n (%) HU - Pap smear; n (%) HU - Prostate exam for DRE; n (%) HU - Firestate exam for DRE; n (%) HU - Hostate exam for DRE; n (%) HU - Hostate exam for DRE; n (%) HU - House exam for DRE; n (%) HU - House exam for DRE; n (%) HU - House exam for DRE; n (%) Lab - Occurrence of creatinine tests ordered; n (%) Lab - Occurrence of creatinine tests ordered; n (%) | 0.15 (0.50)<br>617 (2.9%)<br>2,008 (9.5%)<br>2,088 (9.5%)<br>2,561 (12.11%)<br>380 (1.8%)<br>1,007 (4.7%)<br>987 (4.7%)<br>1,026 (4.8%)<br>4,955 (23.3%)<br>5,388 (25.4%)<br>8,939 (42.1%)<br>1,202 (5.7%)<br>11,639 (54.8%) | 1.52 (0.91)<br>0.12 (0.44)<br>13 (1.5%)<br>76 (8.7%)<br>108 (12.4%)<br>15 (2.2%)<br>38 (4.4%)<br>33 (3.8%)<br>36 (4.4%)<br>197 (22.6%)<br>196 (22.5%)<br>370 (42.5%)<br>370 (42.5%)<br>467 (53.6%) | 0.0213<br>0.0637<br>0.0956<br>0.0278<br>-0.0092<br>-0.0286<br>0.0144<br>0.0446<br>0.0191<br>0.0166<br>0.0680 | 0.96 (0.98)<br>0.14 (0.44)<br>254 (2.8%)<br>841 (9.3%)<br>754 (8.4%)<br>261 (2.9%)<br>315 (3.5%)<br>497 (5.5%)<br>196 (2.2%)<br>1,562 (17.3%)<br>1,246 (13.8%)<br>2,455 (27.3%)<br>466 (5.2%)<br>2,651 (29.0%) | 1.39 (0.95)<br>0.08 (0.31)<br>1.8 (0.9%)<br>1.10 (5.7%)<br>1.81 (9.4%)<br>8.84 (4.4%)<br>8.84 (4.5%)<br>3.92 (2.0%)<br>3.55 (1.8.4%)<br>2.89 (1.5.0%)<br>7.55 (3.9.1%)<br>8.04 (4.1%)<br>8.04 (4.1%) | -0.4455<br>0.1576<br>0.1414<br>0.1370<br>-0.0351<br>-0.0801<br>-0.0558<br>0.0044<br>0.0139<br>-0.0287<br>-0.0342<br>-0.2526<br>0.0523<br>-0.3278 | 1.53 (0.93) 0.25 (0.65) 2,465 (4.7%) 7,233 (13.9%) 5,207 (10.0%) 916 (1.8%) 2,664 (5.1%) 2,514 (4.3%) 2,214 (4.3%) 18,258 (35.2%) 14,318 (27.6%) 19,220 (37.0%) 4,261 (8.2%) 2,150 (14.4%) | 0.85 (1.58)<br>1.72 (0.98)<br>0.13 (0.44)<br>36 (1.3%)<br>245 (9.1%)<br>293 (10.8%)<br>47 (1.7%)<br>182 (6.7%)<br>134 (5.0%)<br>133 (4.9%)<br>935 (34.6%)<br>856 (31.7%)<br>1.105 (40.9%)<br>1.105 (40.9%) | 0.0768 -0.1989 0.2162 0.2003 0.1509 -0.0262 0.0076 -0.0679 -0.0286 0.0126 -0.0899 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%)<br>9,241 (11.3%)<br>7,768 (9.5%)<br>1,296 (1.6%)<br>3,671 (4.5%)<br>3,501 (4.3%)<br>3,240 (3.9%)<br>23,213 (28.3%)<br>19,706 (24.0%)<br>5,463 (6.7%)<br>3,3139 (40.3%) | 0.70 (1.45)<br>1.57 (0.96)<br>0.11 (0.40)<br>0.49 (0.9%)<br>321 (5.8%)<br>401 (7.3%)<br>066 (1.2%)<br>220 (4.0%)<br>167 (3.0%)<br>171 (3.1%)<br>1,132 (20.6%)<br>1,052 (19.1%)<br>1,475 (26.8%)<br>1,475 (26.8%)<br>1,744 (31.7%) | 0.1152<br>0.1984<br>0.1923<br>0.1977<br>0.0794<br>0.0344<br>0.0248<br>0.0694<br>0.0433<br>0.1795<br>0.1194 |
| HU - Recent hospitalization (-30 days to Index Rx date); n (%) HU - Old hospitalizations (-180 to -31 days); n (%) HU - Hu - Mammong m; n (%) HU - Pap smear; n (%) HU - Prostate exam for DRE; n (%) HU - Frostate exam for DRE; n (%) HU - Brostate exam for DRE; n (%) HU - Frostate exam for DRE; n (%) HU - Frostate exam for DRE; n (%) HU - Frostate exam for DRE; n (%) HU - Frostate exam for DRE; n (%) Lob - Occurrence of 24-hour urine test; n (%) Lob - Occurrence of creatinine tests ordered; n (%) | 0.15 (0.50)<br>617 (2.9%)<br>2,008 (9.5%)<br>2,561 (12.1%)<br>380 (1.8%)<br>1,007 (4.7%)<br>987 (4.7%)<br>1,026 (4.8%)<br>4,955 (2.3%)<br>5,388 (25.4%)<br>1,202 (5.7%) | 1.52 (0.91)<br>0.12 (0.44)<br>13 (1.5%)<br>76 (8.7%)<br>108 (12.4%)<br>13 (4.4%)<br>38 (4.4%)<br>38 (4.4%)<br>38 (4.4%)<br>197 (22.6%)<br>196 (22.5%)<br>370 (42.5%)<br>53 (6.1%) | -0.0213<br>0.0637<br>0.0956<br>0.0278<br>-0.0092<br>-0.0286<br>0.0144<br>0.0191<br>0.0166<br>0.0680 | 0.96 (0.98)<br>0.14 (0.44)<br>254 (2.8%)<br>841 (9.3%)<br>754 (8.8%)<br>261 (2.9%)<br>315 (3.5%)<br>497 (5.5%)<br>196 (2.2%)<br>1,562 (17.3%)<br>1,246 (13.8%)<br>2,455 (27.3%)<br>466 (5.2%) | 1.39 (0.95)<br>0.08 (0.31)<br>18 (0.9%)<br>110 (5.7%)<br>181 (9.4%)<br>84 (4.4%)<br>88 (4.6%)<br>104 (5.4%)<br>39 (2.0%)<br>355 (18.4%)<br>289 (15.0%)<br>755 (39.1%)<br>80 (4.1%) | -0.4455<br>0.1576<br>0.1414<br>0.1370<br>-0.0351<br>-0.0801<br>-0.0558<br>0.0044<br>0.0139<br>-0.0287<br>-0.0342<br>-0.2526<br>0.0523 | 1.53 (0.93)<br>0.25 (0.65)<br>2.465 (4.7%)<br>7.233 (13.9%)<br>5.207 (10.9%)<br>916 (1.8%)<br>2.664 (5.1%)<br>2.514 (4.8%)<br>2.214 (4.3%)<br>18,258 (35.2%)<br>14,318 (27.6%)<br>19,220 (37.0%)<br>4,261 (8.2%) | 0.85 (1.58)<br>1.72 (0.98)<br>0.13 (0.44)<br>36 (1.3%)<br>245 (9.1%)<br>293 (10.8%)<br>47 (1.7%)<br>182 (6.7%)<br>133 (4.9%)<br>935 (34.6%)<br>856 (31.7%)<br>1,105 (40.9%)<br>195 (7.2%) | 0.0768 -0.1989 0.2162 0.2003 0.1509 -0.0262 0.0076 -0.0679 -0.093 -0.0286 0.0126 -0.0899 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%)<br>9,241 (11.3%)<br>7,768 (9.5%)<br>1,296 (1.6%)<br>3,671 (4.5%)<br>3,501 (4.3%)<br>3,240 (3.9%)<br>23,213 (28.3%)<br>19,706 (24.0%) | 0.70 (1.45)<br>1.57 (0.96)<br>0.31 (0.40)<br>049 (0.9%)<br>321 (5.8%)<br>401 (7.3%)<br>066 (1.2%)<br>167 (3.0%)<br>171 (3.1%)<br>1,132 (0.6%)<br>1,052 (19.1%)<br>1,475 (26.8%)<br>248 (4.5%) | 0.115;<br>0.1984<br>0.1923<br>0.1977<br>0.0794<br>0.0341<br>0.0248<br>0.0694<br>0.1799<br>0.1194<br>0.1634<br>0.0958 |
| HU - Recent hospitalization (-30 days to Index Rx date); n (%) HU - Old hospitalizations (-180 to -31 days); n (%) HU - Hu - Mammong m; n (%) HU - Pap smear; n (%) HU - Prostate exam for DRE; n (%) HU - Frostate exam for DRE; n (%) HU - Brostate exam for DRE; n (%) HU - Hospitale Expendidoscopy or colonoscopy or CT virtual colonoscopy; n (%) HU - Bone mineral density; n (%) HU - Flu vaccine; n (%) HU - Preumococcal vaccine; n (%) Lab - Occurrence of 24-hour urine test; n (%) Lab - Occurrence of urine albumin test ordered; n (%) Lab - Occurrence of urine albumin test ordered; n (%) | 0.15 (0.50)<br>617 (2.9%)<br>2,008 (9.5%)<br>2,561 (12.1%)<br>380 (1.8%)<br>1,007 (4.7%)<br>987 (4.7%)<br>1,026 (4.8%)<br>4,955 (2.3.3%)<br>5,388 (25.4%)<br>8,939 (42.1%)<br>1,202 (5.7%)<br>11,639 (54.8%) | 1.52 (0.91) 0.12 (0.44) 13 (1.5%) 76 (8.7%) 108 (12.4%) 13 (2.2%) 38 (4.4%) 38 (4.4%) 38 (4.4%) 197 (22.6%) 196 (22.5%) 370 (42.5%) 53 (6.1%) 467 (53.6%) 394 (45.2%) | 0.0213<br>0.0637<br>0.0956<br>0.0278<br>0.0995<br>0.0278<br>0.0092<br>0.0144<br>0.0446<br>0.0191<br>0.0166<br>0.0680<br>-0.0081<br>-0.00241<br>0.1525 | 0.96 (0.98)<br>0.14 (0.44)<br>254 (2.8%)<br>841 (9.3%)<br>754 (8.4%)<br>261 (2.9%)<br>315 (3.5%)<br>497 (5.5%)<br>196 (2.2%)<br>1,562 (17.3%)<br>1,246 (13.8%)<br>2,455 (27.3%)<br>466 (5.2%)<br>2,611 (29.0%)<br>724 (8.0%) | 1.39 (0.95)<br>0.08 (0.31)<br>18 (0.9%)<br>110 (5.7%)<br>181 (9.4%)<br>84 (4.4%)<br>82 (4.6%)<br>104 (5.4%)<br>39 (2.0%)<br>355 (18.4%)<br>289 (15.0%)<br>755 (39.1%)<br>86 (4.1%)<br>86 (2.44,6%)<br>149 (7.7%) | -0.4455<br>0.1576<br>0.1414<br>0.1370<br>-0.0351<br>-0.0801<br>-0.0558<br>0.0044<br>0.0139<br>-0.0287<br>-0.0342<br>-0.2526<br>0.0523<br>-0.3278<br>0.0112 | 1.53 (0.93) 0.25 (0.65) 2.465 (4.7%) 7.233 (13.9%) 5.207 (10.0%) 916 (1.8%) 2.664 (5.1%) 2.514 (4.8%) 2.214 (4.3%) 18,258 (35.2%) 14,318 (27.6%) 19,220 (37.0%) 4,261 (8.2%) 2,1500 (41.4%) 46,435 (89.5%) | 0.85 (1.58) 1.72 (0.98) 0.13 (0.44) 36 (1.3%) 245 (9.1%) 293 (10.8%) 47 (1.7%) 182 (6.7%) 133 (4.9%) 935 (34.6%) 856 (31.7%) 1.105 (40.9%) 1.277 (47.3%) 2,507 (92.8%) | 0.0768 -0.1989 0.2162 0.2003 0.1509 -0.0262 0.0076 -0.0679 -0.0093 -0.0286 0.0126 -0.0899 -0.0800 0.0375 -0.1190 -0.1164 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%)<br>9,241 (11.3%)<br>7,768 (9.5%)<br>1,296 (1.6%)<br>3,501 (4.3%)<br>3,501 (4.3%)<br>3,240 (3.9%)<br>23,213 (28.3%)<br>19,706 (24.0%)<br>28,159 (34.3%)<br>5,463 (6.7%)<br>33,139 (40.3%)<br>57,642 (70.2%) | 0.70 (1.45)<br>1.57 (0.96)<br>0.11 (0.40)<br>0.49 (0.9%)<br>321 (5.8%)<br>401 (7.3%)<br>066 (1.2%)<br>220 (4.0%)<br>167 (3.0%)<br>1,132 (20.6%)<br>1,132 (20.6%)<br>1,475 (26.8%)<br>248 (4.5%)<br>1,744 (31.7%)<br>2,901 (52.7%) | 0.115;<br>0.198;<br>0.192;<br>0.197;<br>0.0794;<br>0.0341;<br>0.0248;<br>0.043;<br>0.1799;<br>0.1194;<br>0.043;<br>0.1799;<br>0.1634;<br>0.1799;<br>0.3655; |
| HU - Recent hospitalization (-30 days to index fix date); n (%) HU - Old hospitalization (-180 to -31 days); n (%) HU - Hu - Mammograp; n (%) HU - Paps smear; n (%) HU - Paps smear in (%) HU - Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%) HU - Flox non-mineral density; n (%) HU - Blownen imieral density; n (%) HU - Flox non-mineral density; n (%) HU - Flox non-mineral density; n (%) HU - Pneumococcal vaccine; n (%) Lab - Occurrence of 24-hour urine test; n (%) Lab - Occurrence of retrianiline tests ordered; n (%) Lab - Occurrence of urine albumin test ordered; n (%) Lab - Occurrence of urine albumin test ordered; n (%) Lab - Occurrence of urine albumin test ordered; n (%) SES Proxy - Copay for pharmacy cost (charges in U. S. \$)mean (sd) | 0.15 (0.50)<br>617 (2.9%)<br>2,008 (9.5%)<br>2,081 (9.5%)<br>2,561 (12.1%)<br>380 (1.8%)<br>1,007 (4.7%)<br>987 (4.7%)<br>1,026 (4.8%)<br>4,955 (23.3%)<br>5,388 (25.4%)<br>8,939 (42.1%)<br>1,202 (5.7%)<br>11,039 (54.8%)<br>11,207 (52.8%) | 1.52 (0.91) 0.12 (0.44) 13 (1.5%) 76 (8.7%) 108 (12.4%) 19 (2.2%) 38 (4.4%) 38 (4.4%) 38 (4.4%) 197 (2.5%) 196 (22.5%) 370 (42.5%) 38 (6.1%) 467 (33.6%) 394 (45.2%) 33.64 (35.58) | -0.0213<br>0.0637<br>0.0936<br>0.0278<br>-0.0092<br>-0.0286<br>0.0144<br>0.0446<br>0.0191<br>0.0166<br>0.0680<br>-0.0081<br>-0.0081<br>-0.0241<br>0.1525 | 0.96 (0.98)<br>0.14 (0.44)<br>254 (2.8%)<br>841 (9.3%)<br>754 (8.4%)<br>261 (2.9%)<br>315 (3.5%)<br>497 (5.5%)<br>196 (2.2%)<br>1,552 (17.3%)<br>1,246 (13.8%)<br>2,455 (27.3%)<br>466 (5.2%)<br>2,611 (29.0%)<br>724 (8.0%) | 1.39 (0.95)<br>0.08 (0.31)<br>18 (0.9%)<br>110 (5.7%)<br>181 (9.4%)<br>84 (4.4%)<br>88 (4.6%)<br>104 (5.4%)<br>39 (2.0%)<br>35 (18.4%)<br>289 (15.0%)<br>755 (39.1%)<br>80 (4.1%)<br>86 (4.6%)<br>149 (7.7%) | 0.4455<br>0.1576<br>0.1414<br>0.1414<br>0.1370<br>-0.0351<br>-0.0801<br>-0.0558<br>0.0044<br>0.0139<br>-0.0287<br>-0.0342<br>-0.2526<br>0.0523<br>-0.3278<br>0.0112 | 1.53 (0.93)<br>0.25 (0.65)<br>2.465 (4.7%)<br>7.233 (13.9%)<br>5.207 (10.0%)<br>916 (1.8%)<br>2.514 (4.8%)<br>2.214 (4.3%)<br>18.258 (35.2%)<br>14,318 (27.6%)<br>19,220 (37.0%)<br>4,261 (8.2%)<br>21,500 (41.4%)<br>46,435 (89.5%) | 0.85 (1.58) 1.72 (0.98) 1.72 (0.98) 0.13 (0.44) 36 (1.3%) 245 (9.1%) 293 (10.8%) 47 (1.7%) 132 (6.7%) 134 (5.0%) 133 (4.9%) 935 (34.6%) 856 (31.7%) 1.105 (40.9%) 1.57 (7.2%) 1.27 (7.2%) 1.27 (7.2%) 2.507 (92.8%) | 0.0768 -0.1989 0.2162 0.2003 0.1509 -0.0262 0.0076 -0.0679 -0.0093 -0.0286 0.0126 -0.0899 -0.0890 -0.0890 -0.1164 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%)<br>9,241 (11.3%)<br>7,768 (9.5%)<br>1,296 (1.6%)<br>3,671 (4.5%)<br>3,501 (4.3%)<br>3,240 (3.9%)<br>23,213 (28.3%)<br>19,706 (24.0%)<br>5,463 (6.7%)<br>3,3139 (40.3%)<br>5,463 (6.7%) | 0.70 (1.45)<br>1.57 (0.96)<br>0.11 (0.40)<br>0.49 (0.9%)<br>321 (5.8%)<br>401 (7.3%)<br>066 (1.2%)<br>107 (3.0%)<br>167 (3.0%)<br>1,052 (19.1%)<br>1,132 (20.6%)<br>1,052 (19.1%)<br>1,475 (26.8%)<br>248 (4.5%)<br>248 (4.5%)<br>29.1 (3.1%) | 0.1152<br>0.1984<br>0.1923<br>0.1977<br>0.0794<br>0.0341<br>0.0694<br>0.0435<br>0.1799<br>0.1194<br>0.0583<br>0.1795<br>0.3655 |
| HU - Recent hospitalization (-30 days to Index Rx date); n (%) HU - Old hospitalizations (-180 to -3.1 days); n (%) HU - Mammograp; n (%) HU - Paps smear; n (%) HU - Prostate exam for DRE; n (%) HU - Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%) HU - Bone mineral density; n (%) HU - Bone mineral density; n (%) HU - Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%) HU - Preumococcal vaccine; n (%) Lab - Occurrence of 24-hour urine test; n (%) Lab - Occurrence of urine albumin test ordered; n (%) Lab - Occurrence of urine albumin test ordered; n (%) SES Proxy - Copay for pharmacy cost (charges in U.S. S)mean (sd) SES Proxy - Copay for pharmacy cost (charges in U.S. S)mean (sd) | 0.15 (0.50)<br>617 (2.9%)<br>2,008 (9.5%)<br>2,561 (12.1%)<br>380 (1.8%)<br>1,007 (4.7%)<br>987 (4.7%)<br>1,026 (4.8%)<br>4,955 (2.3.3%)<br>5,388 (25.4%)<br>8,939 (42.1%)<br>1,202 (5.7%)<br>11,639 (54.8%) | 1.52 (0.91) 0.12 (0.44) 13 (1.5%) 76 (8.7%) 108 (12.4%) 13 (2.2%) 38 (4.4%) 38 (4.4%) 38 (4.4%) 197 (22.6%) 196 (22.5%) 370 (42.5%) 53 (6.1%) 467 (53.6%) 394 (45.2%) | 0.0213<br>0.0637<br>0.0956<br>0.0278<br>0.0995<br>0.0278<br>0.0092<br>0.0144<br>0.0446<br>0.0191<br>0.0166<br>0.0680<br>-0.0081<br>-0.00241<br>0.1525 | 0.96 (0.98)<br>0.14 (0.44)<br>254 (2.8%)<br>841 (9.3%)<br>754 (8.4%)<br>261 (2.9%)<br>315 (3.5%)<br>497 (5.5%)<br>196 (2.2%)<br>1,562 (17.3%)<br>1,246 (13.8%)<br>2,455 (27.3%)<br>466 (5.2%)<br>2,611 (29.0%)<br>724 (8.0%) | 1.39 (0.95)<br>0.08 (0.31)<br>18 (0.9%)<br>110 (5.7%)<br>181 (9.4%)<br>84 (4.4%)<br>82 (4.6%)<br>104 (5.4%)<br>39 (2.0%)<br>355 (18.4%)<br>289 (15.0%)<br>755 (39.1%)<br>86 (4.1%)<br>86 (2.44,6%)<br>149 (7.7%) | -0.4455<br>0.1576<br>0.1414<br>0.1370<br>-0.0351<br>-0.0801<br>-0.0558<br>0.0044<br>0.0139<br>-0.0287<br>-0.0342<br>-0.2526<br>0.0523<br>-0.3278<br>0.0112 | 1.53 (0.93) 0.25 (0.65) 2.465 (4.7%) 7.233 (13.9%) 5.207 (10.0%) 916 (1.8%) 2.664 (5.1%) 2.514 (4.8%) 2.214 (4.3%) 18,258 (35.2%) 14,318 (27.6%) 19,220 (37.0%) 4,261 (8.2%) 2,1500 (41.4%) 46,435 (89.5%) | 0.85 (1.58) 1.72 (0.98) 0.13 (0.44) 36 (1.3%) 245 (9.1%) 293 (10.8%) 47 (1.7%) 182 (6.7%) 133 (4.9%) 935 (34.6%) 856 (31.7%) 1.105 (40.9%) 1.277 (47.3%) 2,507 (92.8%) | 0.0768 -0.1989 0.2162 0.2003 0.1509 -0.0262 0.0076 -0.0679 -0.0093 -0.0286 0.0126 -0.0899 -0.0800 0.0375 -0.1190 -0.1164 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%)<br>9,241 (11.3%)<br>7,768 (9.5%)<br>1,296 (1.6%)<br>3,501 (4.3%)<br>3,501 (4.3%)<br>3,240 (3.9%)<br>23,213 (28.3%)<br>19,706 (24.0%)<br>28,159 (34.3%)<br>5,463 (6.7%)<br>33,139 (40.3%)<br>57,642 (70.2%) | 0.70 (1.45)<br>1.57 (0.96)<br>0.11 (0.40)<br>0.49 (0.9%)<br>321 (5.8%)<br>401 (7.3%)<br>066 (1.2%)<br>220 (4.0%)<br>167 (3.0%)<br>1,132 (20.6%)<br>1,132 (20.6%)<br>1,475 (26.8%)<br>248 (4.5%)<br>1,744 (31.7%)<br>2,901 (52.7%) | 0.115;<br>0.198;<br>0.192;<br>0.197;<br>0.0794;<br>0.0341;<br>0.0248;<br>0.043;<br>0.1799;<br>0.1194;<br>0.043;<br>0.1799;<br>0.1634;<br>0.1799;<br>0.3655; |
| HU - Recent hospitalization (-30 days to Index Rx date); n (%) HU - Old hospitalization (-180 to -31 days); n (%) HU - Days mean; n (%) HU - Pass mean for DRE; n (%) HU - Prostate exam for DRE; n (%) HU - Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%) HU - Bone mineral density; n (%) HU - Flou vaccine; n (%) HU - Flou vaccine; n (%) HU - Preumococcal vaccine; n (%) Lab - Occurrence of 24-hour urine test; n (%) Lab - Occurrence of virtinal bumin test ordered; n (%) Lab - Occurrence of virtinal bumin test ordered; n (%) Lab - Occurrence of virtinal bumin test ordered; n (%) SES Proxy - Copay for pharmacy cost (charges in U.S. \$) mean (sd) SES Proxy - Copay for pharmacy cost (charges in U.S. \$) mean (sd) | 0.15 (0.50)<br>617 (2.9%)<br>2,008 (9.5%)<br>2,561 (12.1%)<br>380 (1.8%)<br>1,007 (4.7%)<br>987 (4.7%)<br>1,026 (4.8%)<br>4,955 (23.3%)<br>5,388 (25.4%)<br>8,939 (42.1%)<br>1,202 (5.7%)<br>11,639 (54.8%)<br>11,207 (52.8%) | 1.52 (0.91) 0.12 (0.44) 1.3 (1.5%) 76 (8.7%) 108 (12.4%) 1.9 (2.2%) 38 (4.4%) 38 (4.4%) 38 (4.4%) 37 (42.5%) 196 (22.5%) 196 (22.5%) 370 (42.5%) 394 (45.2%) 394 (45.2%) | 0.0213<br>0.0637<br>0.0956<br>0.0278<br>0.0278<br>0.0226<br>0.0144<br>0.0446<br>0.0191<br>0.0166<br>0.0680<br>0.0680<br>0.0081<br>0.0241<br>0.1525<br>0.1450 | 0.96 (0.98)<br>0.14 (0.44)<br>254 (2.8%)<br>841 (9.3%)<br>754 (8.4%)<br>261 (2.9%)<br>315 (3.5%)<br>497 (5.5%)<br>196 (2.2%)<br>1,562 (17.3%)<br>1,246 (13.8%)<br>2,455 (27.3%)<br>466 (5.2%)<br>2,611 (29.0%)<br>724 (8.0%)<br>20.33 (20.86)<br>0 (0.0%) | 1.39 (0.95)<br>0.08 (0.31)<br>1.8 (0.9%)<br>1.10 (5.7%)<br>1.81 (9.4%)<br>84 (4.4%)<br>88 (4.6%)<br>1.04 (5.4%)<br>3.9 (2.0%)<br>3.55 (18.4%)<br>2.89 (15.0%)<br>7.55 (3.9.1%)<br>8.62 (44.6%)<br>1.49 (7.7%)<br>24.65 (25.50)<br>0 (0.0%) | 0.4455<br>0.1576<br>0.1414<br>0.1370<br>-0.0801<br>-0.0801<br>-0.0558<br>0.0044<br>0.0139<br>-0.0287<br>-0.0342<br>-0.2526<br>0.0523<br>0.0523<br>-0.0523<br>-0.0112 | 1.53 (0.93) 0.25 (0.65) 2.465 (4.7%) 7.233 (13.9%) 5.207 (10.0%) 916 (18.5%) 2.664 (5.1%) 2.664 (5.1%) 2.514 (4.8%) 2.214 (4.3%) 18,258 (35.2%) 14,318 (27.6%) 19,220 (37.0%) 4,261 (8.2%) 21,500 (41.4%) 46,435 (89.5%) | 0.85 (1.58) 1.72 (0.98) 1.72 (0.98) 1.73 (0.98) 1.74 (0.98) 2.65 (9.1%) 2.93 (10.8%) 4.7 (1.7%) 1.94 (5.0%) 1.95 (3.4.6%) 8.95 (3.4.6%) 8.95 (3.4.7%) 1.105 (40.9%) 1.105 (40.9%) 1.277 (47.3%) 2.507 (92.8%) 31.18 (43.28) 0 (0.0%) | 0.0768 -0.1989 0.2162 0.2003 0.1509 -0.0262 0.0076 -0.0679 -0.0093 -0.0286 0.0126 -0.0899 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%)<br>9,241 (11.3%)<br>7,768 (9.5%)<br>1,296 (1.6%)<br>3,671 (4.5%)<br>3,501 (4.3%)<br>3,501 (4.3%)<br>19,706 (24.0%)<br>28,139 (34.3%)<br>5,463 (6.7%)<br>33,139 (40.3%)<br>5,642 (70.2%)<br>27,23 (33.78)<br>6,063 (7.4%) | 0.70 (1.45) 1.57 (0.96) 0.11 (0.40) 0.49 (0.9%) 321 (5.8%) 401 (7.3%) 401 (7.3%) 220 (4.0%) 167 (3.0%) 1,132 (20.6%) 1,052 (19.1%) 1,475 (26.8%) 1,744 (31.7%) 2,901 (52.7%) 29.28 (36.71) 194 (3.5%) | 0.115;<br>0.1984<br>0.1922<br>0.1927<br>0.0794<br>0.0341<br>0.0244<br>0.0694<br>0.043;<br>0.1799<br>0.1194<br>0.0958<br>0.1799<br>0.3655 |
| HU - Recent hospitalization (-30 days to Index Rx date); n (%) HU - Old hospitalizations (-180 to -31 days); n (%) HU - Dammorgan; n (%) HU - Paps smear; n (%) HU - Prostate exam for DRE; n (%) HU - Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%) HU - Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%) HU - Bloome mineral density; n (%) HU - Plex vaccine; n (%) HU - Pneumococcal vaccine; n (%) HU - Pneumococcal vaccine; n (%) Lab - Occurrence of 24-hour urine test; n (%) Lab - Occurrence of restinine tests ordered; n (%) Lab - Occurrence of urine albumin test ordered; n (%) Lab - Occurrence of HgA1c test; n (%) SES Proxy - Copay for pharmacy cost (charges in U.S. 5)mean (sd) SES Proxy - Low income indicator; n (%) SES Proxy - Business typeCommercial; n (%) | 0.15 (0.50)<br>617 (2.9%)<br>2,008 (9.5%)<br>2,08 (9.5%)<br>2,561 (12.1%)<br>380 (1.8%)<br>1,007 (4.7%)<br>987 (4.7%)<br>1,026 (4.8%)<br>4,955 (23.3%)<br>5,388 (25.4%)<br>1,202 (5.7%)<br>11,202 (5.7%)<br>11,207 (52.8%)<br>28.11 (33.95)<br>6,063 (28.6%) | 1.52 (0.91) 0.12 (0.44) 13 (1.5%) 76 (8.7%) 108 (12.4%) 19 (2.2%) 38 (4.4%) 33 (8.3%) 38 (4.4%) 197 (22.6%) 196 (22.5%) 370 (42.5%) 53 (6.1%) 467 (53.6%) 394 (45.2%) 494 (22.3%) 403 (46.3%) | 0.0213<br>0.0637<br>0.0956<br>0.0278<br>0.0226<br>0.0144<br>0.0144<br>0.0191<br>0.0166<br>0.0680<br>-0.0680<br>-0.0241<br>0.0120<br>0.01241<br>0.01525<br>0.1525<br>0.1450 | 0.96 (0.98)<br>0.14 (0.44)<br>254 (2.8%)<br>841 (9.3%)<br>754 (8.4%)<br>261 (2.9%)<br>315 (3.5%)<br>196 (2.2%)<br>1,552 (17.3%)<br>1,246 (13.8%)<br>2,415 (27.3%)<br>466 (5.2%)<br>2,611 (29.0%)<br>724 (8.0%)<br>0 (0.0%) | 1.39 (0.95)<br>0.08 (0.31)<br>18 (0.9%)<br>110 (5.7%)<br>181 (9.3%)<br>84 (4.4%)<br>88 (4.6%)<br>104 (5.4%)<br>39 (2.0%)<br>355 (18.4%)<br>289 (15.0%)<br>755 (39.1%)<br>80 (4.1%)<br>86 (44.6%)<br>149 (7.7%)<br>24.65 (25.50)<br>0 (0.0%) | 0.4455 0.1576 0.1514 0.1310 0.1414 0.1370 0.0801 0.0058 0.0044 0.0139 0.0342 0.0342 0.0523 0.0523 0.0523 0.0112 0.0118 0.01184 BDIV/01 | 1.53 (0.93)<br>0.25 (0.65)<br>2.465 (4.7%)<br>7.233 (13.9%)<br>5.207 (10.0%)<br>916 (1.8%)<br>2.664 (5.1%)<br>2.514 (4.8%)<br>2.214 (4.3%)<br>2.214 (4.3%)<br>2.214 (4.3%)<br>4.261 (8.2%)<br>14,318 (27.6%)<br>19,220 (37.0%)<br>4.261 (8.2%)<br>21,500 (41.4%)<br>46,435 (89.5%)<br>0 (0.0%) | 0.85 (1.58) 1.72 (0.98) 1.72 (0.98) 0.13 (0.44) 36 (1.3%) 245 (9.1%) 293 (10.8%) 47 (1.7%) 182 (6.7%) 134 (5.0%) 134 (5.0%) 135 (4.6%) 856 (31.7%) 1.105 (40.9%) 1.95 (7.2%) 1.277 (47.3%) 2.507 (92.8%) 31.18 (43.28) 0 (0.0%) | 0.0768 -0.1989 0.2162 0.2003 0.1509 -0.0262 0.0076 -0.0679 -0.0093 -0.0266 0.0126 -0.0899 -0.0800 0.0375 -0.1164 -0.0788 #DIV/01 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%)<br>9,241 (1.13%)<br>7,768 (9.5%)<br>1,296 (1.6%)<br>3,671 (4.5%)<br>3,501 (4.3%)<br>3,240 (3.9%)<br>23,213 (28.3%)<br>19,706 (24.0%)<br>28,159 (34.3%)<br>5,463 (6.7%)<br>33,139 (0.3%)<br>57,642 (70.2%)<br>27,23 (33.78)<br>6,063 (7.4%) | 0.70 (1.45)<br>1.57 (0.96)<br>0.11 (0.40)<br>0.49 (0.9%)<br>321 (5.8%)<br>401 (7.3%)<br>066 (1.2%)<br>220 (4.0%)<br>167 (3.0%)<br>171 (3.1%)<br>1,132 (20.6%)<br>1,052 (19.1%)<br>1,475 (26.8%)<br>248 (4.5%)<br>2,901 (52.7%)<br>29.28 (36.71)<br>194 (3.5%)<br>403 (7.3%) | 0.115:<br>0.198:<br>0.192:<br>0.197:<br>0.0794:<br>0.034:<br>0.0694:<br>0.0694:<br>0.1799:<br>0.1196:<br>0.1634:<br>0.1799:<br>0.365:<br>0.1726:<br>0.1726:<br>0.1726: |
| HU - Recent hospitalization (-30 days to index Rx date); n (%) HU - Old hospitalization (-180 to -31 days); n (%) HU - Hu - Mammorgan; n (%) HU - Pag smear; n (%) HU - Pag smear; n (%) HU - Prostate exam for DRE; n (%) HU - Flexible Sigmoidoscopy or colonoscopy or CTvirtual colonoscopy; n (%) HU - Bone mineral density; n (%) HU - Bone mineral density; n (%) HU - Pneumococcal vaccine; n (%) HU - Pneumococcal vaccine; n (%) Lab - Occurrence of 24-hour urine tests ordered; n (%) Lab - Occurrence of urine albumin test ordered; n (%) Lab - Occurrence of urine albumin test ordered; n (%) Seb Proxy - Copay for pharmacy cost (charges in U.S. \$)mean (sd) SES Proxy - Low income indicator; n (%) SES Proxy - Low income indicator; n (%)Commercial; n (%)Medicare, n (%) | 0.15 (0.50)<br>617 (2.9%)<br>2,008 (9.5%)<br>2,561 (12.1%)<br>380 (1.8%)<br>1,007 (4.7%)<br>987 (4.7%)<br>1,026 (4.8%)<br>4,955 (23.3%)<br>5,388 (25.4%)<br>8,939 (42.1%)<br>1,202 (5.7%)<br>11,639 (54.8%)<br>11,207 (52.8%) | 1.52 (0.91) 0.12 (0.44) 1.3 (1.5%) 76 (8.7%) 108 (12.4%) 1.9 (2.2%) 38 (4.4%) 38 (4.4%) 38 (4.4%) 37 (42.5%) 196 (22.5%) 196 (22.5%) 370 (42.5%) 394 (45.2%) 394 (45.2%) | 0.0213<br>0.0637<br>0.0956<br>0.0278<br>0.0278<br>0.0226<br>0.0144<br>0.0446<br>0.0191<br>0.0166<br>0.0680<br>0.0680<br>0.0081<br>0.0241<br>0.1525<br>0.1450 | 0.96 (0.98)<br>0.14 (0.44)<br>254 (2.8%)<br>841 (9.3%)<br>754 (8.4%)<br>261 (2.9%)<br>315 (3.5%)<br>497 (5.5%)<br>196 (2.2%)<br>1,562 (17.3%)<br>1,246 (13.8%)<br>2,455 (27.3%)<br>466 (5.2%)<br>2,611 (29.0%)<br>724 (8.0%)<br>20.33 (20.86)<br>0 (0.0%) | 1.39 (0.95)<br>0.08 (0.31)<br>1.8 (0.9%)<br>1.10 (5.7%)<br>1.81 (9.4%)<br>84 (4.4%)<br>88 (4.6%)<br>1.04 (5.4%)<br>3.9 (2.0%)<br>3.55 (18.4%)<br>2.89 (15.0%)<br>7.55 (3.9.1%)<br>8.62 (44.6%)<br>1.49 (7.7%)<br>24.65 (25.50)<br>0 (0.0%) | 0.4455<br>0.1576<br>0.1414<br>0.1370<br>-0.0801<br>-0.0801<br>-0.0558<br>0.0044<br>0.0139<br>-0.0287<br>-0.0342<br>-0.2526<br>0.0523<br>0.0523<br>-0.0523<br>-0.0112 | 1.53 (0.93) 0.25 (0.65) 2.465 (4.7%) 7.233 (13.9%) 5.207 (10.0%) 916 (18.5%) 2.664 (5.1%) 2.664 (5.1%) 2.514 (4.8%) 2.214 (4.3%) 18,258 (35.2%) 14,318 (27.6%) 19,220 (37.0%) 4,261 (8.2%) 21,500 (41.4%) 46,435 (89.5%) | 0.85 (1.58) 1.72 (0.98) 1.72 (0.98) 1.73 (0.98) 1.74 (0.98) 2.65 (9.1%) 2.93 (10.8%) 4.7 (1.7%) 1.94 (5.0%) 1.95 (3.4.6%) 8.95 (3.4.6%) 8.95 (3.4.7%) 1.105 (40.9%) 1.105 (40.9%) 1.277 (47.3%) 2.507 (92.8%) 31.18 (43.28) 0 (0.0%) | 0.0768 -0.1989 0.2162 0.2003 0.1509 -0.0262 0.0076 -0.0679 -0.0093 -0.0286 0.0126 -0.0899 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%)<br>9,241 (11.3%)<br>7,768 (9.5%)<br>1,296 (1.6%)<br>3,671 (4.5%)<br>3,501 (4.3%)<br>3,501 (4.3%)<br>19,706 (24.0%)<br>28,139 (34.3%)<br>5,463 (6.7%)<br>33,139 (40.3%)<br>5,642 (70.2%)<br>27,23 (33.78)<br>6,063 (7.4%) | 0.70 (1.45) 1.57 (0.96) 0.11 (0.40) 0.49 (0.9%) 321 (5.8%) 401 (7.3%) 401 (7.3%) 220 (4.0%) 167 (3.0%) 1,132 (20.6%) 1,052 (19.1%) 1,475 (26.8%) 1,744 (31.7%) 2,901 (52.7%) 29.28 (36.71) 194 (3.5%) | 0.115:<br>0.198:<br>0.192:<br>0.197:<br>0.0794:<br>0.034:<br>0.0694:<br>0.0694:<br>0.1799:<br>0.1196:<br>0.1634:<br>0.1799:<br>0.365:<br>0.1726:<br>0.1726:<br>0.1726: |
| HU - Recent hospitalization (-30 days to index Rx date); n (%) HU - Old hospitalization (-180 to -31 days); n (%) HU - Old hospitalizations (-180 to -31 days); n (%) HU - Pags smear; n (%) HU - Pags smear; n (%) HU - Prostate exam for DRE; n (%) HU - Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%) HU - Bone mineral density; n (%) HU - Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%) HU - Preumococcal vaccine; n (%) HU - Preumococcal vaccine; n (%) Lab - Occurrence of 24-hour urine test; n (%) Lab - Occurrence of virtual abumin test ordered; n (%) Lab - Occurrence of virtual abumin test ordered; n (%) Lab - Occurrence of virtual abumin test ordered; n (%) SES Proxy - Low income indicator; n (%) SES Proxy - Low income indicator; n (%) SES Proxy - Low income indicator; n (%) SES Proxy - Low income indicator; n (%)Commercial; n (%)Commercial; n (%)Commercial; n (%)Medicare; n (%) | 0.15 (0.50) 617 (2.9%) 617 (2.9%) 2,008 (9.5%) 2,061 (12.11%) 380 (1.8%) 1,007 (4.7%) 987 (4.7%) 1,026 (4.8%) 4,955 (23.3%) 5,388 (25.4%) 1,202 (5.7%) 1,202 (5.7%) 1,207 (52.8%) 28.11 (33.95) 6,063 (28.6%) 1,284 (6.0%) 19,940 (94.0%) | 1.52 (0.91) 0.12 (0.44) 13 (1.5%) 76 (8.7%) 108 (12.4%) 19 (12.4%) 13 (3.8%) 38 (4.4%) 38 (4.4%) 38 (4.4%) 197 (2.5%) 196 (22.5%) 370 (42.5%) 370 (42.5%) 394 (457.2%) 394 (457.2%) 467 (53.6%) 394 (457.2%) 403 (46.3%) 403 (46.3%) 408 (53.7%) | 0.0213<br>0.0637<br>0.0956<br>0.0278<br>0.0295<br>0.0286<br>0.0144<br>0.0191<br>0.0166<br>0.0680<br>-0.0081<br>0.0170<br>0.0241<br>0.1525<br>-1.0319<br>1.0319 | 0.96 (0.98) 0.14 (0.44) 254 (2.8%) 841 (9.3%) 754 (8.4%) 261 (2.9%) 315 (3.5%) 497 (5.5%) 196 (2.2%) 1,552 (7.3%) 1,246 (13.8%) 2,455 (27.3%) 466 (5.2%) 2,611 (2.9%) 724 (8.0%) 0 (0.0%) 0 (0.0%) | 1.39 (0.95) 0.08 (0.31) 18 (0.9%) 110 (5.7%) 110 (5.7%) 181 (9.4%) 84 (4.4%) 88 (4.6%) 104 (5.4%) 39 (2.0%) 35 (18.4%) 289 (15.0%) 755 (39.1%) 80 (4.1%) 86 (24.6%) 149 (7.7%) 24.65 (25.50) 0 (0.0%) 0 (0.0%) | 0.4455 0.1576 0.1414 0.1370 0.0414 0.1370 -0.0801 -0.0558 0.0044 0.0139 -0.0287 -0.0342 -0.0287 -0.0342 -0.1854 -0.0112 -0.1854 -0.0112 -0.1854 -0.0112 | 1.53 (0.93) 0.25 (0.65) 2.465 (4.7%) 7.233 (13.9%) 5.207 (10.0%) 916 (1.8%) 2.664 (5.1%) 2.514 (4.8%) 2.214 (4.3%) 2.214 (4.3%) 4.214 (4.3%) 4.261 (8.2%) 4.261 (8.2%) 4.261 (8.2%) 4.261 (8.2%) 0.00%) 0 (0.0%) | 0.85 (1.58) 1.72 (0.98) 1.72 (0.98) 0.13 (0.44) 36 (1.3%) 245 (9.1%) 293 (10.8%) 47 (1.7%) 132 (6.7%) 134 (5.0%) 133 (4.9%) 935 (34.6%) 856 (31.7%) 1.105 (40.9%) 1.95 (7.2%) 1.277 (47.3%) 2.507 (92.8%) 0 (0.0%) 0 (0.0%) | 0.0768 -0.1899 -0.0899 | 0.91 (1.77) 1.46 (0.95) 0.21 (0.59) 3,082 (3.8%) 9,241 (11.3%) 7,768 (9.5%) 1,296 (1.6%) 3,671 (4.5%) 3,501 (4.3%) 3,204 (3.9%) 23,213 (28.3%) 19,706 (24.0%) 28,159 (34.3%) 5,463 (6.7%) 3,139 (40.3%) 57,642 (70.2%) 27,23 (33.78) 6,063 (7.4%) 1,284 (1.6%) 1,9,940 (24.3%) | 0.70 (1.45) 1.57 (0.96) 0.11 (0.40) 0.49 (0.9%) 321 (5.8%) 401 (7.3%) 0.66 (1.2%) 1.67 (3.0%) 1.71 (3.1%) 1.132 (20.6%) 1.052 (19.1%) 1.475 (26.8%) 1.475 (26.8%) 1.744 (31.7%) 2.901 (52.7%) 4.03 (7.3%) 4.03 (7.3%) 4.08 (8.5%) | 0.115 0.198 0.192 0.197 0.079 0.034 0.024 0.069 0.043 0.119 0.163 0.095 0.079 0.365 0.095 0.079 0.365 |
| HU - Recent hospitalization (-30 days to index Rx date); n (%) HU - Old hospitalization (-180 to -31 days); n (%) HU - Hu - Mammorgan; n (%) HU - Pag smear; n (%) HU - Pag smear; n (%) HU - Prostate exam for DRE; n (%) HU - Flexible Sigmoildoscopy or colonoscopy or CTvirtual colonoscopy; n (%) HU - Bloome mineral density; n (%) HU - Flexible Sigmoildoscopy or colonoscopy or CTvirtual colonoscopy; n (%) HU - Pneumococcal vaccine; n (%) HU - Pneumococcal vaccine; n (%) Lab - Occurrence of 24-hour urine test; n (%) Lab - Occurrence of creatinine tests ordered; n (%) Lab - Occurrence of urine albumin test ordered; n (%) Lab - Occurrence of HgA1c test; n (%) SES Proxy - Copay for pharmacy cost (charges in U.S. S)mean (sd) SES Proxy - Low income indicator; n (%) SES Proxy - Low income indicator; n (%)Commercial; n (%)Medicare; n (%)Medicare; n (%) | 0.15 (0.50) 617 (2.9%) 617 (2.9%) 2,008 (9.5%) 2,561 (12.1%) 380 (13%) 1,007 (4.7%) 987 (4.7%) 1,026 (4.8%) 4,955 (23.3%) 5,388 (25.4%) 8,939 (42.1%) 1,202 (5.7%) 11,639 (54.8%) 11,207 (52.8%) 11,207 (52.8%) 11,207 (52.8%) | 1.52 (0.91) 0.12 (0.44) 13 (1.5%) 76 (8.7%) 108 (12.4%) 13 (1.4%) 19 (2.2%) 38 (4.4%) 38 (4.4%) 197 (22.6%) 370 (42.5%) 53 (6.1%) 467 (53.6%) 394 (45.2%) 36.4 (35.58) 194 (22.3%) 468 (53.7%) 468 (53.7%) | 0.0213 0.0637 0.0956 0.0278 0.0278 0.00956 0.0278 0.0091 0.0092 0.0092 0.0091 0.0044 0.0191 0.0166 0.0580 0.0466 0.0170 0.0241 0.1525 0.1459 0.1459 0.1459 1.0319 | 0.96 (0.98) 0.14 (0.44) 254 (2.8%) 841 (9.3%) 754 (8.4%) 261 (2.9%) 315 (3.5%) 196 (2.2%) 1,552 (17.3%) 1,246 (13.8%) 2,455 (27.3%) 466 (5.2%) 2,611 (29.0%) 724 (8.0%) 0 (0.0%) 0 (0.0%) | 1.39 (0.95) 0.08 (0.31) 1.8 (0.9%) 1.10 (5.7%) 1.10 (5.7%) 1.81 (9.4%) 84 (4.4%) 88 (4.6%) 39 (2.0%) 39 (2.0%) 35 (1.8.4%) 289 (15.0%) 755 (39.1%) 80 (4.1%) 862 (44.6%) 149 (7.7%) 24.65 (25.50) 0 (0.0%) 0 (0.0%) | 0.4455 0.1576 0.1576 0.1414 0.1370 -0.0351 -0.0801 -0.0558 0.0044 0.0139 -0.0287 -0.0342 -0.0287 -0.03278 0.0112 -0.1854 #DIV/01 #DIV/01 #DIV/01 #DIV/01 | 1.53 (0.93) 0.25 (0.65) 2.465 (4.7%) 7.233 (13.9%) 5.207 (10.0%) 916 (1.8%) 2.664 (5.1%) 2.514 (4.8%) 2.214 (4.3%) 14.318 (27.6%) 14.318 (27.6%) 4.261 (8.2%) 21.500 (41.4%) 46.435 (89.5%) 0 (0.0%) 0 (0.0%) | 0.85 (1.58) 1.72 (0.98) 1.72 (0.98) 0.13 (0.44) 36 (1.3%) 245 (9.1%) 293 (10.8%) 47 (1.7%) 132 (6.7%) 134 (5.0%) 133 (4.9%) 935 (34.6%) 856 (31.7%) 1,105 (40.9%) 1,277 (47.3%) 2,507 (92.8%) 31.18 (43.28) 0 (0.0%) 0 (0.0%) | 0.0768 -0.1989 -0.1989 -0.2062 -0.0003 -0.0262 -0.0076 -0.0067 -0.0093 -0.0286 -0.0126 -0.0800 -0.0375 -0.1190 -0.1164 -0.0788 | 0.91 (1.77) 1.46 (0.95) 0.21 (0.59) 3,082 (3.8%) 9,241 (1.13%) 7,768 (9.5%) 1,296 (1.6%) 3,671 (4.5%) 3,501 (4.3%) 3,240 (3.9%) 23,213 (28.3%) 19,706 (24.0%) 28,159 (34.3%) 5,463 (6.7%) 33,139 (40.3%) 57,642 (70.2%) 57,642 (70.2%) 1,284 (1.6%) 1,284 (1.6%) 1,940 (24.3%) | 0.70 (1.45) 1.57 (0.96) 0.11 (0.40) 0.49 (0.9%) 321 (1.8%) 401 (7.3%) 0.66 (1.2%) 1.67 (3.0%) 1.67 (3.0%) 1.71 (3.1%) 1.72 (2.6.6%) 1.752 (19.1%) 1.475 (26.8%) 2.90 (152.7%) 2.91 (52.7%) 2.92 (3.5%) 4.03 (7.3%) 4.03 (7.3%) 4.03 (7.3%) 4.03 (7.3%) 4.03 (7.3%) | 0.115: 0.198: 0.199: 0.197: 0.079: 0.079: 0.0244: 0.069: 0.1034: 0.199: 0.1190: 0.163: 0.095: 0.1799: 0.365: 0.172: 0.279: 0.436: 0.0183: |
| HU - Recent hospitalization (-30 days to index Rx date); n (%) HU - Old hospitalization (-180 to -31 days); n (%) HU - Old hospitalization (-180 to -31 days); n (%) HU - Pap smear; n (%) HU - Prostate exam for DRE; n (%) HU - Frostate exam for DRE; n (%) HU - Flour section (-180 to -180 to -18 | 0.15 (0.50) 617 (2.9%) 2,081 (9.5%) 2,081 (9.5%) 2,561 (12.1%) 380 (1.8%) 1,007 (4.7%) 987 (4.7%) 1,026 (4.8%) 4,955 (2.3.3%) 5,388 (25.4%) 5,388 (25.4%) 1,202 (5.7%) 11,639 (54.8%) 11,207 (52.8%) 28.11 (33.95) 6,063 (28.6%) 1,284 (6.0%) 1,284 (6.0%) 1,940 (94.0%) 0 (0.0%) | 1.52 (0.91) 0.12 (0.44) 13 (1.5%) 76 (8.7%) 108 (12.4%) 13 (2.4%) 13 (2.4%) 13 (2.4%) 13 (4.4%) 13 (4.4%) 13 (4.5%) 19 (2.2.5%) 196 (22.5%) 196 (22.5%) 196 (22.5%) 196 (22.5%) 196 (22.5%) 196 (23.5%) 194 (23.5%) 194 (45.2%) 194 (23.3%) 403 (46.3%) 468 (53.7%) 0 (0.0%) | 0.0213 0.0637 0.0956 0.0278 0.0278 0.0226 0.0144 0.0446 0.0191 0.0166 0.0680 0.0680 0.0680 0.0241 0.1255 0.1450 0.1450 0.1450 | 0.96 (0.98) 0.14 (0.44) 254 (2.8%) 841 (9.3%) 754 (8.4%) 261 (2.9%) 315 (3.5%) 497 (5.5%) 196 (2.2%) 1,562 (17.3%) 1,246 (13.8%) 2,455 (27.3%) 466 (5.2%) 2,611 (29.0%) 724 (8.0%) 0 (0.0%) 0 (0.0%) 0 (0.0%) | 1.39 (0.95) 0.08 (0.31) 1.8 (0.9%) 1.10 (5.7%) 1.10 (5.7%) 1.81 (9.4%) 8.8 (4.6.4%) 8.8 (4.6.4%) 3.9 (2.0%) 3.55 (18.4.4%) 2.89 (15.0%) 2.89 (15.0%) 2.89 (15.0%) 2.99 (1.1%) 8.62 (4.4.6%) 1.49 (7.7%) 2.4.65 (25.50) 0 (0.0%) 0 (0.0%) 0 (0.0%) | 0.4455 0.1576 0.1576 0.1414 0.1370 0.0351 0.0051 0.0058 0.0044 0.0139 0.00287 0.0342 0.0327 0.0327 0.03278 0.0112 #DIV/01 #DIV/01 #DIV/01 0.5226 | 1.53 (0.93) 0.25 (0.65) 2.465 (4.7%) 7.233 (13.9%) 5.207 (10.0%) 916 (1.8%) 2.664 (5.1%) 2.664 (5.1%) 2.514 (4.8%) 2.214 (4.3%) 18,258 (35.2%) 14,318 (27.6%) 19,220 (37.0%) 4,261 (8.2%) 21,500 (41.4%) 46,435 (89.5%) 28.06 (35.48) 0 (0.0%) 0 (0.0%) | 0.85 (1.58) 1.72 (0.98) 1.73 (0.98) 1.74 (0.98) 3.6 (1.3%) 2.45 (9.1%) 2.93 (10.8%) 4.7 (1.7%) 1.82 (6.7%) 1.84 (5.0%) 1.85 (31.7%) 1.95 (40.9%) 1.105 (40.9%) 1.105 (40.9%) 1.277 (47.3%) 2.507 (92.8%) 31.18 (43.28) 0 (0.0%) 0 (0.0%) | 0.0768 -0.189 0.2162 0.2003 0.1509 -0.0262 0.0076 -0.0079 -0.0093 -0.0286 0.0126 -0.0809 -0.0800 -0.0375 -0.1190 -0.1164 -0.0788 #DIV/OI #DIV/OI | 0.91 (1.77) 1.46 (0.95) 0.21 (0.59) 3,082 (3.8%) 9,241 (11.3%) 7,768 (9.5%) 1,296 (1.6%) 3,671 (4.5%) 3,501 (4.3%) 3,501 (4.3%) 3,240 (3.9%) 23,213 (28.3%) 19,706 (24.0%) 28,159 (34.3%) 5,463 (6.7%) 3,139 (40.3%) 57,642 (70.2%) 27,23 (33.78) 6,063 (7.4%) 1,284 (1.6%) 1,940 (24.3%) 2,315 (2.8%) 957 (1.2%) | 0.70 (1.45) 1.57 (0.96) 0.11 (0.40) 0.49 (0.9%) 321 (5.8%) 401 (7.3%) 401 (7.3%) 166 (1.2%) 220 (4.0%) 167 (3.0%) 1,052 (19.1%) 1,132 (20.6%) 1,052 (19.1%) 1,475 (26.8%) 1,474 (31.7%) 2,901 (52.7%) 29.28 (36.71) 194 (3.5%) 403 (7.3%) 403 (7.3%) 468 (8.5%) 136 (2.5%) | 0.115:<br>0.1984<br>0.192;<br>0.197;<br>0.0794<br>0.0694<br>0.0693<br>0.1799<br>0.1194<br>0.1634<br>0.0955<br>0.1799<br>0.3655<br>0. |
| HU - Recent hospitalization (-30 days to index Rx date); n (%) HU - Old hospitalization (-180 to -31 days); n (%) HU - Hu - Mammorgan; n (%) HU - Pags smear; n (%) HU - Pags smear; n (%) HU - Flexible Sigmoidoscopy or cotonoscopy or CT virtual colonoscopy; n (%) HU - Flexible Sigmoidoscopy or cotonoscopy or CT virtual colonoscopy; n (%) HU - Bone mineral density; n (%) HU - Flexible Sigmoidoscopy or cotonoscopy or CT virtual colonoscopy; n (%) HU - Put vaccine; n (%) HU - Put vaccine; n (%) HU - Put vaccine; n (%) Lab - Occurrence of 24-hour urine test; n (%) Lab - Occurrence of creatinine tests ordered; n (%) Lab - Occurrence of HgA1c test; n (%) SES Proxy - Copay for pharmacy cost (charges in U.S. 5)mean (sd) SES Proxy - Low income indicator; n (%) SES Proxy - Business typeCommercial; n (%)Medicare; n (%)Medicare; n (%)Medicare; n (%)Medicare; n (%)PO; n (%) | 0.15 (0.50) 617 (2.9%) 6217 (2.9%) 2,008 (9.5%) 2,056 (12.13%) 380 (1.8%) 1,007 (4.7%) 987 (4.7%) 1,026 (4.8%) 4,955 (23.3%) 5,388 (25.4%) 1,202 (5.7%) 1,202 (5.7%) 1,202 (5.8%) 28.11 (33.95) 6,063 (28.6%) 1,284 (6.0%) 1,940 (94.0%) 0 (0.0%) 0 (0.0%) | 1.52 (0.91) 0.12 (0.44) 13 (1.5%) 76 (8.7%) 108 (12.4%) 13 (1.4%) 13 (2.3%) 38 (4.4%) 38 (4.4%) 38 (4.4%) 197 (2.5%) 196 (22.5%) 370 (42.5%) 53 (6.1%) 467 (53.6%) 394 (45.2%) 468 (53.7%) 403 (46.3%) 468 (53.7%) 0 (0.0%) 0 (0.0%) | 0.0213 0.0637 0.0956 0.0278 0.00956 0.0278 0.00956 0.0286 0.0144 0.0191 0.0166 0.0680 -0.0680 -0.0160 0.0165 0.0550 0.1450 -1.0319 1.0319 #DIV/OI #DIV/OI #DIV/OI #DIV/OI | 0.96 (0.98) 0.14 (0.44) 2.54 (2.8%) 841 (9.3%) 754 (8.4%) 261 (2.9%) 315 (3.5%) 497 (5.5%) 196 (2.2%) 1,552 (17.3%) 1,246 (13.8%) 2,611 (29.0%) 2,615 (2.9%) 2,616 (2.9%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 2,315 (25.7%) 957 (10.6%) | 1.39 (0.95) 0.08 (0.31) 1.8 (0.9%) 1.10 (5.7%) 1.10 (5.7%) 1.8 (1.94%) 8.4 (4.4%) 8.8 (4.6%) 1.04 (5.4%) 3.9 (2.0%) 3.95 (1.84%) 2.89 (1.5.0%) 7.55 (3.9.1%) 8.0 (4.1%) 8.0 (4.1%) 1.49 (7.7%) 1.49 (7.7%) 0 (0.0%) 0 (0.0%) 1.16 (7.0%) 1.16 (7.0%) 1.16 (7.9%) | 0.4455 0.1576 0.1574 0.1414 0.1370 -0.0801 -0.0558 0.0044 0.0139 -0.0287 -0.0287 -0.0342 -0.2526 0.0523 -0.3278 0.0112 -0.1854 -0.0102 -0.1854 -0.0102 -0.003 | 1.53 (0.93) 0.25 (0.65) 2.465 (4.7%) 7.233 (13.9%) 5.207 (10.0%) 916 (1.8%) 2.664 (5.1%) 2.514 (4.8%) 2.214 (4.3%) 2.214 (4.3%) 4.241 (8.2%) 14.318 (27.6%) 19.220 (37.0%) 4.261 (8.2%) 21.500 (41.4%) 46.435 (89.5%) 0 (0.0%) 0 (0.0%) 0 (0.0%) | 0.85 (1.58) 1.72 (0.98) 1.72 (0.98) 0.13 (0.44) 36 (1.3%) 245 (9.1%) 293 (10.8%) 47 (1.7%) 132 (6.7%) 134 (5.0%) 134 (5.0%) 134 (5.0%) 135 (34.6%) 856 (31.7%) 159 (7.2%) 1,105 (40.9%) 195 (7.2%) 1,277 (47.3%) 2,507 (92.8%) 31.18 (43.28) 0 (0.0%) 0 (0.0%) | 0.0768 -0.1989 -0.1989 -0.2162 -0.2003 -0.0056 -0.0076 -0.0679 -0.0093 -0.0286 -0.0150 -0.0809 -0.0800 -0.0375 -0.1190 -0.1164 -0.0788 #DIV/01 #DIV/01 #DIV/01 #DIV/01 #DIV/01 | 0.91 (1.77)<br>1.46 (0.95)<br>0.21 (0.59)<br>3,082 (3.8%)<br>9,241 (1.13%)<br>7,768 (9.5%)<br>1,296 (1.6%)<br>3,671 (4.5%)<br>3,501 (4.3%)<br>3,501 (4.3%)<br>3,240 (3.9%)<br>23,213 (28.3%)<br>19,706 (24.0%)<br>28,159 (34.3%)<br>5,463 (6.7%)<br>33,139 (0.3%)<br>57,642 (70.2%)<br>27,23 (33.78)<br>6,063 (7.4%)<br>1,284 (1.6%)<br>19,940 (24.3%)<br>2,315 (2.8%)<br>957 (1.2%) | 0.70 (1.45) 1.57 (0.96) 0.11 (0.40) 0.49 (0.9%) 321 (5.8%) 401 (7.3%) 0.66 (1.2%) 1.07 (1.2%) 1.07 (1.3.1%) 1.132 (20.6%) 1.052 (19.1%) 1.475 (26.8%) 2.48 (4.5%) 2.901 (52.7%) 2.901 (52.7%) 4.03 (7.3%) 4.03 (7.3%) 4.03 (7.3%) 4.03 (7.3%) 4.03 (7.3%) 4.03 (7.3%) 4.03 (7.3%) 4.09 (19.4%) | 0.115:<br>0.1984<br>0.192:<br>0.197:<br>0.0794<br>0.0694<br>0.0694<br>0.1199<br>0.1199<br>0.1634<br>0.0958<br>0.1799<br>0.3659<br>0.1799<br>0.3659<br>0.1724<br>0.0438<br>0. |
| HU - Recent hospitalization (-30 days to Index Rx date); n (%) HU - Old hospitalizations (-180 to -31 days); n (%) HU - Pays smear; n (%) HU - Pays smear; n (%) HU - Pays smear; n (%) HU - Postate sexam for DRE; n (%) HU - Bone mineral density; n (%) HU - Bone mineral density; n (%) HU - Bone mineral density; n (%) HU - Bone mineral density; n (%) HU - Postate sexam for DRE; n (%) HU - Postate sexam for DRE; n (%) Lab - Occurrence of 24-hour urine test; n (%) Lab - Occurrence of 24-hour urine tests ordered; n (%) Lab - Occurrence of rine albumin test ordered; n (%) Lab - Occurrence of urine albumin test ordered; n (%) Lab - Occurrence of urine albumin test ordered; n (%) Lab - Occurrence of urine albumin test ordered; n (%) Lab - Occurrence of urine albumin test ordered; n (%) Lab - Occurrence of urine albumin test ordered; n (%) SES Proxy - Low income indicator; n (%) | 0.15 (0.50) 617 (2.9%) 2,081 (9.5%) 2,081 (9.5%) 2,561 (12.1%) 380 (1.8%) 1,007 (4.7%) 987 (4.7%) 1,026 (4.8%) 4,955 (2.3.3%) 5,388 (25.4%) 5,388 (25.4%) 1,202 (5.7%) 11,639 (54.8%) 11,207 (52.8%) 28.11 (33.95) 6,063 (28.6%) 1,284 (6.0%) 1,284 (6.0%) 1,940 (94.0%) 0 (0.0%) | 1.52 (0.91) 0.12 (0.44) 13 (1.5%) 76 (8.7%) 108 (12.4%) 13 (2.4%) 13 (2.4%) 13 (2.4%) 13 (4.4%) 13 (4.4%) 13 (4.5%) 19 (2.2.5%) 196 (22.5%) 196 (22.5%) 196 (22.5%) 196 (22.5%) 196 (22.5%) 196 (23.5%) 194 (23.5%) 194 (45.2%) 194 (23.3%) 403 (46.3%) 468 (53.7%) 0 (0.0%) | 0.0213 0.0637 0.0956 0.0278 0.0278 0.0226 0.0144 0.0446 0.0191 0.0166 0.0680 0.0680 0.0680 0.0241 0.1255 0.1450 0.1450 0.1450 | 0.96 (0.98) 0.14 (0.44) 254 (2.8%) 841 (9.3%) 754 (8.4%) 261 (2.9%) 315 (3.5%) 497 (5.5%) 196 (2.2%) 1,562 (17.3%) 1,246 (13.8%) 2,455 (27.3%) 466 (5.2%) 2,611 (29.0%) 724 (8.0%) 0 (0.0%) 0 (0.0%) 0 (0.0%) | 1.39 (0.95) 0.08 (0.31) 1.8 (0.9%) 1.10 (5.7%) 1.10 (5.7%) 1.81 (9.4%) 8.8 (4.6.4%) 8.8 (4.6.4%) 3.9 (2.0%) 3.55 (18.4.4%) 2.89 (15.0%) 2.89 (15.0%) 2.89 (15.0%) 2.99 (1.1%) 8.62 (4.4.6%) 1.49 (7.7%) 2.4.65 (25.50) 0 (0.0%) 0 (0.0%) 0 (0.0%) | 0.4455 0.1576 0.1576 0.1414 0.1370 0.0351 0.0051 0.0058 0.0044 0.0139 0.00287 0.0342 0.0327 0.0327 0.03278 0.0112 #DIV/01 #DIV/01 #DIV/01 0.5226 | 1.53 (0.93) 0.25 (0.65) 2.465 (4.7%) 7.233 (13.9%) 5.207 (10.0%) 916 (1.8%) 2.664 (5.1%) 2.664 (5.1%) 2.514 (4.8%) 2.214 (4.3%) 18,258 (35.2%) 14,318 (27.6%) 19,220 (37.0%) 4,261 (8.2%) 21,500 (41.4%) 46,435 (89.5%) 28.06 (35.48) 0 (0.0%) 0 (0.0%) | 0.85 (1.58) 1.72 (0.98) 1.72 (0.98) 1.73 (0.98) 2.93 (10.8%) 4.7 (1.7%) 4.7 (1.7%) 1.94 (5.0%) 1.95 (3.4.6%) 8.56 (31.7%) 1.105 (40.9%) 1.105 (40.9%) 1.27 (47.3%) 2.507 (92.8%) 31.18 (43.28) 0 (0.0%) 0 (0.0%) | 0.0768 -0.189 0.2162 0.2003 0.1509 -0.0262 0.0076 -0.0079 -0.0093 -0.0286 0.0126 -0.0809 -0.0800 -0.0375 -0.1190 -0.1164 -0.0788 #DIV/OI #DIV/OI | 0.91 (1.77) 1.46 (0.95) 0.21 (0.59) 3,082 (3.8%) 9,241 (11.3%) 7,768 (9.5%) 1,296 (1.6%) 3,671 (4.5%) 3,501 (4.3%) 3,501 (4.3%) 3,240 (3.9%) 23,213 (28.3%) 19,706 (24.0%) 28,159 (34.3%) 5,463 (6.7%) 3,139 (40.3%) 57,642 (70.2%) 27,23 (33.78) 6,063 (7.4%) 1,284 (1.6%) 1,940 (24.3%) 2,315 (2.8%) 957 (1.2%) | 0.70 (1.45) 1.57 (0.96) 0.11 (0.40) 0.49 (0.9%) 321 (5.8%) 401 (7.3%) 401 (7.3%) 166 (1.2%) 220 (4.0%) 167 (3.0%) 1,052 (19.1%) 1,132 (20.6%) 1,052 (19.1%) 1,475 (26.8%) 1,474 (31.7%) 2,901 (52.7%) 29.28 (36.71) 194 (3.5%) 403 (7.3%) 403 (7.3%) 468 (8.5%) 136 (2.5%) | 0.115 0.198 0.192 0.197 0.079 0.034 0.043 0.043 0.197 0.119 0.119 0.163 0.095 0.179 0.365 0.172 0.279 0.436 0.018 |

Due to CMS cell suppression policy, all values less than 11 are denoted with \*\*

| | | | | | Δ. | FTER MA | ATCHING | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | OPTUM | | N. | MARKETSCAN | | | MEDICARE | | | POOLED | |
| Variable | Reference - Sitagliptin | Exposure - Dapagliflozin | St. Diff | Reference -<br>Sitagliptin | Exposure -<br>Dapagliflozin | St. Diff | Reference -<br>Sitagliptin | Exposure -<br>Dapagliflozin | St. Diff | Reference - Sitagliptin | Exposure - Dapagliflozin | n<br>St. Diff |
| Number of patients | 828 | 828 | | 1,687 | 1,687 | | 2,630 | 2,630 | | 5,145 | 5,145 | |
| Age - Continuousmean (sd) | 65.33 (9.96) | 65.27 (9.97) | 0.0060 | 59.19 (9.34) | 59.52 (8.66) | -0.0366 | 73.17 (5.93) | 73.25 (6.25) | -0.0131 | 67.32 (7.91) | 67.46 (7.78) | -0.0178 |
| Age Categories18 - 54: n (%) | 119 (14.4%) | 130 (15.7%) | -0.0364 | 489 (29.0%) | 413 (24.5%) | 0.1018 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 608 (11.8%) | 543 (10.6%) | 0.0381 |
| 55 - 64: n (%) | 232 (28.0%) | 224 (27.1%) | 0.0304 | 836 (49.6%) | 958 (56.8%) | -0.1447 | 0 (0.0%) | 0 (0.0%) | #DIV/01 | 1.068 (20.8%) | 1.182 (23.0%) | -0.0532 |
| 65 - 74: n (%) | 327 (39.5%) | 336 (40.6%) | -0.0225 | 262 (15.5%) | 228 (13.5%) | 0.0568 | 1.686 (64.1%) | 1,674 (63.7%) | 0.0083 | 2.013 (39.1%) | 2.010 (39.1%) | 0.0000 |
| >= 75; n (%) | 150 (18.1%) | 138 (16.7%) | 0.0369 | 100 (5.9%) | 88 (5.2%) | 0.0306 | 944 (35.9%) | 956 (36.3%) | -0.0083 | 1,094 (21.3%) | 1,094 (21.3%) | 0.0000 |
| Gender | | | | , , , , , | | | , | | | | | 1 |
| Male; n (%) | 440 (53.1%) | 452 (54.6%) | -0.0301 | 1,042 (61.8%) | 1,051 (62.3%) | -0.0103 | 1,371 (52.1%) | 1,349 (51.3%) | 0.0160 | 1,811 (35.2%) | 1,801 (35.0%) | 0.0042 |
| Female; n (%) | 388 (46.9%) | 376 (45.4%) | 0.0301 | 645 (38.2%) | 636 (37.7%) | 0.0103 | 1,259 (47.9%) | 1,281 (48.7%) | -0.0160 | 1,647 (32.0%) | 1,657 (32.2%) | -0.0043 |
| Geographic Region | | | | | | | | | | | | ↓ |
| Northeast; n (%) | 77 (9.3%) | 71 (8.6%) | 0.0245 | 197 (11.7%) | 192 (11.4%) | 0.0094 | 400 (15.2%) | 412 (15.7%) | -0.0138<br>-0.0141 | 477 (9.3%)<br>1.652 (32.1%) | 483 (9.4%)<br>1.668 (32.4%) | -0.0034 |
| Soutn; n (%)Midwest; n (%) | 463 (55.9%)<br>99 (12.0%) | 460 (55.6%)<br>119 (14.4%) | -0.0709 | 1,024 (60.7%)<br>252 (14.9%) | 1,010 (59.9%)<br>259 (15.4%) | -0.0139 | 1,189 (45.2%)<br>422 (16.0%) | 1,208 (45.9%)<br>379 (14.4%) | 0.0141 | 1,652 (32.1%)<br>521 (10.1%) | 1,668 (32.4%)<br>498 (9.7%) | 0.0134 |
| West: n (%) | 189 (22.8%) | 178 (21.5%) | 0.0703 | 206 (12.2%) | 219 (13.0%) | -0.0133 | 619 (23.5%) | 631 (24.0%) | -0.0117 | 808 (15.7%) | 809 (15.7%) | 0.0000 |
| Calendar Time - Year of Initiation (2014/15 - 2020) | 105 (22.0%) | 170 (21.3%) | 0.0313 | 200 (12.2%) | 219 (13.0%) | 0.0241 | 019 (23.370) | 031 (24.0%) | 0.0117 | 000 (15.770) | 003 (13.770) | |
| 2014-2015; n (%) | 257 (31.0%) | 270 (32.6%) | -0.0344 | 531 (31.5%) | 539 (32.0%) | -0.0107 | 755 (28.7%) | 790 (30.0%) | -0.0286 | 1,012 (19.7%) | 1,060 (20.6%) | -0.0224 |
| 2016; n (%) | 67 (8.1%) | 75 (9.1%) | -0.0357 | 399 (23.7%) | 408 (24.2%) | -0.0117 | 682 (25.9%) | 659 (25.1%) | 0.0184 | | | L |
| 2017; n (%) | 119 (14.4%) | 131 (15.8%) | -0.0391 | 364 (21.6%) | 343 (20.3%) | 0.0319 | 1,193 (45.4%) | 1,181 (44.9%) | 0.0100 | 1,312 (25.5%) | 1,312 (25.5%) | 0.0000 |
| 2018; n (%) | 140 (16.9%) | 125 (15.1%) | 0.0491 | 393 (23.3%) | 397 (23.5%) | -0.0047 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 140 (2.7%) | 125 (2.4%) | 0.0190 |
| 2019 - March 2020; n (%) | 245 (29.6%) | 227 (27.4%) | 0.0488 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 245 (4.8%) | 227 (4.4%) | 0.0191 |
| Combined comorbidity score, 180 daysmean (sd) | 2.54 (2.24) | 2.57 (2.25) | -0.0134<br>0.0000 | 1.64 (1.78) | 1.63 (1.82) | 0.0056 | 2.07 (2.19) | 2.02 (2.14) | 0.0231 | 2.00 (2.07) | 1.98 (2.06)<br>0.17 (0.04) | 0.0097 |
| Frailty Score: Empirical Version, 180 daysmean (sd) | 0.16 (0.05) | 0.16 (0.05) | 0.0000 | 0.15 (0.03) | 0.15 (0.03) | 0.0000 | 0.19 (0.06) | 0.19 (0.05) | 0.0000 | 0.17 (0.05) | 0.17 (0.04) | 0.0000 |
| DiabRen - CKD II; n (%) | 162 (19.6%) | 181 (21.9%) | -0.0567 | 339 (20.1%) | 341 (20.2%) | -0.0025 | 513 (19.5%) | 482 (18.3%) | 0.0307 | 675 (13.1%) | 663 (12.9%) | 0.0059 |
| DiabRen - CKD III: n (%) | 351 (42.4%) | 350 (42.3%) | 0.0020 | 492 (29.2%) | 508 (30.1%) | -0.0197 | 1.107 (42.1%) | 1,090 (41.4%) | 0.0142 | 1,458 (28.3%) | 1,440 (28.0%) | 0.0067 |
| DiabRen - Occurrence of Diabetic Nephropathy ; n (%) | 371 (44.8%) | 381 (46.0%) | -0.0241 | 558 (33.1%) | 570 (33.8%) | -0.0148 | 907 (34.5%) | 883 (33.6%) | 0.0190 | 1,278 (24.8%) | 1,264 (24.6%) | 0.0046 |
| DiabRen - Occurrence of Diabetic Neuropathy ; n (%) | 252 (30.4%) | 242 (29.2%) | 0.0262 | 357 (21.2%) | 328 (19.4%) | 0.0448 | 869 (33.0%) | 821 (31.2%) | 0.0386 | 1,121 (21.8%) | 1,063 (20.7%) | 0.0269 |
| DiabRen - Diabetic retinopathy ; n (%) | 99 (12.0%) | 90 (10.9%) | 0.0346 | 118 (7.0%) | 102 (6.0%) | 0.0406 | 285 (10.8%) | 309 (11.7%) | -0.0285 | 384 (7.5%) | 399 (7.8%) | -0.0113 |
| DiabRen - Diabetic foot ; n (%) | 18 (2.2%) | 26 (3.1%) | -0.0561 | 33 (2.0%) | 42 (2.5%) | -0.0337 | 92 (3.5%) | 88 (3.3%) | 0.0110 | 110 (2.1%) | 114 (2.2%) | -0.0069 |
| DiabRen - Diabetes with peripheral circulatory disorders ; n (%) | 74 (8.9%) | 86 (10.4%) | -0.0508<br>-0.0481 | 86 (5.1%) | 86 (5.1%) | 0.0000 | 335 (12.7%)<br>496 (18.9%) | 328 (12.5%) | 0.0060 | 409 (7.9%) | 414 (8.0%) | -0.0037<br>0.0088 |
| DiabRen - Hypertensive nephropathy; n (%) DiabRen - Hypertension : n (%) | 204 (24.6%)<br>750 (90.6%) | 221 (26.7%)<br>749 (90.5%) | 0.0034 | 316 (18.7%)<br>1,442 (85.5%) | 318 (18.9%)<br>1,429 (84.7%) | -0.0051<br>0.0225 | 2,483 (94.4%) | 465 (17.7%)<br>2,474 (94.1%) | 0.0310<br>0.0129 | 700 (13.6%)<br>3,233 (62.8%) | 686 (13.3%)<br>3,223 (62.6%) | 0.0088 |
| DiabRen - Hypotension : n (%) | 27 (3.3%) | 20 (2.4%) | 0.0541 | 21 (1.2%) | 23 (1.4%) | -0.0177 | 77 (2.9%) | 70 (2.7%) | 0.0123 | 104 (2.0%) | 090 (1.7%) | 0.0223 |
| DiabRen - Gout (acute/chronic) ; n (%) | 14 (1.7%) | 14 (1.7%) | 0.0000 | 31 (1.8%) | 38 (2.3%) | -0.0353 | 49 (1.9%) | 44 (1.7%) | 0.0150 | 063 (1.2%) | 058 (1.1%) | 0.0094 |
| DiabRen - Nephrolithiasis; n (%) | 20 (2.4%) | 17 (2.1%) | 0.0202 | 29 (1.7%) | 34 (2.0%) | -0.0223 | 54 (2.1%) | 49 (1.9%) | 0.0143 | 074 (1.4%) | 066 (1.3%) | 0.0087 |
| DiabRen - Proteinuria ; n (%) | 72 (8.7%) | 75 (9.1%) | -0.0140 | 40 (2.4%) | 42 (2.5%) | -0.0065 | 251 (9.5%) | 244 (9.3%) | 0.0069 | 323 (6.3%) | 319 (6.2%) | 0.0041 |
| DiabRen - Urinary tract infections (UTIs) ; n (%) | 78 (9.4%) | 79 (9.5%) | -0.0034 | 92 (5.5%) | 83 (4.9%) | 0.0270 | 405 (15.4%) | 396 (15.1%) | 0.0083 | 483 (9.4%) | 475 (9.2%) | 0.0069 |
| DiabRen - Genital infections; n (%) | 10 (1.2%) | 9 (1.1%) | 0.0094 | 25 (1.5%) | 26 (1.5%) | 0.0000 | 39 (1.5%) | 44 (1.7%) | -0.0159 | 049 (1.0%) | 053 (1.0%) | 0.0000 |
| DiabRen - Hypoglycemia v2; n (%) | 132 (15.9%) | 117 (14.1%) | 0.0504 | 155 (9.2%) | 145 (8.6%) | 0.0211 | 284 (10.8%) | 278 (10.6%) | 0.0065 | 416 (8.1%) | 395 (7.7%) | 0.0148 |
| DiabRen - Hyperglycemia; n (%) | 31 (3.7%)<br>22 (2.7%) | 30 (3.6%)<br>33 (4.0%) | -0.0053 | 70 (4.1%)<br>36 (2.1%) | 59 (3.5%)<br>37 (2.2%) | -0.0069 | 130 (4.9%)<br>78 (3.0%) | 144 (5.5%)<br>87 (3.3%) | -0.0270<br>-0.0172 | 161 (3.1%)<br>100 (1.9%) | 174 (3.4%)<br>120 (2.3%) | -0.0169<br>-0.0279 |
| DiabRen - Hyperkalemia; n (%) DiabRen - Hypovolemia/volume depletion; n (%) | 22 (2.7%) | 27 (3.3%) | -0.0723 | 44 (2.6%) | 39 (2.3%) | 0.0194 | 96 (3.7%) | 88 (3.3%) | 0.0218 | 118 (2.3%) | 115 (2.2%) | 0.0067 |
| Diables - 119 povolesma) voiume depiedon, ii (/a) | 22 (2.770) | 27 (5.570) | 0.0552 | 44 (2.0%) | 33 (2.3%) | 0.0154 | 30 (3.770) | 88 (3.370) | 0.0210 | 110 (2.570) | 113 (2.270) | 0.0007 |
| NephroTox - ACE inhibitors ; n (%) | 443 (53.5%) | 433 (52.3%) | 0.0240 | 899 (53.3%) | 905 (53.6%) | -0.0060 | 1,366 (51.9%) | 1,327 (50.5%) | 0.0280 | 1,809 (35.2%) | 1,760 (34.2%) | 0.0210 |
| NephroTox - ARBs ; n (%) | 428 (51.7%) | 430 (51.9%) | -0.0040 | 852 (50.5%) | 848 (50.3%) | 0.0040 | 1,371 (52.1%) | 1,400 (53.2%) | -0.0220 | 1,799 (35.0%) | 1,830 (35.6%) | -0.0126 |
| NephroTox - Loop Diuretics ; n (%) | 153 (18.5%) | 159 (19.2%) | -0.0179 | 222 (13.2%) | 241 (14.3%) | -0.0319 | 653 (24.8%) | 634 (24.1%) | 0.0163 | 806 (15.7%) | 793 (15.4%) | 0.0083 |
| NephroTox - Thiazide diuretics ; n (%) | 169 (20.4%) | 159 (19.2%) | 0.0301 | 293 (17.4%) | 300 (17.8%) | -0.0105 | 474 (18.0%) | 476 (18.1%) | -0.0026 | 643 (12.5%) | 635 (12.3%) | 0.0061 |
| NephroTox - Mineralocorticoid receptor antagonist; n (%) | 42 (5.1%) | 49 (5.9%) | -0.0351<br>0.0269 | 83 (4.9%) | 89 (5.3%) | -0.0182 | 129 (4.9%) | 126 (4.8%) | 0.0047 | 171 (3.3%) | 175 (3.4%) | -0.0056 |
| NephroTox - NSAIDs; n (%) | 142 (17.1%)<br>202 (24.4%) | 133 (16.1%) | 0.0258 | 299 (17.7%) | 288 (17.1%) | 0.0158<br>-0.0152 | 439 (16.7%)<br>671 (25.5%) | 411 (15.6%)<br>676 (25.7%) | 0.0299<br>-0.0046 | 581 (11.3%)<br>873 (17.0%) | 544 (10.6%)<br>869 (16.9%) | 0.0224 |
| NephroTox - PPIs; n (%) NephroTox - H2RAs: n (%) | 202 (24.4%)<br>51 (6.2%) | 193 (23.3%) | 0.0258 | 318 (18.9%)<br>58 (3.4%) | 329 (19.5%)<br>59 (3.5%) | -0.0152 | 6/1 (25.5%)<br>195 (7.4%) | 205 (7.8%) | -0.0046 | 246 (4.8%) | 245 (4.8%) | 0.0027 |
| NephroTox - H2RAs; n (%) NephroTox - Antivirals/Antiretrovirals/Antimicrobials: n (%) | 51 (6.2%)<br>12 (1.4%) | 40 (4.8%)<br>13 (1.6%) | -0.0165 | 58 (3.4%)<br>14 (0.8%) | 59 (3.5%)<br>17 (1.0%) | -0.0055 | 195 (7.4%)<br>28 (1.1%) | 205 (7.8%)<br>32 (1.2%) | -0.0151 | 040 (0.8%) | 045 (0.9%) | -0.0109 |
| responsible in the contrast contrast contrast contrast, in (10) | 12 (1.4/0) | 13 (1.0/0) | 0.0103 | 17 (0.0/0) | 1/ (1.0/0) | 0.0212 | 20 (1.1/0) | JE (1.E/0) | 0.0054 | 0.00 (0.070) | 0.45 (0.570) | 0.0103 |
| DM Medications - 1st and 2nd Generation SUs ; n (%) | 362 (43.7%) | 366 (44.2%) | -0.0101 | 641 (38.0%) | 630 (37.3%) | 0.0144 | 1,144 (43.5%) | 1,160 (44.1%) | -0.0121 | 1,506 (29.3%) | 1,526 (29.7%) | -0.0088 |
| DM Medications - AGI & Meglinitides; n (%) | 17 (2.1%) | 17 (2.1%) | 0.0000 | 34 (2.0%) | 30 (1.8%) | 0.0146 | 126 (4.8%) | 131 (5.0%) | -0.0093 | 143 (2.8%) | 148 (2.9%) | -0.0060 |
| DM Medications - DPP-4 Inhibitors (excluding sitagliptin); n (%) | 113 (13.6%) | 120 (14.5%) | -0.0259 | 148 (8.8%) | 154 (9.1%) | -0.0105 | 372 (14.1%) | 404 (15.4%) | -0.0367 | 485 (9.4%) | 524 (10.2%) | -0.0269 |
| DM Medications - Glitazones ; n (%) | 98 (11.8%) | 101 (12.2%) | -0.0123 | 198 (11.7%) | 203 (12.0%) | -0.0093 | 318 (12.1%) | 307 (11.7%) | 0.0124 | 416 (8.1%) | 408 (7.9%) | 0.0074 |
| DM Medications - GLP-1 RA ; n (%) | 207 (25.0%) | 198 (23.9%) | 0.0256 | 312 (18.5%) | 332 (19.7%) | -0.0305 | 497 (18.9%) | 460 (17.5%) | 0.0363 | 704 (13.7%) | 658 (12.8%) | 0.0265 |
| DM Medications - Insulins; n (%) | 268 (32.4%) | 276 (33.3%) | -0.0192 | 529 (31.4%) | 507 (30.1%) | 0.0282 | 994 (37.8%) | 966 (36.7%) | 0.0228 | 1,262 (24.5%) | 1,242 (24.1%) | 0.0093 |
| DM Medications - Metformin ; n (%) | 487 (58.8%) | 497 (60.0%) | -0.0244<br>0.0159 | 1,019 (60.4%) | 1,020 (60.5%) | -0.0020<br>-0.0460 | 1,447 (55.0%) | 1,468 (55.8%) | -0.0161<br>0.0042 | 1,934 (37.6%)<br>219 (4.3%) | 1,965 (38.2%)<br>213 (4.1%) | -0.0124<br>0.0100 |
| DM Medications-SGLT-2 Inhibitors (excluding dapagliflozin); n (%) DM Medications-Number of antiDM medications at index datemean (sd) | 58 (7.0%)<br>2.80 (0.96) | 55 (6.6%)<br>2.80 (0.96) | 0.0159 | 136 (8.1%)<br>2.69 (0.87) | 158 (9.4%)<br>2.70 (0.93) | -0.0460 | 161 (6.1%)<br>2.82 (0.94) | 158 (6.0%)<br>2.83 (0.99) | -0.0104 | 2.77 (0.92) | 2.78 (0.97) | -0.0106 |
| DIM Medications - Number of anti-DM infedications at index dateinean (su) | 2.00 (0.50) | 2.00 (0.50) | 0.0000 | 2.03 (0.07) | 2.70 (0.55) | -0.0111 | 2.02 (0.54) | 2.03 (0.33) | 0.0104 | 2.77 (0.32) | 2.70 (0.57) | 0.0100 |
| CV Comorbidity - Acute and Old MI ; n (%) | 26 (3.1%) | 28 (3.4%) | -0.0169 | 20 (1.2%) | 25 (1.5%) | -0.0260 | 126 (4.8%) | 124 (4.7%) | 0.0047 | 152 (3.0%) | 152 (3.0%) | 0.0000 |
| CV Comorbidity - Any Heart failure (HF); n (%) | 85 (10.3%) | 90 (10.9%) | -0.0195 | 82 (4.9%) | 86 (5.1%) | -0.0092 | 419 (15.9%) | 379 (14.4%) | 0.0418 | 504 (9.8%) | 469 (9.1%) | 0.0239 |
| CV Comorbidity - Hospitalization for CHF ; n (%) | 21 (2.5%) | 23 (2.8%) | -0.0187 | 19 (1.1%) | 23 (1.4%) | -0.0270 | 86 (3.3%) | 78 (3.0%) | 0.0172 | 107 (2.1%) | 101 (2.0%) | 0.0071 |
| CV Comorbidity - Atrial fibrillation; n (%) | 65 (7.9%) | 62 (7.5%) | 0.0150 | 71 (4.2%) | 75 (4.4%) | -0.0099 | 352 (13.4%) | 349 (13.3%) | 0.0029 | 417 (8.1%) | 411 (8.0%) | 0.0037 |
| CV Comorbidity - Other dysrythmias ; n (%) | 107 (12.9%) | 108 (13.0%) | -0.0030 | 113 (6.7%) | 115 (6.8%) | -0.0040 | 418 (15.9%) | 408 (15.5%) | 0.0110 | 525 (10.2%) | 516 (10.0%) | 0.0066 |
| CV Comorbidity - Valve disorder; n (%) | 18 (2.2%) | 17 (2.1%) | 0.0069 | 10 (0.6%) | 15 (0.9%) | -0.0348 | 90 (3.4%) | 94 (3.6%) | -0.0109 | 108 (2.1%) | 111 (2.2%) | -0.0069 |

| Automatic Auto | CV Comorbidity - Implantable cardioverter defibrillator ; n (%) | 9 (1.1%) | 10 (1.2%) | -0.0094 | 9 (0.5%) | 10 (0.6%) | -0.0135 | 47 (1.8%) | 47 (1.8%) | 0.0000 | 056 (1.1%) | 057 (1.1%) | 0.0000 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Description of the control of the | | . (,-) | | | - () | | | | (=.0,-) | | , | | 0.0082 |
| Secretary Secr | | ***(******) | 00 () | | 00 (2.07.7) | 00 (2.0) | | 200 (20.27.) | () | | ( , | | 0.0270 |
| Company Comp | | | 686 (82,9%) | 0.0107 | | | | | | | | | 0.0060 |
| Community Amperes internal From Principal Conference (1998) Co | | | | | | | | | | | 178 (3.5%) | | 0.0167 |
| Comment person | CV Comorbidity - Unstable Angina ; n (%) | 24 (2.9%) | 17 (2.1%) | 0.0513 | 14 (0.8%) | 12 (0.7%) | 0.0116 | 42 (1.6%) | 37 (1.4%) | 0.0165 | 066 (1.3%) | 054 (1.0%) | 0.0281 |
| Marchen Marc | | | | -0.0501 | | | -0.0306 | | | 0.0110 | 491 (9.5%) | 494 (9.6%) | -0.0034 |
| Page | CV Comorbidity - Stroke/TIA; n (%) | 23 (2.8%) | 25 (3.0%) | -0.0119 | 20 (1.2%) | 17 (1.0%) | 0.0192 | 84 (3.2%) | 82 (3.1%) | 0.0057 | 107 (2.1%) | 107 (2.1%) | 0.0000 |
| Application | CV Comorbidity - Pulmonary hypertension/Other pulmonary heart disease; n (%) | 20 (2.4%) | 19 (2.3%) | 0.0066 | 16 (0.9%) | 16 (0.9%) | 0.0000 | 81 (3.1%) | 63 (2.4%) | 0.0428 | 101 (2.0%) | 082 (1.6%) | 0.0301 |
| Application | | | | | | | | | | | | | |
| Company Comp | | | | | | | | | | | , , , | ,- ( , | |
| Visibility Vis | | | | | | | | 00. (00,10) | | | , . , , | , , | |
| Continues and present (Column Column Colum | | | | | | | | 0. (0.071) | | | , | | |
| Contention between preference Content Co | | | | | | | | | | | | | |
| Comment Comm | 7 17 | | | | | | | | | | , , . , | ,- (- , | |
| Controlled Application A | | | | 0.00.0 | | | | | | | | | |
| | CV Medication - Use of other hypertension drugs ; n (%) | 75 (9.1%) | 79 (9.5%) | -0.0138 | 156 (9.2%) | 167 (9.9%) | -0.0238 | 372 (14.1%) | 341 (13.0%) | 0.0321 | 447 (8.7%) | 420 (8.2%) | 0.0180 |
| | | | | 0.0751 | | | 0.0120 | / | | 0.0001 | 0.45 (1.5.40/) | 022 (4 6 20/) | 0.0054 |
| Page | | () | | | (, | | | 000 (201111) | (= 0.0,1-) | | ( / | | |
| 22.28 20.29 20.2 | | | | 0.00-0 | | | | | | | (0.2) | 102 (01.112) | |
| 1956/279 1961/279 | | 00 (2011) | 00 (20.0) | | 0.0 (0.0) | | | 000 (22.07.) | | | - ( , | ( / | |
| 15.5 | | | | | | | | | | | | | |
| | | | | | | | | | | | - ( , | ( / | |
| 15/23/10 | The state of the s | | | | | | | | | | , | | |
| Marchester Mar | | | | | | | | | | | | | 0.0131 |
| The Markstein Land articonomers, in No. 177,05/75 1791/150 0.015 779,15/50 0.027 779,07/76 0.015 0.001 0.0 | | | | | | | | | | | - ( , | | 0.0163 |
| | | (27.070) | (20.5/0) | | 120,070/ | | | (15.670) | 222 (24.070) | | | | |
| | Other Medication - Use of anticonvulsants; n (%) | 171 (20.7%) | 178 (21.5%) | -0.0196 | 279 (16.5%) | 262 (15.5%) | 0.0273 | 729 (27.7%) | 681 (25.9%) | 0.0406 | 900 (17.5%) | 859 (16.7%) | 0.0212 |
| | Other Medication - Use of antidepressants; n (%) | 219 (26.4%) | 214 (25.8%) | 0.0137 | 415 (24.6%) | 390 (23.1%) | 0.0352 | 804 (30.6%) | 778 (29.6%) | 0.0218 | 1,023 (19.9%) | 992 (19.3%) | 0.0151 |
| | Other Medication - Use of antiparkinsonian meds ; n (%) | 25 (3.0%) | 24 (2.9%) | 0.0059 | 32 (1.9%) | 38 (2.3%) | -0.0279 | 118 (4.5%) | 115 (4.4%) | 0.0048 | 143 (2.8%) | 139 (2.7%) | 0.0061 |
| 20th Methodiscon: Used methodiscophysics, (c) (1) (2) | Other Medication - Use of dementia meds ; n (%) | 21 (2.5%) | 16 (1.9%) | 0.0409 | 0 (0.0%) | 3 (0.2%) | -0.0633 | 124 (4.7%) | 125 (4.8%) | -0.0047 | 145 (2.8%) | 141 (2.7%) | 0.0061 |
| | Other Medication - Use of antipsychotics ; n (%) | 22 (2.7%) | 22 (2.7%) | 0.0000 | 21 (1.2%) | 22 (1.3%) | -0.0090 | 87 (3.3%) | 89 (3.4%) | -0.0056 | 109 (2.1%) | 111 (2.2%) | -0.0069 |
| | Other Medication - Use of anxiolytics/hypnotics ; n (%) | 52 (6.3%) | 51 (6.2%) | 0.0041 | 122 (7.2%) | 111 (6.6%) | 0.0237 | 207 (7.9%) | 197 (7.5%) | 0.0150 | 259 (5.0%) | 248 (4.8%) | 0.0093 |
| Commendation - Used Participations (agents, p. 16) 164 (12.68) 164 | Other Medication - Use of Benzodiazepines ; n (%) | | 98 (11.8%) | -0.0746 | 167 (9.9%) | | | 340 (12.9%) | 334 (12.7%) | | | | -0.0109 |
| 20th Medication : Used for all anticognomists, (10) 2017 36 (8 8 2 24) 30189 51 (8 8 3) 39 (5 5 3) 40177 34 (6 12 24) 3181 (2 7 8) 400 (7 7 9 24) 400 (7 7 9 24) 400 (7 7 9 24) 400 (7 9 24) | Other Medication - Use of COPD/asthma meds; n (%) | | | 0.000 | 277 (16.4%) | | | | | 0.00.0 | (= ,) | | 0.000 |
| 1902 | Other Medication - Use of antiplatelet agents; n (%) | | | | 238 (14.1%) | | | | | | | | 0.0000 |
| Identife-Ancion/Drug Rouse or Dependence: n Ci 15 15 15 15 15 15 15 1 | Other Medication - Use of or al anticoagulants ; n (%) | | | | 0= () | | | | | 0.000 | (0, | | |
| | Other Medication - Use of opioids ; n (%) | 190 (22.9%) | 188 (22.7%) | 0.0048 | 419 (24.8%) | 410 (24.3%) | 0.0116 | 708 (26.9%) | 717 (27.3%) | -0.0090 | 898 (17.5%) | 905 (17.6%) | -0.0026 |
| | | | | | | | | | | | // | / | |
| No. Number of Cardiologist vistsmen (pl) 1.74 (4.21) 1.67 (4.26) 0.0161 | | | | 0.000- | | | 0.00 | | | 0.0000 | -/ (// | | 0.00.0 |
| Number of Prophenologist visitmen (gr) | Lifestyle*-3moxing, if (/a) | 88 (10.0%) | 52 (11.176) | -0.0101 | 00 (3.2%) | 77 (4.0%) | 0.0270 | 350 (14.6%) | 300 (14.070) | 0.0000 | 470 (3.370) | 400 (5.570) | 0.0000 |
| Number of Prophenologist visitmen (gr) | HU - Number of Cardiologist visits mean (sd) | 1.74 (4.42) | 1.67 (4.26) | 0.0161 | 0.90 (3.32) | 0.86 (2.40) | 0.0138 | 2.18 (5.13) | 2.06 (5.04) | 0.0236 | 1.69 (4.50) | 1.60 (4.22) | 0.0206 |
| HV-Number of fractional pages visitsmean (pd) 0.904 at 0.68 (1.87) 0.0914 0.0814 0.0812 0.0914 0.0914 0.0915 0.0915 0.0914 0.091 | | | | | | | | | | | 0.57 (2.48) | | 0.0072 |
| HU-Number of friends 13.24 (19.07) 12.07 (15.06) 0.0664 7.27 (7.55) 7.76 (8.95) 0.0584 10.35 (14.68) 0.72 (14.87) 0.023 0.381 (13.74) 0.021 | | | | -0.0414 | | | | | | 0.0359 | 1.19 (4.95) | 1.13 (3.85) | 0.0135 |
| NU-Number of Distinct Medication Prescriptions (premarized to generics)mean (pd) 33.68 (29.55) 33.55 (0.44) 0.0120 26.94 (17.22) 26.88 (16.42) 0.0026 35.51 (26.27) 35.61 (25.53) 0.0039 32.44 (14.43) 0.0012 0.0014 0 | | | | | | | -0.0584 | | | -0.0230 | | 9.97 (13.43) | -0.0103 |
| NU-Number of Distinct Medication Prescriptions (ong generalized to generics)mean (sd) 0.35 (29.55) 33.55 (20.44) 0.013 0.012 0.013 (2.55) 0.012 0.022 (2.05) 0.022 (0.05) 0.023 (0.05) 0.020 0.021 (0.022) 0.022 (0.05) 0.022 (0.05) 0.023 (0.05) 0.020 0.021 (0.022) 0.022 (0.05) 0.023 (0.05) 0.020 0.021 (0.022) 0.022 (0.05) 0.023 (0.05) 0.020 0.021 (0.022) 0.022 (0.05) 0.020 0.021 (0.022) 0.022 (0.05) 0.023 (0.05) 0.020 0.021 (0.022) 0.022 (0.05) 0.023 (0.05) 0.020 0.020 (0.022) 0.020 0.020 (0.022) 0.022 (0.022) 0.022 (0. | HU - Number of Emergency Department (ED) visitsmean (sd) | 0.56 (1.88) | 0.54 (1.87) | 0.0107 | 0.20 (1.55) | 0.19 (1.62) | 0.0063 | 0.60 (1.52) | 0.55 (1.35) | 0.0348 | 0.46 (1.59) | 0.43 (1.53) | 0.0192 |
| Hu-Number of flectrocardingam Performedmean (g) | | 33.68 (29.55) | 33.35 (20.44) | 0.0130 | 26.94 (17.22) | 26.88 (16.42) | 0.0036 | 35.51 (26.27) | 35.61 (25.53) | -0.0039 | 32.41 (24.30) | 32.38 (22.11) | 0.0013 |
| HU-Number of Flettrocardiogram Performedman (sd) | HU - Number of Echocardiogrammean (sd) | 0.29 (1.50) | 0.31 (1.59) | -0.0129 | 0.13 (0.52) | 0.12 (0.42) | 0.0212 | 0.22 (0.60) | 0.23 (0.65) | -0.0160 | 0.20 (0.80) | 0.21 (0.82) | -0.0123 |
| HU-Number of Hospitalizations during CAPmean (cd) 0.12 (0.44) 0.12 (0.44) 0.12 (0.44) 0.12 (0.44) 0.0000 0.08 (0.33) 0.08 (0.32) 0.0000 0.14 (0.47) 0.13 (0.44) 0.0220 0.12 (0.42) 0.11 (0.40) 0.0244 HU-Recent hospitalization (3.0 days to index Red arely, (n/s) 9 (1.1%) 19 | | 0.77 (1.86) | 0.77 (1.85) | | 0.51 (1.17) | 0.47 (0.96) | | 0.87 (1.61) | 0.85 (1.59) | 0.0125 | 0.74 (1.53) | | |
| HU-Rent hospitalization (30 days to index Red ate); n (%) 9 (1.1%) 13 (1.6%) 9 (2.1%) 9 (2.9%) 9 (2.9%) 9 (2.9%) 9 (2.9%) 9 (2.9%) 9 (2.9%) 15 (4.9%) 9 (2.9%) 16 (4.9%) 16 (4.9%) 17 (4.6%) 9 (2.3%) 18 (2.2%) 0.0026 18 (1.7%) 19 (2.9%) 0.0026 18 (1.7%) 0.0000 18 (1.7%) 18 (1.1%) 18 (1.1%) 10 (1.2.6%) 19 (2.9%) 0.0026 18 (1.9%) 15 (1.9%) 15 (1.9%) 15 (1.9%) 15 (1.9%) 15 (1.9%) 15 (1.9%) 16 (1.9%) 17 (1.6%) 18 (1.2%) 0.0026 17 (1.6%) 18 (1.2%) 0.0026 17 (1.6%) 18 (1.2%) 0.0026 18 (1.7%) 0.0010 18 | | 2.00 (2.22) | | 0.0.00 | 2.00 (0.00) | 2.00 (0.00) | | 2.1.0 (0.00) | | | | | 0.0000 |
| HU-Old hospitalizations (180 to -31 days); n (%) 99 (5.9%) 99 (5.9 | | | | | | | | | | | | | 0.0244 |
| HU-Mammogram; n (%) 92 (11.1%) 104 (12.6%) -0.0464 164 (9.7%) 154 (9.1%) -0.0266 -0.02 | | | | | | | | | | 0.000. | . ( , | , | 0.0000 |
| HU-Papsmear; n(%) 15(1.8%) 15( | | | | | | | | | | | ( , | | _ |
| HU-Prostate exam for DRE; n (%) 41 (5.0%) 37 (4.5%) 0.0235 80 (4.7%) 76 (4.5%) 0.0095 171 (6.5%) 178 (6.8%) 0.0120 212 (4.1%) 215 (4.2%) 0.0055 HU-Flexible Sigmoidoscopy or Colonoscopy; n (%) 29 (3.5%) 32 (3.9%) 20 (3.5%) 37 (4.5%) 0.0248 32 (3.9%) 37 (2.2%) 0.0215 21 (4.7%) 130 (4.9%) 130 (4.9%) 157 (3.2%) 0.0055 HU-Flexible Sigmoidoscopy or Colonoscopy; n (%) 29 (3.5%) 30 (3.9%) 109 (4.1%) 128 (4.9%) 0.0386 138 (2.7%) 130 (4.9%) 157 (3.2%) 0.0055 HU-Flexible Sigmoidoscopy or Colonoscopy; n (%) 128 (4.9%) 128 (4.9%) 130 (4.9%) 157 (3.2%) 0.0055 HU-Flexible Sigmoidoscopy or Colonoscopy; n (%) 128 (4.9%) 128 (4.9%) 128 (4.9%) 130 (4.9%) 128 (4.9%) 100 (4.1%) 128 (4.9%) 128 (4.9%) 130 (4.9%) 100 (4.1%) 128 (4.9%) 100 (4.1%) 128 (4.9%) 128 (4.9%) 130 (4.9%) 100 (4.1%) | | | | | | | | | | | | | -0.0114 |
| HU-Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%) 29 (3.5%) 32 (3.9%) -0.0212 90 (5.3%) 32 (3.9%) -0.0212 90 (5.3%) 37 (2.2%) -0.0212 124 (4.7%) 130 (4.9%) -0.094 157 (3.1%) 150 (2.1%) 150 (2.1%) 150 (2.1.%) 1 | | | | | | | | | | | , | | |
| HU-Bone mineral density; n (%) 33 (4.0%) 37 (4.5%) -0.0248 32 (1.9%) 37 (2.5%) -0.0212 124 (4.7%) 130 (4.9%) -0.0094 157 (3.1%) 167 (3.2%) -0.0055 HU-Flu vaccine; n (%) 191 (23.1%) 186 (22.5%) 0.0143 37 (18.2%) 305 (18.1%) 0.0026 925 (35.2%) 906 (34.4%) 0.0168 1,116 (21.7%) 1,092 (21.2%) 0.017 140 (20.0%) 1,016 (1.7%) 1,016 (1.9%) 1,020 (21.2%) 0.0075 144 (1.9%) 1,020 (21.2%) 1,016 (19.7%) 1,020 (21.2%) | | | | | | | | | | | | | |
| HU-Flu vaccine; n (%) 191(23.1%) 186(22.5%) 0.0143 307(18.2%) 305(18.1%) 0.026 925(35.2%) 906(34.4%) 0.0168 1,116(21.7%) 1,092(21.2%) 0.017 185(23.2%) 185(23.9%) 0.0215 227(13.5%) 244(14.5%) 0.028 838(31.9%) 831(16.6%) 0.0064 1,030(20.0%) 1,016(19.7%) 0.0075 1,0076(10.9%) 0.0081 1,416(27.5%) 1,023(27.7%) 0.0084 1,030(20.0%) 1,016(19.7%) 0.0075 1,020(20.0%) 1,016(19.7%) 0.0075 1,020(20.0%) 1,016(19.7%) 0.0075 1,020(20.0%) 1,016(19.7%) 0.0075 1,020(20.0%) 1 | | | | | | | | | | | ( | | |
| HU-Pneumococcal vaccine; n (%) 122 (2.2.%) 185 (22.3%) 244 (14.5%) 244 (14.5%) 244 (14.5%) 244 (14.5%) 244 (14.5%) 244 (14.5%) 245 (13.5%) 244 (14.5%) 244 (14.5%) 245 (13.5%) 244 (14.5%) 244 (14.5%) 245 (13.5%) 244 (14.5%) 244 (14.5%) 245 (13.5%) 244 (14.5%) 244 (14.5% | | | | | | | | | | | | | |
| Lab - Occurrence of 24-hour urine test; n (%) Lab - Occurrence of 24-hour urine test; n (%) Lab - Occurrence of Creatinine tests ordered; n (%) A8 (5.8%) 50 (6.0%) -0.086 53 (8.7%) -0.085 71 (4.2%) 70 (4.1%) -0.095 20 (37.7%) -0.004 -0.0081 -0.00 | | | | 0.00.0 | | | 0.0000 | | | 0.0200 | | | 0.00 |
| Lab - Occurrence of creatinine tests ordered; n (%) 48 (5.8%) 50 (6.0%) -0.0085 71 (4.2%) 70 (4.1%) -0.0050 203 (7.7%) 188 (7.1%) 0.0229 251 (4.9%) 238 (4.6%) 0.0141 1,634 (31.8%) 1,637 (32.8%) -0.021 1,634 (31.8%) 1,637 (32.8%) -0.021 1,637 (31.8%) 1,637 (32.8%) -0.021 1,637 (31.8%) 1,637 (32.8%) | HU - Pneumococcal vaccine ; n (%) | 192 (23.2%) | 185 (22.3%) | 0.0215 | 227 (13.5%) | 244 (14.5%) | -0.0288 | 838 (31.9%) | 831 (31.6%) | 0.0064 | 1,030 (20.0%) | 1,016 (19.7%) | 0.0075 |
| Lab - Occurrence of creatinine tests ordered; n (%) 48 (5.8%) 50 (6.0%) -0.0085 71 (4.2%) 70 (4.1%) -0.0050 203 (7.7%) 188 (7.1%) 0.0229 251 (4.9%) 238 (4.6%) 0.0141 1,634 (31.8%) 1,637 (32.8%) -0.021 1,634 (31.8%) 1,637 (32.8%) -0.021 1,637 (31.8%) 1,637 (32.8%) -0.021 1,637 (31.8%) 1,637 (32.8%) | | | | | | | 1 | | | | | | 4 |
| Lab - Occurrence of urine albumin test ordered; n(%) 412 (49.8%) 445 (53.7%) -0.0781 -0.0 | | | | | | | | | | | | | |
| Lab - Occurrence of HgAlc test; n (%) 372 (44.9%) 376 (45.4%) -0.0100 134 (7.9%) 135 (8.0%) -0.0037 2,454 (93.3%) 2,439 (92.7%) 0.0235 2,826 (54.9%) 2,815 (54.7%) 0.0040 (54.9%) 2.815 (54.7%) 0.0040 (54.9%) 2.815 (54.7%) 0.0040 (54.9%) 2.815 (54.9%) 2.815 (54.7%) 0.0040 (54.9%) 2.815 (54.9%) 2.8 | | (0.07.7) | 0.0 (0.07.) | | | | | | () | | | | |
| SES Proxy-Copay for pharmacy cost (charges in U.S. \$)mean (sd) 33.75 (44.90) 32.86 (35.48) 0.022 23.59 (24.04) 23.70 (24.63) 0.0045 31.51 (40.70) 31.37 (43.52) 0.0033 29.27 (36.89) 29.09 (37.01) 0.0045 SES Proxy-Low income indicator; n (%) 0.0535 0 (0.0%) | | | | 0.0.0 | | | | , | , , , , | | | ,, | |
| SES Proxy - Low income indicator; n (%) 213 (25.7%) 194 (23.4%) 0.0535 0 (0.0%) 0 (0.0%) #DIV/0! 0 (0.0%) #DIV/0! 213 (4.1%) 194 (3.8%) 0.0154 (5.5F) roxy - Business type | Lab - Occurrence of HgA1c test; n (%) | 372 (44.9%) | 376 (45.4%) | -0.0100 | 134 (7.9%) | 135 (8.0%) | -0.0037 | 2,454 (93.3%) | 2,439 (92.7%) | 0.0235 | 2,826 (54.9%) | 2,815 (54.7%) | 0.0040 |
| SES Proxy - Low income indicator; n (%) 213 (25.7%) 194 (23.4%) 0.0535 0 (0.0%) 0 (0.0%) #DIV/0! 0 (0.0%) #DIV/0! 213 (4.1%) 194 (3.8%) 0.0154 (5.5F) roxy - Business type | | | | | | | | | | | | | |
| SES Proxy - Business type | | | | | | | | | | | | | 0.0049 |
| Commercial; n (%) 354 (42.8%) 361 (43.6%) -0.0162 0 (0.0%) 0 (0.0%) #DIV/0! 0 (0.0%) #DIV/0! 354 (6.9%) 361 (7.0%) -0.0033 | , | 213 (25.7%) | 194 (23.4%) | 0.0535 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 213 (4.1%) | 194 (3.8%) | 0.0154 |
| | , , | ļ | | | | <b></b> | <u> </u> | | ļ | 1 | | ļ | |
| Nedicare; n (%) 474 (57.2%) 467 (56.4%) 0.0162 0 (0.0%) 0 (0.0%) #DIV/0! 0 (0.0%) #DIV/0! 474 (9.2%) 467 (9.1%) 0.0035 | | 00.(.2.0,1.) | | | | | | | | | | | |
| | Medicare; n (%) | 474 (57.2%) | 467 (56.4%) | 0.0162 | U (U.0%) | U (U.0%) | #DIV/0! | υ (υ.0%) | U (U.0%) | #DIV/0! | 4/4 (9.2%) | 46 / (9.1%) | 0.0035 |

| SES Proxy - Insurance Plan type | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Comprehensive; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 117 (6.9%) | 132 (7.8%) | -0.0345 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 117 (2.3%) | 132 (2.6%) | -0.0194 |
| HMO; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 161 (9.5%) | 176 (10.4%) | -0.0301 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 161 (3.1%) | 176 (3.4%) | -0.0169 |
| PPO; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 924 (54.8%) | 918 (54.4%) | 0.0080 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 924 (18.0%) | 918 (17.8%) | 0.0052 |
| Others; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 485 (28.7%) | 461 (27.3%) | 0.0312 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 485 (9.4%) | 461 (9.0%) | 0.0138 |
| SES Proxy - Dual status code (with Medicaid); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 778 (29.6%) | 817 (31.1%) | -0.0326 | 778 (15.1%) | 817 (15.9%) | -0.0221 |